

#### CLINICAL STUDY PROTOCOL

Study Title: A Phase 1b, Randomized, Blinded, Placebo-Controlled

Dose-Escalation Study of the Safety and Biological Activity of GS-9620 in HIV-1 Infected, Virologically Suppressed Adults

**Sponsor:** Gilead Sciences, Inc.

333 Lakeside Drive Foster City, CA 94404

**IND Number:** 122452

EudraCT Number:Not ApplicableClinical Trials.gov Identifier:NCT02858401Indication:HIV-1 Infection

**Protocol ID:** GS-US-382-1450

Clinical Program Manager: Name:

Name: PPD Telephone: PPD

Fax:

PPD

**Gilead Medical Monitor:** Name:

Name: PPD Telephone: PPD

Fax: PPD

Mobile: PPD

Gilead Study Director: Name: PPD

Telephone: PPD

Fax: PPD Mobile: PPD

**Protocol Version/Date:** Amendment 7: 16 January 2019

Amendment 6: 07 June 2018

Amendment 5: 18 October 2017

Amendment 4: 13 October 2016

Amendment 3: 29 June 2015

Amendment 2: 15 December 2014

Amendment 1: 14 November 2014

Original: 16 September 2014

#### CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# TABLE OF CONTENTS

| TABLI | E OF CONTENTS | 2 |
|--------|--------------------------------------------------------------|----|
| LIST C | OF IN-TEXT TABLES | 5 |
| LIST C | OF IN-TEXT FIGURES | 5 |
| PROTO | OCOL SYNOPSIS | 6 |
| | SARY OF ABBREVIATIONS AND DEFINITION OF TERMS | |
| | NTRODUCTION | |
| | .1. Background | |
| 1. | .2. GS-9620 | |
| | 1.2.2. Preclinical Pharmacology and Toxicology | |
| | 1.2.3. Clinical Trials of GS-9620 | 27 |
| 1. | .3. Rationale for This Study | |
| 1. | .4. Rationale for Dose Selection/Dosing Interval | |
| 1. | .5. Rationale for Biomarker Testing. | |
| 1. | .6. Compliance | 34 |
| 2. O | DBJECTIVES | 35 |
| | TUDY DESIGN | 36 |
| | .1. Endpoints | |
| | 2. Study Design | |
| | .4. Duration of Treatment. | |
| | UBJECT POPULATION | |
| | .1. Number of Subjects and Subject Selection | |
| | 3. Exclusion Criteria (All Cohorts) | |
| | .4. Other Protocol Restrictions | |
| | NVESTIGATIONAL MEDICINAL PRODUCTS | |
| 5. | .1. Randomization, Blinding and Treatment Codes | 44 |
| - | 5.1.1. Procedures for Breaking Treatment Codes | |
| 3. | .2. Description and Handling of GS-9620 and Placebo to match | |
| | 5.2.2. Packaging and Labeling | |
| 5. | 3. Dosage and Administration of GS-9620 | |
| | 5.3.1. Fasting and food/liquids Requirement | |
| | CCI | |
| | 5.3.3. Storage and Handling | |
| | .4. Prior and Concomitant Medications | |
| 5. | .5. Accountability for GS-9620 | |
| | 5.5.1. Investigational Medicinal Product Return or Disposal | |
| 6. S' | TUDY PROCEDURES | 51 |
| 6. | .1. Subject Enrollment and Treatment Assignment | 51 |
| 6. | .2. Pretreatment Assessments Screening Visit (all cohorts) | 51 |
| | 6.2.2. Pre-Baseline/Day -13 Assessments (all Cohorts) | |
| | 6.2.3 Baseline/Day 1 Assessments (all Cohorts) | 54 |

| | 6.3. | Treatment Assessments (Cohorts 1 to 3) | 56 |
|---|---|---|---|
| | | 6.3.1. Treatment Assessments on Non Dosing Days 3, 5, 11, 17, 19, 25, 31, 33, 39, 45, 47, 53, 59, 61, 67, 73, 75 and 81 | |
| | | 6.3.2. Treatment Assessments on Non Dosing Days 8, 22, 36, 50, 64 and 78 | |
| | | 6.3.3. Treatment Assessments on Dosing Days 15, 29, 43, 57 and 71 | |
| | 6.4. | Treatment Assessments (Cohorts 4 to 9) | |
| | | 6.4.1. Treatment Assessments on Non Dosing Days 2, 58 and 128 | |
| | | 6.4.2. Treatment Assessments on Non Dosing Days 3, 59 and 129 | |
| | | 6.4.3. Treatment Assessments on Non Dosing Days 8, 22, 36, 50, 64, 78, 92, | |
| | | 106, 120 and 134 | 60 |
| | | 6.4.4. Treatment Assessments on Dosing Days 15, 29, 43, 57, 71, 85, 99, 113 and 127 | |
| | | 6.4.5. Treatment Assessments on Non Dosing Days 31, 45, 73, 87, 101 and 115 | |
| | | (For Cohorts 5 to 9 only) | 63 |
| | 6.5. | Post-treatment Assessments | 64 |
| | | 6.5.1. End of Study Visit (all Cohorts) | 64 |
| | | 6.5.2. Early Study Drug Discontinuation Visit (all Cohorts) | 65 |
| | 6.6. | Criteria for Discontinuation of Study Treatment | 66 |
| | CCI | | |
| | 6.8. | Prolonged Viremia | 67 |
| | | 6.8.1. Management of Prolonged Viremia | 67 |
| 7. | ADVI | ERSE EVENTS AND TOXICITY MANAGEMENT | 68 |
| | 7.1. | Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events | 68 |
| | , , , , , | 7.1.1. Adverse Events. | 68 |
| | | 7.1.2. Serious Adverse Events | |
| | | 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as | |
| | | Adverse Events or Serious Adverse Events | 69 |
| | 7.2. | Assessment of Adverse Events and Serious Adverse Events | |
| | | 7.2.1. Assessment of Causality for Study Drugs and Procedures | |
| | | 7.2.2. Assessment of Severity | |
| | 7.3. | Investigator Requirements and Instructions for Reporting Adverse Events and Serious | |
| | | Adverse Events to Gilead | 70 |
| | 7.4. | Gilead Reporting Requirements | |
| | 7.5. | Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or | |
| | | Serious Adverse Events | 72 |
| | 7.6. | Toxicity Management | |
| | | 7.6.1. Management of Dose-Limiting Toxicities (DLTs) | |
| | | 7.6.2. Management of Other Toxicities | |
| | 7.7. | Special Situations Reports | 75 |
| | | 7.7.1. Definitions of Special Situations | |
| | | 7.7.2. Instructions for Reporting Special Situations | |
| 8. | STAT | ISTICAL CONSIDERATIONS | |
| | 8.1. | Analysis Objectives and Endpoints | 79 |
| | 0.1. | 8.1.1. Analysis Objectives | |
| | | 8.1.2. Primary Endpoint | |
| | | 8.1.3. Secondary Endpoint | |
| | | 8.1.4. Other Endpoints of Interest | |
| | | 8.1.5. Exploratory Endpoints | |
| | 8.2. | Analysis Conventions. | |
| | 0.2. | 8.2.1. Analysis Sets | |
| | 8.3. | Data Handling Conventions | |
| | 8.4. | Demographic Data and Baseline Characteristics | |
| | J. r. | 2 - 1110 D. aprile Data and Date inte Characteristics | |

| | 8.5. | Efficacy | Analysis | 81 |
|---|---|---|---|---|
| | | 8.5.1. | Primary Analysis | |
| | | 8.5.2. | Secondary Analyses | |
| | 8.6. | Safety A | analysis | 81 |
| | | 8.6.1. | Extent of Exposure | 81 |
| | | 8.6.2. | Adverse Events | 81 |
| | | 8.6.3. | Laboratory Evaluations | 82 |
| | 8.7. | Pharmac | cokinetic Analysis | 82 |
| | 8.8. | Sample | Size | 83 |
| | 8.9. | Safety E | Evaluation Committee | 83 |
| | 8.10. | Analysis | s Schedule | 83 |
| 9. | RESP | ONSIBIL | ITIES | 84 |
| | 9.1. | Investig | ator Responsibilities | 84 |
| | | 9.1.1. | Good Clinical Practice. | |
| | | 9.1.2. | Institutional Review Board (IRB) Review and Approval | 84 |
| | | 9.1.3. | Informed Consent | |
| | | 9.1.4. | Confidentiality | 85 |
| | | 9.1.5. | Study Files and Retention of Records | |
| | | 9.1.6. | Case Report Forms | 86 |
| | | 9.1.7. | Investigational Medicinal Product Accountability and Return | 87 |
| | | 9.1.8. | Inspections | 87 |
| | | 9.1.9. | Protocol Compliance | 87 |
| | 9.2. | Sponsor | Responsibilities | 87 |
| | | 9.2.1. | Protocol Modifications | 87 |
| | | 9.2.2. | Study Report and Publications | 87 |
| | 9.3. | | vestigator/Sponsor Responsibilities | 88 |
| | | 9.3.1. | Payment Reporting | 88 |
| | | 9.3.2. | Access to Information for Monitoring | 88 |
| | | 9.3.3. | Access to Information for Auditing or Inspections | |
| | | 9.3.4. | Study Discontinuation | 89 |
| 10. | REFE | RENCES | | 90 |
| 11. | APPE | ENDICES . | | 92 |
| | A | . 31 1 | Investigator Signature Page | 02 |
| | | ndix 1. | | |
| | Appendix 2. | | Study Procedures Table | |
| | Appendix 3. Appendix 4. | | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities | |
| | | ndix 4.<br>ndix 5. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and | 100 |
| | Appel | iuix J. | Contraceptive Requirements | 120 |
| | Anner | ndix 6 | Definitions of Stage 3 Opportunistic Illnesses in HIV (CDC Guidelines) | |
| | | IMIA U. | | |

# LIST OF IN-TEXT TABLES

| Table 1-1. | Estimated Margins of GS-9620 Following Oral Administration at the Highest | |
|---|---|---|
| Tuole 1 1. | Anticipated Human Dose | 27 |
| Table 5-1. | Fasting and food/liquids Requirement | |
| Table 5-2. | Recommended Moderate-Fat Meal | |
| Table 5-3. | Prohibited Concomitant Medications | 49 |
| | LIST OF IN-TEXT FIGURES | |
| Figure 3-1. | High-Level Study Schema. | 38 |
| Figure 3-2. | Cohort 6 Visit Schema | |

#### PROTOCOL SYNOPSIS

Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404

| <b>Study Title:</b> | A Phase 1b. | Randomized. | Blinded. | Placebo-Controlled |
|---|---|---|---|---|

Dose-Escalation Study of the Safety and Biological Activity of GS-9620 in HIV-1 Infected, Virologically Suppressed Adults

IND Number: EudraCT Number:

Clinical Trials.gov

**Identifier:** 

122452

Not Applicable NCT02858401

**Study Centers Planned:** Multiple centers in North America

### **Objectives:**

The primary objectives are:

- To evaluate the safety and tolerability of escalating, multiple doses of GS-9620 in HIV-1 infected virologically suppressed adults on antiretroviral therapy (ART)
- To evaluate the virologic effect of GS-9620 as measured by changes in plasma HIV-1 RNA

The secondary objectives are:

- To evaluate the plasma pharmacokinetics (PK) of GS-9620
- To evaluate the pharmacodynamics (PD) of GS-9620 as measured by changes in interferon-stimulated genes (ISGs) and serum cytokines in whole blood compared to placebo
- To evaluate effects of GS-9620 on whole blood immune cell activation (T cell, B cell, NK cell)

The exploratory objectives are:





### **Study Design:**

This is a randomized, double-blinded, multi-cohort dose-escalation study with dose cohorts: Cohort 1 (1 mg Dose), Cohort 2 (2 mg Dose), Cohort 3 (4 mg Dose), Cohort 4 (6 mg Dose), Cohort 5 (8 mg Dose), Cohort 6 (three administrations of 10 mg Dose, followed by seven administrations of 12 mg Dose; SEC review of the 10mg safety data will be required prior to dose escalating to 12mg), and optional Cohort 7





For each cohort, eight subjects will be randomized in a 6:2 ratio to receive GS-9620 or placebo.

Subjects will receive a total of either 6 doses in Cohorts 1 to 3, 10 doses in Cohorts 4 to 6, CCI of their assigned study treatment administered once every other week. For all subjects in Cohort 6, Dose 4 (Day 43) will

occur after SEC review has been completed. If dose escalation is approved by the SEC, subjects in Cohort 6 will receive 12 mg of GS-9620 or placebo from Doses 4 to 10; if dose escalation is not approved by the SEC, subjects will continue receiving 10 mg of GS-9620 or placebo from Doses 4 to 10.

Enrollment will initially be opened for Cohort 1 only. A SEC will review study progress, safety and virology results of enrolled subjects. After all subjects in a cohort have received at least three doses (Cohorts 1 to 3, and 6) or five doses (Cohorts 4 and 5), the SEC will review safety data from that cohort, including adverse events (AEs) and clinical laboratory results (including plasma HIV-1 RNA) before approving the next dose escalation.

### A cohort may be suspended if

≥ 2 out of 6 subjects receiving GS-9620 experience one or more dose-limiting toxicities (DLTs) considered related to study drug.

Number of Subjects Planned:

Approximately up to 72 subjects total (6 GS-9620; 2 placebo per cohort)

Subjects who discontinue study participation before completion of dosing for reasons other than study treatment-related AEs may be replaced

Target Population:

HIV-1 infected male and non-pregnant, non-lactating female adults who have been virologically suppressed (HIV-1 RNA < 50 copies/mL) on ART for ≥ 12 consecutive months prior to screening

Main Eligibility Criteria:

- HIV-1 infection
- Aged ≥ 18 years at Pre-Baseline/Day -13
- On antiretroviral (ARV) treatment for
   ≥ 12 consecutive months prior to Pre-Baseline/Day -13
  - The following agents are allowed as part of the current ARV regimen: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc
  - The following agents are NOT allowed as part of the current ARV regimen: HIV protease inhibitors (including low dose ritonavir), cobicistat-containing regimens, elvitegravir, efavirenz, etravirine, and nevirapine

- A change in ARV regimen ≥ 45 days prior to
   Baseline/Day 1 for reasons other than virologic failure (eg, tolerability, simplification, drug-drug interaction profile) is allowed
- Plasma HIV-1 RNA < 50 copies/mL at screening
- Documented plasma HIV-1 RNA levels < 50 copies/mL (according to the local assay being used) for ≥ 12 months preceding the screening visit (measured at least twice using a licensed assay with a lower limit of quantitation of at least 40 copies/mL)
  - Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable. (If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL, the plasma HIV-1 RNA level cannot exceed 50 copies/mL on two consecutive HIV-1 RNA tests)
  - If ARV regimen is changed ≥ 45 days prior to Pre-Baseline/Day -13, plasma HIV-1 RNA <50 copies/mL at Pre-baseline/Day -13 visit is required.
- No documented history of resistance to any components of the current ARV regimen
- Availability of a fully active alternative ARV regimen, in the opinion of the Investigator, in the event of discontinuation of the current ARV regimen with development of resistance.
- Hgb  $\geq$  11.5 g/dL (males) or  $\geq$  11 g/dL (females)
- WBC  $\geq 4000 \text{ cells/}\mu\text{L}$
- Platelets  $\geq 150,000/\text{mL}$
- ANC  $\geq 1500 \text{ cells/}\mu\text{L}$
- CD4 count  $\geq$  400 cells/ $\mu$ L
- Albumin  $\geq 3.9 \text{ g/dL}$
- ALT and AST  $\leq 2 \times ULN$
- Estimated glomerular filtration rate  $\geq 60 \text{ mL/min}$
- No autoimmune disease(e.g. lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, sarcoidosis, moderate or severe psoriasis)
- No evidence of current HBV infection
  - Positive anti-HBs antibody and negative HBsAg results are acceptable

- No evidence of current HCV infection
  - Positive anti-HCV antibody and negative HCV PCR results are acceptable
- No documented history of pre-ART CD4 nadir < 200 cells/μL
  - Unknown pre-ART CD4 nadir is acceptable
- No history of Class C AIDS-Defining Condition
  - No acute febrile illness within 35 days prior to Pre-Baseline/Day -13

Study Visits and Procedures:

#### **Visit Schedule:**

The main study phase consists of a screening period of up to 35 days, a pre-treatment period of 14 Days (from Day -13 to Day 1), treatment period of 71 days (Cohorts 1 to 3), 127 days (Cohorts 4 to 6), CCI and a follow-up period of 30 days after the last dose of study drug is taken. Enrolled subjects will undergo the following scheduled study visits:

#### Cohort 1 to Cohort 3

Day -13 (Pre-Baseline)

Day 1 (Baseline/Dose 1), Day 3, Day 5, Day 8, Day 11

Day 15 (Dose 2), Day 17, Day 19, Day 22, Day 25

Day 29 (Dose 3), Day 31, Day 33, Day 36, Day 39

Day 43 (Dose 4), Day 45, Day 47, Day 50, Day 53

Day 57 (Dose 5), Day 59, Day 61, Day 64, Day 67

Day 71 (Dose 6), Day 73, Day 75, Day 78, Day 81

Day 101 (End of Study)

#### Cohort 4

Day -13 (**Pre-Baseline**)

Day 1 (Baseline/Dose 1), Day 2, Day 3, Day 8

Day 15 (Dose 2), Day 22

Day 29 (Dose 3), Day 36

Day 43 (**Dose 4**), Day 50

Day 57 (Dose 5), Day 58, Day 59, Day 64

Day 71 (Dose 6), Day 78

Day 85 (**Dose 7**), Day 92

Day 99 (Dose 8), Day 106

Day 113 (**Dose 9**), Day 120

Day 127 (Dose 10), Day 128, Day 129, Day 134

Day 157 (End of Study)

#### Cohorts 5 to 9

Day -13 (Pre-Baseline)

Day 1 (Baseline/Dose 1), Day 2, Day 3, Day 8

Day 15 (Dose 2), Day 22

Day 29 (Dose 3), Day 31, Day 36

Day 43 (Dose 4), Day 45, Day 50

Day 57 (Dose 5), Day 58, Day 59, Day 64

Day 71 (Dose 6), Day 73, Day 78

Day 85 (Dose 7), Day 87, Day 92

Day 99 (Dose 8), Day 101, Day 106

Day 113 (Dose 9), Day 115, Day 120

Day 127 (Dose 10), Day 128, Day 129, Day 134

Day 157 (End of Study)

Subjects who prematurely discontinue study drug will be required to complete an Early Study Drug Discontinuation Visit within 30 days after their last dose of study treatment.

The Pre-Baseline/Day -13 visit has an allowable window of  $\pm$  3 days.

• Visits scheduled for 2, 4, 7, or 10 days after a Dosing visit, except for Day 2, 3, 58, 59, 128 and 129 have an allowable window of  $\pm$  1 day.

The Day 101 and 157 visits have an allowable window of  $\pm$  3 days.

Non-dosing visits may occur at the investigator site or at other location agreed by the subject and mobile nurse vendor.

# **Screening Procedures:**

Screening procedures include: complete physical examination, vital signs, height, weight, medical history (including route and estimated duration of HIV infection, pre-ART viral set point, and complete ARV history), HIV-1 RNA, ARV trough PK, hematology, serum chemistry, serum pregnancy test, urinalysis, HBV and HCV serologies, eGFR, and electrocardiogram (ECG). Pre-ART CD4 nadir and historical genotype will be collected if available.

In order to establish eligibility, Investigators may repeat screening procedures or laboratory assessments for subjects who have an acute illness or abnormal laboratory value that is expected to resolve without sequelae within the screening window.

# **On-Study Procedures:**

### **Dosing:**

For Cohorts 1 to 3, dosing visits will occur at Day 1, Day 15, Day 29, Day 43, Day 57, and Day 71. For Cohorts 4 to 9, dosing visits will occur at Day 1, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 113 and Day 127.

For **Cohorts 1 to 4**, subjects will fast for at least 2 hours before dosing. For **Cohorts 5 to 8**, subjects will fast overnight (at least 8 hours) before dosing.

The Investigator will verify the subject's continued eligibility for dosing at post-Baseline dosing visits, including the absence of dose-limiting toxicities (DLTs) and (for females of childbearing potential) a negative urine pregnancy test, prior to dosing. All doses will be directly administered by blinded site staff. Subjects will fast for 2 hours after dosing for all cohorts. After Dose 1, subjects will remain on site for 12 hours after dosing for safety assessment and phlebotomy.

### **Safety:**

Solicitation of AEs and concomitant medications and symptom-directed physical examination at every visit.

Hematology, serum chemistry, and urinalysis weekly for Cohorts 1 to 3. For **Cohorts 4 to 9** these labs will be collected on dosing days, seven days post dose (starting from Dose 4), at end of study, and ESDD. For **Cohorts 6** these labs will also be collected on Day 2 and two days post dose (starting from Dose 5).

Urine pregnancy test (for females of childbearing potential) prior

to each dose.

Vital signs (blood pressure, pulse, respiration rate and temperature) at all dosing visits.

Subjects will be instructed to contact the site immediately if any flu-like symptoms are noted (eg, fatigue, pyrexia, chills, myalgia, joint pain or headache).

#### **Pharmacokinetics:**

Plasma GS-9620 concentrations will be collected at the following time points **for all cohorts:** 

- Pre-dose (≤5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 12 hours post dose at Day 1; then one sample 48 hours post dose at Day 3
- If the SEC approves the dose escalation to 12 mg in Cohort 6, starting from Dose 4 and onwards, plasma GS-9620 concentrations will also be collected on Day 43 (Dose 4): Pre-dose (≤5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 12 hours post dose; then one sample 48 hours post dose at Day 45

CCI

A single trough ARV PK sample will be collected at Pre-Baseline/Day -13 (Cohorts 1 to 3) or at Screening, Day 29, Day 57, Day 85 and Day 99 (Cohort 5), or at Screening, Day 57 and Day 99 (Cohorts 6CCI CCI

The timing of the ARV trough collection is to be 20-24 hours following the subject's previous QD regimen dose and before next ARV dose (and, for any subject on a regimen containing a BID component, the trough collection must also occur 8-12 hours following the subject's previous dose of that BID component and before next ARV dose). These samples may be analyzed to assess interim ART adherence.

### **Pharmacodynamics:**

Whole blood ISG mRNA panel: For Cohorts 1 to 3, immediately before and 2 days and 7 days after each dose of study drug, and at the end of the study (Day 101). For Cohorts 4 to 9, immediately before and 1 day, 2 days and 7 days after doses 1, 4 (only if Cohort 6 subjects receive 12 mg starting at Dose 4), 5 and 10.

TLR7 genotyping: at Pre-Baseline/Day -13

# Virology:

Plasma HIV-1 RNA: at every visit except Pre-Baseline (Day -13).

Cell-associated HIV-1 RNA/DNA (CAVR/CAVD), and plasma HIV-1 RNA by Single Copy Assay (SCA) will be collected immediately before and two days post Doses 1, 4, 6 and at end of the study (Cohort 1 to 3); immediately before and two days post Doses 1, 5, 10 and at end of the study (Cohorts 4 to 9).

HIV-1 reservoir measurements: at Pre-Baseline/Day -13 and at the end of the study (Cohorts 4 to 9).

# **Immunology:**

Peripheral blood immune cell numbers for T/B/NK/pDC/mDC including: CD4 and CD8 populations, CD4/CD8 ratio, CD4% and lymphocyte activation (T, B and NK cells) by flow cytometry will be collected immediately before and two days post Doses 1, 3, and 6 (Cohorts 1 to 3), and immediately before, one and two days post Doses 1, 5 and 10 (Cohorts 4 to 9).

FoxP3+ Treg cells by flow cytometry will be collected immediately before Doses 1, 3, and 6 (Cohorts 1 to 3), and immediately before Doses 1, 5 and 10 (Cohort 4 to 9).

Changes in the levels of antiviral cytokines and inflammatory markers by chemiluminescence: immediately before and 2 days and 7 days after each dose, and at the end of the study (Cohorts 1 to 3). For subjects in Cohorts 4 to 9, immediately before, post dose days 1, 2 and 7 after Doses 1, 4 (only if Cohort 6 subjects receive 12 mg at Dose 4), 5 and 10.

PBMC Intracellular cytokine staining (ICS) for Treg cells: immediately before and 2 days after Doses 1 and 6 for subjects in Cohorts 1 to 3.

HIV-specific T-cell responses by ELISPOT will be collected at Pre-Baseline/Day -13, immediately before Dose 6 and at the end of study for subjects in **Cohorts 1 to 3**.

For subjects in Cohorts 4 to 9, HIV-specific polyfunctional T cell Intracellular Cytokine Staining (ICS) and HIV-specific T-cell responses by ELISPOT will be collected at Pre-Baseline/Day -13 and at the end of the study.

Stool sample will be obtained for microbiome analysis. (Day 1 and Day 157 for Cohorts 5 to 9). CCI

### **Additional End of Study Procedures:**

Symptom-directed physical examination, review of AEs and concomitant medications, weight, eGFR, hematology, serum chemistry, urinalysis, urine pregnancy test (for females of childbearing potential, if not performed within the previous 30 days).

#### **Early Study Drug Discontinuation Visit Procedures:**

Symptom-directed physical examination, review of AEs and concomitant medications, weight, eGFR, HIV-1 RNA, hematology, serum chemistry, whole blood ISG mRNA panel, serum cytokine/soluble biomarker studies, urinalysis, urine pregnancy test.

#### **Procedure Definitions and Specifications:**

**HIV-1 RNA** will be performed by a licensed assay with a lower limit of quantitation of at least 20 copies/mL.

**Hematology** panel includes: complete blood count (CBC) with differential and platelets, CD4+ cell count, CD8+ cell count, CD4/CD8 ratio, and CD4%.

**Serum chemistry** panel includes: alkaline phosphatase, AST, ALT, total and direct bilirubin, total protein, albumin, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphate, magnesium, potassium, sodium, CPK, and uric acid.

Urinalysis includes dipstick. Serum and urine pregnancy tests are performed only on female subjects of childbearing potential.

Phlebotomy volume limits will be maintained in accordance with American Red Cross blood donation guidelines, which limit blood donation to 473 mL every 56 days. Subjects will undergo periodic phlebotomy over a 149-day period and will provide no more than 473 mL every 56 days. Subjects will be prohibited from blood donation in excess of that required for clinical care within 30 days prior to screening and 30 days after study ends.

# **Study Treatment:**

Investigational Medicinal Products:

GS-9620: 1 mg, 2 mg, 4 mg, 6 mg (administered as three 2 mg tablets), 8 mg (administered as two 4 mg tablets), 10 mg (administered as five 2 mg tablets), 12 mg (administered as six 2 mg tablets, or three 4 mg tablets) dose administered orally once every other week.

Reference Treatment:

Placebo-to-match GS-9620, administered orally once every other week.

**Duration of Treatment:** 

The treatment duration is 71 days (Cohorts 1 to 3), 127 days (Cohorts 4 to 6), CCI

Other Treatment:

Subjects will continue their existing ARV regimen (as currently prescribed and supplied) for the duration of study participation.

#### **Criteria for Evaluation:**

Safety:

AEs and clinical laboratory tests will be collected at every visit and summarized through Day 101 or Day 157 (30 days after the last dose of GS-9620 or placebo).

### The following are DLTs:

- ALT elevation defined as:
  - -- ALT > 10 × ULN **OR**
  - confirmed ALT elevation (i.e. grade shift or 2 × previous value) with evidence of worsened hepatic function (e.g. total bilirubin > 2 mg/dL above Baseline, serum albumin > 1 g/dL decrease from Baseline)
- A confirmed ≥ Grade 3 AE considered by the investigator to be study drug-related

- A confirmed ≥ Grade 3 lab abnormality considered by the investigator to be study drug-related and clinically significant
- A persistent (≥ 72 hours) ≥ Grade 2 flu-like symptom (eg pyrexia, fatigue, myalgia, arthralgia, headache, chills) considered by the investigator to be study drug-related
- A post-dose increase in plasma HIV-1 RNA that fails to resolve to < 50 copies/mL within 10 days in Cohorts 1 to 3
- A post-dose increase in plasma HIV-1 RNA that fails to resolve to < 200 copies/mL within 10 days in Cohorts 4 to 9

The Investigator will notify the SEC within 24 hours of any DLT. The SEC may unblind the treatment assignment for a subject experiencing a DLT.

Study drug dosing for a subject may be discontinued if the subject receives GS-9620 and experiences one or more DLTs considered to be related to study drug.

A Dose Cohort may be discontinued if  $\geq 2$  out of 6 subjects receiving GS-9620 experience one or more DLTs considered related to study drug.

#### **Statistical Methods:**

Safety:

To evaluate overall safety, the incidences of treatment-emergent AEs and treatment-emergent laboratory abnormalities will be summarized by treatment group.

The proportion of subjects in each treatment group with an AE leading to premature discontinuation of study drug and proportion of subjects with serious adverse events (SAEs) will be summarized by treatment group.

Virology:

The change in plasma HIV-1 RNA and the incidence of detectable plasma HIV-1 RNA at each visit will be summarized by treatment group.

The change in plasma HIV-1 RNA SCA from pre-dose to 2 days post-dose may be explored.

The change in cell (PBMC) associated HIV-1 RNA from pre-dose to 2 days post-dose may be explored.

The change in HIV-1 reservoir measured by cell (PBMC) associated HIV-1 DNA from pre-dose to 2 days post-dose, and in Cohorts 4 to 9 by use of secondary assays using stored PBMC samples may be explored

| PK: Exposure parameters of GS-9620 will be summarized using |
|-------------------------------------------------------------|
|-------------------------------------------------------------|

descriptive statistics by active treatment.

PD: The change from baseline in the levels of serum cytokines will be

summarized using descriptive statistics by treatment group. The post-baseline change and fold induction in mRNA for ISGs will be summarized using descriptive statistics by treatment group.

Immunology: The post-baseline change in peripheral blood immune cell

numbers for T/B/NK/pDC/mDC including: CD4 and CD8 populations, CD4/CD8 ratio, CD4 % and lymphocyte activation (T, B and NK cells) will be summarized using descriptive

statistics by treatment group.

The post-baseline change in magnitude and poly-functionality (Cohorts 4 to 9) of the HIV-1-specific T cell immune response

may be explored.

TLR7 genotype may be reported and its association with key pharmacodynamic and virologic parameters may be explored.

Sample Size: This is an exploratory study to characterize the safety and efficacy

of GS-9620; therefore, no power calculation was performed. Sample size is determined based on empirical considerations. A total of up to 54 subjects (6 per cohort) receiving GS-9620 will

provide a reasonable preliminary assessment of safety.

This study will be conducted in accordance with the guidelines of Good Clinical Practice (GCP) including archiving of essential documents.

### GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

°C degree(s) Celsius
°F degree(s) Fahrenheit

ACTG AIDS Clinical Trials Group

AE adverse event

AIDS Acquired Immune Deficiency Syndrome

ALT alanine aminotransferase (SGPT)

ANOVA analysis of variance ART antiretroviral therapy

AST aspartate aminotransferase (SGOT)
ATI analytical treatment interruption

AUC<sub>0-t</sub> area under the plasma concentration-time curve from zero
AUC<sub>24h</sub> area under the plasma concentration-time curve in 24 hours

AUC<sub>tau</sub> area under the plasma concentration versus time curve over the dosing

interval (tau)

BID bis in die (two-or twice-a-day)
BLQ below the limit of quantitation

BUN blood urea nitrogen

CAVR/CAVD Cell-associated HIV-1 RNA/DNA

CBC complete blood count

CDC Center for Disease Control and Prevention
CFR Code of Federal Regulations (United States)

C<sub>last</sub> last observed quantifiable concentration of the drug

CL<sub>cr</sub> creatinine clearance

C<sub>max</sub> maximum observed concentration of drug

CNS central nervous system

CPK creatine phosphokinase (= creatine kinase, CK)

CSR clinical study report

C<sub>tau</sub> observed drug concentration at the end of the dosing interval (tau)

CYP3A cytochrome P450

dL deciliter(s)

DLT dose-limiting toxicities
DNA deoxyribonucleic acid

DTG dolutegravir EC ethics committee

EC<sub>50</sub> 50% effective inhibitory concentration

ECG Electrocardiogram
EDC Electronic data capture

eCRF electronic case report form(s)

eGFR estimated glomerular filtration rate **ESDD** Early Study Drug Discontinuation

**EudraCT** European Union Drug Regulating Authorities Clinical Trials

**FDA** Food and Drug Administration (United States)

**FSH** Follicle stimulating hormone

**FTC** emtricitabine ET early termination

G Gram

**GCP** Good Clinical Practice (Guidelines)

gamma-glutamyl transferase (= gamma-glutamyl transpeptidase, GGTP) **GGT** 

Gilead Sciences, Inc. GSI **HBV** hepatitis B virus HCV hepatitis C virus

hepatitis B virus surface antigen **HBsAg** 

HLT high level term

**HLGT** high level group term **HPF** high-power field

HIV human immunodeficiency virus

Hour hr

**ICH** International Conference on Harmonization

**ICS** intracellular cytokine staining  $IC_{50}$ 50% inhibitory concentration **Institutional Ethics Committee IEC** 

**IFN** Interferon interferon-alpha IFN-α

IND Investigational New Drug (Application) IP-10 interferon γ-inducible protein-10 IRB Institutional Review Board

**ISGs** interferon-inducible genes **IUD** intrauterine device IU

Kilogram kg

lower limit of the normal range LLN

lower limit of detection LLOD

LLT lower level term

LRA latency reversal agents MAD multiple ascending dose

MedDRA Medical Dictionary for Regulatory Activities; MedDRA®

international unit

Milligram mg Microgram μg

Protocol GS-US-382-1450 Final Gilead Sciences, Inc. Amendment 7

min Minute

mDC conventional (myeloid) dendritic cell

mL Milliliter

mRNA messenger ribonucleic acid

NK natural killer (cell)
NDA New Drug Application

NOAEL no observed adverse effect level

NRTI Nucleoside Reverse-Transcriptase Inhibitors

PEG pegylated interferon

PBMC peripheral blood mononucleated cell

PCR polymerase chain reaction
PD pharmacodynamics(s)
pDC plasmacytoid dendritic cell

PK pharmacokinetic(s)
POC Proof of concept
PT prothrombin time
PT preferred term

PVE Pharmacovigilance and Epidemiology, Gilead Sciences

PXR pregnane X receptor

QD quaque die (one- or once-a-day)

QOD every other day (dosing)

qPCR quantitative PCR
RBC red blood cell (count)
RNA ribonucleic acid
SAD single ascending dose

SADR serious adverse drug reaction

SAE serious adverse event SCA single copy assay SD standard deviation

SEC Safety Evaluation Committee
SIV Simian immunodeficiency virus

SOC System Organ Class

SUSAR Suspected Unexpected Serious Adverse Reaction

 $T_{1/2}$  estimate of the terminal elimination half-life of the drug, calculated by

dividing the natural log of 2 by the terminal elimination rate constant  $(\lambda_z)$ 

Th1/Th2/Th17 T helper cells (1, 2, 17)
Tr1 Type 1 T regulatory cells

 $T_{last} \hspace{1cm} time \hspace{1cm} (observed \hspace{1cm} time \hspace{1cm} point) \hspace{1cm} of \hspace{1cm} C_{last}$   $T_{max} \hspace{1cm} time \hspace{1cm} (observed \hspace{1cm} time \hspace{1cm} point) \hspace{1cm} of \hspace{1cm} C_{max}$ 

 $T_{reg}$  T regulatory (cells)

TFV tenofovir

TLR toll-like receptor

ULN upper limit of the normal range

US United States

USA United States of America

vs versus

WHO World Health Organization

wt weight

 $\lambda_z$  terminal elimination rate constant, estimated by linear regression of the

terminal elimination phase of the concentration of drug versus time curve

### 1. INTRODUCTION

# 1.1. Background

Human immunodeficiency virus type-1 (HIV-1) infection is a life-threatening and serious disease that is of major public health interest around the world. There are approximately 2.4 million people in North America and Western and Central Europe living with HIV-1 and 36 million people worldwide {Joint United Nations Programme on HIV/AIDS (UNAIDS) 2016}. Untreated infection leads to deterioration in immune function and death. The availability of antiretroviral therapy (ART) has been associated with a dramatic decrease in acquired immune deficiency syndrome (AIDS)-related morbidity and mortality {Mocroft 1998, Palella 1998, Sterne 2005}.

While ART effectively suppresses HIV replication, HIV infection remains incurable. Persistent viral reservoirs fuel rebound viremia when treatment ceases. Despite the availability of chronic treatment, morbidity and mortality due to HIV infection remain high due to the latent HIV reservoir, which may contribute to ongoing inflammation-driven disease. Current therapy is associated with challenges with tolerability, long-term adherence and safety, drug-drug interactions, and expense. Persistent HIV infection may also be associated with psychosocial stigma. Thus, the discovery and development of therapeutic interventions that can eradicate or control HIV reservoirs, leading to long-term ART-free remission or HIV cure, is a major priority.

Following entry into a target cell, HIV-1 stably integrates into the host genome, thus establishing the basis for latent infection and the main barrier to HIV cure. Neither the host immune system nor ART can eliminate transcriptionally inactive virus. Therefore, adjunctive therapies that efficiently reactivate ("kick") virus out of this latent reservoir to enable its destruction ("kill") may be required for viral eradication. This "kick and kill" strategy to cure or induce long-term HIV remission has been tested in clinical trials of latency reversal agents (LRA) such as histone deacetylase inhibitors (HDACi). While short-term treatment with HDACi such as romidepsin appears to be safe and may activate viral transcription in individuals virologically suppressed on ART, the size of the latent viral reservoir as measured by total peripheral blood mononuclear cell (PBMC)-associated HIV-1 DNA or quantitative viral outgrowth assay (QVOA) appears to be unchanged (Sogaard 2015). However, a TLR9 agonist has been dosed in HIV-1 positive participants on ART in a single-arm open-label study demonstrating increases in plasma IFN-α levels, transcriptional (messenger ribonucleic acid [mRNA] induction of interferon stimulated genes (ISGs), activation of pDCs, activation of cytotoxic natural killer (NK) and CD8+ T cells with transient increases in plasma HIV-1 RNA in a subset of individuals {Vibholm 2017}. It is postulated that a combination of therapies exerting viral latency reversing activity and engagement of the host immune system will be necessary to have a demonstrable effect on reducing the HIV-1 reservoir. To date there is no fully validated biomarker for the latent HIV-1 reservoir. Therefore, measurement of the time to viral rebound and/or new viral load set-points following analytical treatment interruption (ATI) is the most accurate endpoint to evaluate the efficacy of "kick and kill" interventions. The AIDS Clinical Trials Group (ACTG) has reported that ATI can be conducted safely in patients {Bar 2016, Li 2016} and that certain measures of the HIV reservoir may be correlated with time to viral rebound {Li 2016}.

GS-9620 is an orally-administered toll-like receptor (TLR) 7 agonist currently in clinical development for the treatment of HIV. In vitro, GS-9620 appears to mediate both HIV-1 "kick" and "kill" activity. In a rhesus macaque model of chronic SIV infection, treatment with GS-9620 or its close analog GS-436986 has also demonstrated the ability to both "kick" and "kill": treatment resulted in transient detection of plasma viremia within 24-72 hours of dosing, decreases in ex vivo SIV production from T-cell receptor stimulated PBMC cultures or immune cell isolates of peripheral lymph nodes comparing pre-treatment to post-dosing samples and a ~0.5 log<sub>10</sub> lower viral load set-point after discontinuation of ART {Lim 2018}. Most importantly, in a subset of animals, there was a lack of detectable plasma virus (< 50 SIV RNA copies/mL) for > 2 years after discontinuation of ART. During the off ART phase, two animals from one of the studies had no viral rebound after administration of antibodies depleting NK and CD8+ lymphocytes or transfer of viral infection after infusion of mononuclear immune cells from lymph node and peripheral blood into naïve animals; implying a substantial reduction in viral reservoir. The administration of multiple doses of GS-9620 has been shown to be safe in clinical studies of healthy subjects (single doses up to 12 mg), and hepatitis B virus (HBV)-infected subjects (multiple doses up to 4 mg). This study will therefore investigate the safety and efficacy of GS-9620 in HIV-infected individuals who are virologically suppressed on ART.

#### 1.2. GS-9620

#### 1.2.1. General Information

GS-9620 is an orally-administered TLR7 agonist in development for the treatment of HIV infection.

Data in-vitro have shown that GS-9620 is a potent and selective TLR7 receptor agonist with a > 30-fold selectivity for TLR7 (32-fold based on EC<sub>50</sub> and 81-fold based on minimum effective concentration) over toll-like receptor 8 (TLR8), with no detectable stimulation of other human TLRs at concentrations up to 100  $\mu$ M (PC-243-2031).

Nonclinical data in mice and in chimpanzees chronically infected with HBV demonstrated that oral administration of GS-9620 induce a type I IFN dependent innate response in the liver, as measured by induction of interferon-stimulated genes (ISGs), in the absence of concomitant serum detectable levels of IFN- $\alpha$  (i.e. a pre-systemic response) {Fosdick 2013, Lanford 2013}. The induction of type I IFN-dependent innate immune responses without the induction of detectable systemic IFN- $\alpha$  has been confirmed in healthy human subjects (GS-US-320-0101) and patients affected by chronic hepatitis C (GS-US-243-0102) or by chronic hepatitis B (GS-US-283-0102, GS-US-283-0106, GS-US-283-1059, and GS-US-283-1062).

For further information on GS-9620, refer to the investigator's brochure for GS-9620.

# 1.2.2. Preclinical Pharmacology and Toxicology

Preclinical in vivo pharmacology studies in different non-human primate species have consistently demonstrated that GS-9620 induces IFN-α, multiple cytokines, chemokines, peripheral blood mononuclear cell (PBMC) derived ISG mRNAs and peripheral immune cell activation in a dose-dependent manner. Of note, with escalating doses of GS-9620 cynomolgus monkeys were shown to have an exaggerated IFN-α response both in vitro and in vivo compared to other species (mice, chimpanzees, and humans).

In in vitro PBMC cultures, GS-9620 stimulated markedly higher maximal levels of secreted IFN- $\alpha$  in cynomolgus monkey PBMC compared to human PBMC cultures; the in vitro mean peak IFN- $\alpha$  was 9105 pg/mL and 1552 pg/mL in cynomolgus monkey and human PBMCs, respectively.

Similarly, the mean peak IFN-α concentration in serum following a single oral dose in vivo was notably higher in cynomolgus monkeys than healthy human volunteers at an equivalent dose; at 0.5 mg/kg (human equivalent dose 9.6 mg) the mean peak of serum IFN-α was 4859 pg/mL in cynomolgus monkey versus 93.7 pg/mL in human healthy volunteers receiving 12 mg dose [study GS-US-243-0101] (human equivalent dose was calculated using a conversion factor of 0.32 for cynomolgus monkey and assuming a human body weight of 60 kg {U. S. Department of Health and Human Services (DHHS) 2005}).

Single oral doses of GS-9620 given in preclinical studies in cynomolgus monkeys (0.05 to 0.5 mg/kg, human equivalent dose 1-9.6 mg) and mice (0.3 mg/kg, human equivalent dose 1.4 mg) human equivalent dose was calculated using a conversion factor of 0.08 for mice and assuming a human body weight of 60 kg {U. S. Department of Health and Human Services (DHHS) 2005}) have shown that GS-9620 can induce an innate immunity gene expression signature, e.g. up-regulation of interferon-stimulated genes (ISG) in the absence of detectable serum IFN- $\alpha$  concentrations. These observations are consistent with the concept of a pre-systemic response elicited by oral GS-9620.

Body temperature increases were noted in the cardiovascular/respiratory safety pharmacology study in cynomolgus monkeys ( $\geq 0.5$  mg/kg) at  $C_{max}$  exposures that were approximately equivalent to the  $C_{max}$  at the highest dose tested in HBV infected patients (4 mg; study GS-US-283-0102). Increases in heart rate were observed concurrently with the increases in body temperature and with the peak of IFN- $\alpha$  levels. Of note, body temperature and heart rate increase were not seen at the 4-mg dose in the human clinical studies. Increases in body temperature and heart rate are well-described side effects of exogenous IFN- $\alpha$  administration in humans {Vial 1994} and in nonhuman primates {Kubicek 1958, Vial 1994} and may reflect the sequelae of elevated IFN- $\alpha$  in the cynomolgus monkeys.

In an in vitro electrophysiology assay GS-9620 inhibited the human ether-à-go-go-related gene (hERG)-mediated current at an IC $_{50}$  (50% inhibitory concentration) value that was 150-fold higher than the  $C_{max}$  at the highest dose used in HBV infected patients (4 mg; study GS-US-283-0102). These margins are likely even higher once adjusted for protein binding.

No adverse cardiovascular effects were noted in cynomolgus monkeys at  $C_{max}$  exposures up to 1.7-fold higher than projected  $C_{max}$  (11.97 ng/mL) for a 12 mg dose of GS-9620, the highest dose planned to be used in this clinical study. No notable effects on the central nervous or respiratory systems were seen in the safety pharmacology studies. Safety pharmacology studies did not identify any major effects that would impede the use of GS-9620 in human subjects.

Preclinical toxicology studies were conducted in single dose and multiple dose settings in different animal species.

### **Single Dose Toxicology Studies**

Single oral doses of GS-9620 were well tolerated at up to 30 mg/kg and up to 2 mg/kg in mice and cynomolgus monkeys, respectively. At higher doses, mortality was noted in single dose oral studies in mice at 100 mg/kg (TX-243-2008) or greater (AD-243-2017) and in a single woodchuck administered 10 mg/kg orally (AD-243-2014). Additionally, mortality was observed following intravenous administration of 3 mg/kg to rhesus monkeys (AD-243-2034). These deaths were attributed to high systemic exposure to GS-9620 ( $\geq$  21-fold higher than the AUC<sub>0-24</sub> in HBV infected patients [study GS-US-283-0102]; 44.3 pg•h/mL at 4 mg).

## **Multiple Dose Toxicology Studies**

Oral administration of GS-9620 every-other-day (QOD) was well tolerated in the 4-week and 6-week studies in mice, with the highest doses of 5 and 3 mg/kg QOD, respectively, being the no observed adverse effect levels (NOAELs) (Table 1-1).

In cynomolgus monkeys, GS-9620 was well tolerated in the 4-week study with the highest dose of 1.5 mg/kg QOD being the NOAEL (Table 1-1).

In the 26-week cynomolgus monkey toxicity study, GS-9620 administration at ≤ 0.15 mg/kg/dose was well tolerated. Administration of 0.50 mg/kg every other day (reduced to 0.3 mg/kg every other day at Week 11) resulted in morbidity/mortality of 3 animals beyond 8 weeks of QOD dosing. In this study the pharmacodynamic effects appeared to increase over time and were associated with high levels of circulating IFN-α. Cynomolgus monkeys were the most sensitive toxicology species and have an apparent exaggerated IFN-α response to GS-9620 (Table 1-1). The observed mortalities in cynomolgus monkeys are consistent with data obtained from the New Drug Application (NDA) approvals of peginterferon alpha 2a (Pegasys®) and peginterferon alpha 2b (Peg-Intron®) showing that repeated high doses of IFN-α or PEG cause a similar spectrum of effects in cynomolgus monkeys as those observed in the 26-week toxicology study with GS-9620 {European Medicines Agency (EMA) 2006, Pilaro 2000}. The margins of exposure in the preclinical species, based on IFN-α stimulation, range from 0.33 to 122-fold depending on the duration of exposure due to GS-9620 dosing every other day. Less frequent administration, once every other week, in the clinical setting would be expected to minimize chronic IFN-α exposure side-effects.

Table 1-1. Estimated Margins of GS-9620 Following Oral Administration at the Highest Anticipated Human Dose

| | | | | | Mean | Margin of Exposure | | |
|---|---|---|---|---|---|---|---|---|
| Species | Duration | Dose<br>(mg/kg/dose) | AUC <sub>0-tau</sub> a<br>ng•h/mL | C <sub>max</sub> <sup>a</sup><br>ng/mL | Peak<br>IFN-α<br>pg/mL | AUCinf <sup>b</sup> | C <sub>max</sub> <sup>b</sup> | IFN-α <sup>c</sup> |
| Mouse | QOD x 4 weeks | 5<br>(NOAEL) | 43.5 | 13.4 | 237 | 0.3x | 1.1x | 2.4x |
| Mouse | QOD x 26 weeks | 3<br>(NOAEL) | 15.8 | 6.64 | 60.7 | 0.1x | 0.6x | 0.6x |
| | QOD x 4 weeks | 1.5<br>(NOAEL) | 73.8 | 86.7 | 11900 | 0.5x | 7.2x | 122x |
| Cynomolgus<br>Monkey | QOD x 26 weeks | 0.15<br>(NOAEL) | 0.171 | 0.077 | 32 | 0.001x | 0.006x | 0.33 |
| | - | 0.5/0.3 | 1.82 <sup>d</sup> | 0.504 <sup>d</sup> | 2085 <sup>d</sup> | 0.013x | 0.04x | 21x |

- a Males and females combined, Week 4 or Week 26 as applicable
- b Margins of exposure were calculated using clinical GS-9620 C<sub>max</sub> and AUC<sub>inf</sub> at 12 mg of 12.0 ng/mL and 140 ng•h/mL, respectively (GS-US-243-0101)
- c Margins of exposure were calculated using the mean peak for IFN-α (97.3 pg/mL) from healthy subjects dosed with 12 mg GS-9620 (GS-US-243-0101)
- d Week 17 at 0.3 mg/kg

Source: Studies TX-243-2005, TX-243-2011, TX-243-2004, TX-243-2012

# **Monotherapy Proof-of-Concept Studies in Monkeys**

In a rhesus macaque model of chronic SIV infection, treatment with GS-9620 or its close analog GS-436986 has also demonstrated the ability to both "kick" and "kill". Treatment resulted in transient detection of plasma viremia within 24-72 hours of dosing, decreases in ex vivo SIV production from T-cell receptor stimulated PBMC cultures or immune cell isolates of peripheral lymph nodes comparing pre-treatment to post-dosing samples and a ~0.5 log<sub>10</sub> lower viral load set-point after discontinuation of ART {Lim 2018}. Most importantly, in a subset of animals, there was a lack of detectable plasma virus (< 50 SIV RNA copies/mL) for > 2 years after discontinuation of ART. During the off ART phase two animals from one of the studies had no viral rebound after administration of antibodies depleting NK and CD8+ lymphocytes or transfer of viral infection after infusion of mononuclear immune cells from lymph node and peripheral blood into naïve animals; implying a substantial reduction in viral reservoir.

#### 1.2.3. Clinical Trials of GS-9620

As of 27 March 2018, 4 Phase 1 clinical studies, 1 Phase 2 clinical study, and 1 registry study have been completed in which 55 healthy subjects, 42 HCV infected subjects, and 230 subjects with chronic hepatitis B (CHB) (189 virologically suppressed and 41 treatment naive subjects) were dosed with GS-9620. In addition, a Phase 2 clinical trial (GS-US-283-1059) in virologically suppressed CHB subjects has completed dosing and a Phase 1 clinical trial (GS-US-382-3961) in HIV-1 infected controllers on ART is currently on-going. In these studies, single doses ranged from 0.3 mg to 12 mg in healthy volunteers, and from 0.3 mg to 4 mg in HCV- and HBV-infected subjects. Multiple doses (two doses one week apart and up to 12 doses one week apart) were assessed in HCV-infected and HBV-infected subjects and ranged from 0.3 mg to 4 mg.

In HIV-infected subjects, multiple doses of GS-9620 ranging from 1 mg to 6 mg were assessed, with the 8 mg dosing cohort currently in progress.

#### 1.2.3.1. GS-US-243-0101

Study GS-US-243-0101 was a first-in-human, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study of GS-9620 in 75 healthy male and female subjects. The primary objective of the study was to evaluate the safety and tolerability of GS-9620 and the secondary objectives were to characterize the plasma PK/PD profile of GS-9620. Doses used were: 0.3, 1, 2, 4, 6, 8, and 12 mg.

The treatment was generally well tolerated. There were no Grade 4 AEs or serious adverse events (SAEs) reported, and most AEs were mild. No individual subject discontinued due to AEs or laboratory abnormalities. Treatment-emergent Grade 3 AEs included pyrexia in 2 subjects who received GS-9620 12 mg. A higher incidence of flu-like symptoms was also reported in subjects administered the higher doses (8 and 12 mg). Myalgia and headache were reported by subjects in both the 8 and 12 mg cohorts, while pyrexia and chills were only reported by subjects in the 12 mg cohort.

Plasma concentrations of GS-9620 peaked between 1.5 and 6 hours after dosing and declined gradually over 48 hours. The mean maximum plasma concentration ( $C_{max}$ ) ranged from 184.2 pg/mL at the 0.3 mg dose to 11.97 ng/mL at the 12 mg dose. Exposures were higher in the fasted state than in the fed state. After the 1 mg, 2 mg, and 4 mg doses, GS-9620 was detectable at 48 hours after dosing and had a median terminal half-life between 17.16 and 26.96 hours.

Three ISGs were analyzed: ISG15, MX-1 and OAS-1. Significant ISG induction was observed at the 2-mg dose and above. ISG15 mRNA expression showed the highest induction compared to MX-1 and OAS-1. Serum IFN- $\alpha$  was detected transiently in subjects who received the 8 or 12 mg doses, and only the 12 mg cohort had a >2-fold mean change in serum IFN- $\alpha$  from baseline. A dose-dependent induction was observed for serum IP-10 but not for IFN- $\alpha$  or TNF- $\alpha$ . Dose-dependent T cell activation was also observed at the 2 mg dose and above.

In summary, single doses of GS-9620 up to 12 mg were well tolerated, with significant ISG induction and T cell activation at doses of 2, 4, and 6 mg in the absence of detectable serum IFN- $\alpha$  or systemic AEs.

#### 1.2.3.2. Other Phase 1 studies

The following studies have also demonstrated good tolerability of GS-9620 (see IB for details):

- GS-US-243-0102: A Phase 1b ascending, single and multiple-dose study evaluating the safety, PK, PD, and antiviral activity in treatment-naive HCV subjects.
- GS-US-283-0102: A Phase 1b ascending, single and multiple-dose study evaluating the safety, PK/PD, and antiviral activity in virologically-suppressed HBV subjects.

- GS-US-283-0106: A Phase 1b ascending, single and multiple-dose study evaluating the safety, PK/PD, and antiviral activity in treatment-naive HBV subjects.
- GS-US-283-0110: An observational registry study of subjects who did not achieve loss of HBsAg and sustained HBV viral load reduction below the level of quantitation in Gilead-Sponsored trials of GS-9620 in subjects with chronic HBV infection.

#### 1.2.3.3. GS-US-283-1059

GS-US-283-1059 was a Phase 2, randomized, double-blind, placebo-controlled multi-center study to evaluate the safety and efficacy of GS-9620 in HBV-infected subjects who are virologically suppressed. In this study, approximately 162 subjects received weekly dosing with GS-9620 (1, 2 or 4 mg) or placebo for a total of 4 (Cohort A), 8 (Cohort B) or 12 (Cohort C) weeks. The efficacy of GS-9620 was evaluated by assessing the change from baseline to Week 24 in HBsAg levels. Overall, once-weekly dosing of GS-9620 1, 2, or 4 mg for 4, 8, or 12 weeks was generally well tolerated in virologically-suppressed subjects with CHB on OAV. Most subjects had Grade 1 (mild) AEs and, except for the Cohort C 4 mg group in which a higher proportion of subjects had Grade 2 (moderate) and 3 (severe) AEs compared with Cohorts A and B. No other dose-related or treatment duration-related safety findings were observed. No Grade 4 (life threatening) AEs were reported in any of the cohorts. Four subjects had SAEs, 3 of these subjects had AEs that led to discontinuation of study drug, and 3 of the 4 subjects had study drug interrupted due to AEs. No deaths occurred in any study participant.

Two subjects interrupted study treatment after having experienced SAEs due to an overdose caused by a dispensing error at the study site. One of these subjects randomized to 2 mg GS-9620 mistakenly received 10 mg and one subject randomized to 4 mg mistakenly received 20 mg. These 2 subjects experienced transient Grade 3 AEs of flu-like symptoms, and decline in lymphocytes count; the subject who received 10 mg experienced Grade 3 AEs of pyrexia, chills and hot flush, all SAEs that were assessed as related to study drug by the investigator. The subject who received 20 mg experienced SAEs of Grade 3 AE of tremor and Grade 2 hypotension requiring hospitalization. This subject also experienced additional Grade 2 AEs of abdominal pain, diarrhea, and vomiting, and an increase in ALT value. For both subjects, each of the AEs resolved within 24 hours after overdose. A meeting of the Data Monitoring Committee reviewed these events and determined them to be due to the overdose of GS-9620 with expected effects of interferon-alpha induction and cytokine release and allowed for the study to proceed as planned. The other two subjects with SAEs were in Cohort C (cataract, which was reported in one subject with a medical history of cataract, and cholecystitis, which was reported in the other subject). The subject who experienced cholecystitis also withdrew from study drug and the study.

Most AEs reported were Grade 1 or Grade 2 in severity. No Grade 4 (life threatening) AEs occurred in any of the cohorts. For Cohort A, 1 subject in each group had Grade 3 AEs. None of the Grade 3 AEs led to withdrawal from study drug and none occurred in more than 1 subject. All of the Grade 3 AEs resolved. Excluding the 2 overdosed subjects discussed above, 2 subjects (placebo and GS-9620 1 mg) experienced transient Grade 3 AE of anxiety and diarrhea, respectively, during the treatment period with GS-9620/placebo; both AEs resolved within

24 hours. For Cohort B, no subjects had Grade 3 AEs. For Cohort C, 6 subjects had Grade 3 AEs: 2 subjects in the GS-9620 1 mg group, 1 subject in the GS-9620 2 mg group, 2 subjects in the GS-9620 4 mg group, and 1 subject in the placebo group. Two subjects, both in the GS-9620 4 mg group, with Grade 3 AEs (cholecystitis [discussed above] and panic attack) withdrew from the study and study drug.

Overall, patients from both the GS-9620-treated and placebo groups experienced a similar number of treatment emergent AEs (TEAEs) (68% study drug vs. 70% placebo). Upon assessment of relation to study drug, 37% of patients treated with GS-9620 reported at least one AE compared to 50% of placebo patients, all of which were mild to moderate in severity. No dose-dependency for AEs was observed across cohorts. The most commonly reported related AEs (for ≥2 or more patients) in Cohort A were fatigue (4 of 16 [25.0%] subjects) and diarrhea, headache, oropharyngeal pain, pruritus, and pyrexia (each of which occurred in 2 of 16 patients [12.5%]) (1-mg group); headache (4 of 15 [26.7%] subjects), fatigue (3 of 15 [20.0%] patients) and chills (2 of 15 [13.3%] patients) (2-mg group); and fatigue and pyrexia (each in 3 of 16 [18.8%] patients) and headache (2 of 16 [12.5%] patients) (4-mg group). In Cohort B, headache (6 of 18 [33.3%] patients), nausea (3 of 18 [16.7%] patients) and acne, dizziness, fatigue, insomnia, and oropharyngeal pain (each in 2 of 18 [11.1%] patients) (1-mg group); headache and dizziness (each in 2 of 17 [11.8%] patients) (2-mg group); and headache (4 of 17 [23.5%] patients) and fatigue, influenza-like illness, and rhinorrhea (each in 2 of 17 [11.8%] patients) (4-mg group) were most common. In Cohort C, headache, fatigue, influenza-like illness (each in 4 of 16 [25.0%] patients) and asthenia, pyrexia and somnolence (each in 2 of 16 [12.5%] patients) (1-mg group); abdominal pain upper and headache (each in 3 of 17 [17.6%] patients) and fatigue (2 of 17 [11.8%] patients) (2-mg group); and asthenia (5 of 14 [35.7%] patients), headache, influenza-like illness, and pyrexia (each in 3 of 14 [21.4%] patients) and myalgia (2 of 14 [14.3%] patients) (4-mg group). Headache was the most commonly reported placebo group AE (40-50% of patients).

Among the patients dosed with GS-9620, treatment-emergent graded ALT elevations were seen in 5 subjects (4 subjects with Grade 1 and one subject with Grade 2). All grade 1 elevations were transient (1 placebo, 1 GS-9620 2 mg, and 2 GS-9620 4 mg) and the grade 2 elevation occurred 22 days after the last dose of GS-9620 4 mg and reduced to grade 1 elevation 3 days later.

Please refer to the current GS-9620 Investigator's Brochure for the treatment of chronic hepatitis B virus infection for additional information regarding the above studies.

#### 1.2.3.4. GS-US-283-1062

This Phase 2, randomized, double-blind, placebo-controlled study is being conducted to evaluate the safety and efficacy of administering either 1 mg, 2 mg or 4 mg of GS-9620 orally once a week (every 7 days) for 12 doses (Weeks 0-11) in adult subjects with CHB who were not currently on treatment for CHB. 192 subjects were randomized in a 1:2:2:2 ratio to 1 of the 4 treatment arms (placebo, GS-9620 1 mg, 2 mg, or 4 mg) for weekly dosing for a total of 12 doses and stratified by HBeAg status (positive versus negative) and ALT (> versus  $\leq$  19 IU/mL for female; > versus  $\leq$  30 IU/mL for male). All subjects were also treated with TDF 300 mg oral daily for 48 weeks.

Preliminary interim safety results from Week 48 show that overall, once-weekly dosing of GS-9620 1, 2, or 4 mg was generally well tolerated. 65% of subjects overall had at least 1 AE during the study and most of the reported AEs were Grade 1 (mild) or 2 (moderate) in severity. Overall, the majority of subjects had Grade 1 (mild) or moderate (Grade 2) AEs. Six subjects experienced Grade 3 (severe) AEs. No Grade 4 (life threatening) AEs were reported in any of the treatment groups.

Four subjects had treatment-emergent SAEs: an SAE of laceration (deep laceration on the right foot) on Day 133 which resolved on Day 252, an SAE of asthma (worsening of asthma) on Day 257 which resolved on Day 288, an SAE of breast cancer on Day 422 continuing at the time of the interim data cut, and an SAE of abdominal pain (exacerbation of chronic generalized abdominal pain) on Day 71 which resolved on Day 85. All SAEs were considered by the investigator to be unrelated to study drugs or to study procedures. No action was taken with study drugs, with the exception of TDF dose interruption for the abdominal pain case and dose withdrawn for the breast cancer case. No deaths occurred.

Six subjects overall (3.1%) discontinued study drug due to an AE, all of which were considered related to study drugs by the investigator.

Across the treatment groups, most laboratory abnormalities were Grade 1 or 2 in severity. Five subjects had ALT  $\geq$  10x ULN and thirty had ALT between 3x ULN and < 10x ULN and > 2x nadir.

#### 1.2.3.5. GS-US-382-3961

This ongoing Phase 1b, randomized, double-blind, placebo-controlled study is being conducted to evaluate the safety and efficacy of GS-9620 in antiretroviral treated HIV-1 infected controllers. The study is conducted in two periods. In Period 1, up to 30 subjects will be randomized 2:1 to receive GS-9620 or placebo-to-match. All subjects will receive up to 10 doses of their assigned study treatment administered orally every 14 days. Subjects will continue to take their prescribed ART during Period 1. In Period 2, all subjects will discontinue ART and be monitored for rebound in HIV-1 plasma viremia. Enrollment is ongoing and several subjects have completed dosing (4-6 mg) and are undergoing ART interruption (Period 2).

# 1.3. Rationale for This Study

Despite the extensive advances made in the treatment of chronic HIV-1 infection, eradication of the latent HIV-1 reservoir is still needed to achieve a cure that abrogates the requirement for lifelong ART. To this end, "kick and kill" strategies to reactivate and target latent virus have been tested in a number of clinical trials, but none have resulted in lasting virologic remission. GS-9620 is a promising candidate for this approach given the demonstration of both SIV reactivation (as measured by transient plasma viremia in the presence of ART), decrease in SIV reservoir (as measured by proviral DNA in PBMCs, lymph node and colon), and ~0.5 log reduction in SIV set point relative to pre-ART plasma viral load set point following ART interruption in studies of SIV-infected rhesus macaques treated with GS-436986, a close analog of GS-9620. In a second study in SIV-infected rhesus on ART the TLR7 agonists GS-9620 or GS-436986 administered for 10 or 19 doses produced transient plasma viremia within

24-72 hours after dosing. Sampling PBMCs and immune cell isolates from lymph node biopsies prior to TLR7 agonist administration and after completing all doses demonstrated a decrease in the amount of SIV production following T-cell receptor stimulation. Interestingly, two of these animals, one from the GS-9620 dosing group and one from the GS-436986 dosing group had no detectable ex vivo SIV production from both PBMCs and isolated immune cells from lymph node biopsies. Most importantly, after ART discontinuation these same two animals had no detectable plasma virus (< 50 SIV RNA copies/mL) rebound which has been sustained for at least twenty four months. These results suggest the possible use of TLR7 agonists in combination with ART toward reduction of HIV reservoirs and ultimately finite therapies for HIV-1 infection. In addition, GS-9620 appears to be safe in healthy and HBV-infected subjects.

### 1.4. Rationale for Dose Selection/Dosing Interval

In 50 HCV and in 100 HBV patients, doses of up to 4 mg of GS-9620 were evaluated, either as a single dose or two doses one week apart. Safety data from these studies demonstrated that GS-9620 is well-tolerated with no evidence of dose dependent adverse events or laboratory abnormalities that are consistent with systemic immune activation such as flu-like symptoms, hematologic reductions or increases in liver enzymes including transaminases. In the majority of patients there was no detectable IFN- $\alpha$  in serum, consistent with the mechanism of action of pre-systemic innate immune system activation in the GALT and/or in the liver. Evidence of biological activity was observed in a dose dependent manner in these studies, with maximal induction of ISG15 occurring within 48 hours and return to baseline levels of expression within 168 hours (7 days). In addition, the safety of a weekly dosing interval was supported by the observed elimination half-life (median range ~ 8 to 25 hours for 1, 2, or 4 mg doses in HBV- or HCV-infected subjects) and that no accumulation of GS-9620 occurred following once-weekly dosing.

A dosing schedule of once every 2 weeks is planned for this protocol in order to verify the resolution of GS-9620-induced HIV-1 viremia prior to additional dosing. This schedule is more conservative than the weekly administrations used in the Phase 1 evaluations across the above-referenced studies in chronic hepatitis B and C patients.

In the current study GS-US-382-1450, approximately 32 HIV-1-infected subjects have received biweekly dosing with GS-9620 (1, 2 and 4 mg) or placebo for a total of 6 doses, and GS-9620 6 mg or placebo for a total of 10 doses. No safety issues including dose-limiting toxicities were identified; however, pharmacodynamic and virologic effects were limited. The protocol-defined safety evaluation committee (SEC) recommended proceeding with enrollment of the 6 mg cohort on February 7, 2017. In the 6 mg dose cohort (Cohort 4) of this study, 6 subjects experienced treatment-emergent AEs. Three of these subjects had AEs which were considered to be related to study drug by the investigator: one subject had decreased concentration, vivid dreams, sweats, and fatigue; another subject had headache and increased peripheral neuropathy; the third subject had fatigue, myalgia, and nasal congestion. All of these AEs were grade 1 or 2 and all resolved during the dosing period. There have been no grade 3 or 4 AEs, AEs leading to study drug discontinuation, SAEs or deaths. The protocol-defined SEC reviewed blinded safety data from the 6 mg cohort on 25 September 2017 and recommended proceeding with the addition of the 8 mg cohort (Cohort 5). In the 8 mg dose cohort (Cohort 5) of this study, a total of 8 subjects

have been enrolled and are currently being dosed with study drug. At the time of the interim safety data cut (30 April 2018), all subjects had completed 5 out of 10 doses, and 3 subjects had completed 6 doses. There have been no grade 3 or 4 AEs, AEs leading to study drug discontinuation, SAEs or deaths. Three subjects have had mild AEs considered related to study drug by the investigator. These AEs include chills and malaise in one subject, pyrexia and myalgia in another subject, and headache in the last subject. All resolved within one day and have not recurred after Dose 3, thus far. If the SEC recommends proceeding with the 10 mg dose escalation of GS-9620, Cohort 6 will be opened for enrollment with the potential to escalate to the 12 mg dose of GS-9620, starting with dose 4 (out of 10 total doses of GS-9620). In Cohort 6, the SEC will review blinded safety data after all subjects have completed three doses of 10 mg of GS-9620 or placebo. Dose escalation to 12 mg of GS-9620 within Cohort 6 will only be initiated if SEC approval is obtained.

The highest GS-9620 dose planned to be assessed in this clinical study may be up to 12 mg. Dose selection has been based on the results from the study in healthy volunteers (GS-US-243-0101) that showed dose-dependent ISG mRNA induction from 0.3 mg up to 12 mg in the absence of dose-dependent induction in serum IFN- $\alpha$ . As described above, dose escalation to Cohort 6 (GS-9620 10 mg) for the proposed study is also based on interim safety data from the ongoing 8 mg cohort (Cohort 5) as described above.

With regard to the proposed adaptive cohorts, food affects absorption of GS-9620 and administration of GS-9620 4 hours post-ingestion of a high fat meal in Study GS-US-243-0101 resulted in approximately 30% reduction of systemic exposures of GS-9620, minimal effect on PD biomarkers and improved tolerability. Dosing GS-9620 with an acidic solution may improve the solubility and absorption of the compound.

### 1.5. Rationale for Biomarker Testing

It is hypothesized that the mechanism of action of GS-9620 is partly due to the initial activation of the innate immune system via TLR7 positive pDCs, promoting activation and maturation of pDCs and the release of antiviral cytokines and chemokines including IFN-α. The matured pDCs present HIV antigens to HIV-specific CD4 and CD8 T cells, thereby enhancing the HIV-specific adaptive response (cytotoxic CD8 T cells). These multifaceted effector mechanisms (cytotoxic CD8 T cells, NK cells, and antiviral cytokines) together strengthen the lymphocyte anti-HIV immune response and may lead to lowering the viral set point.

To provide proof of concept on the mechanism of action of GS-9620 in HIV-1 infected patients, several exploratory immunological biomarkers will be examined and listed below. The testing outlined below is based upon the current state of scientific knowledge. It may be modified during or after the end of the study to remove tests no longer indicated and/or to add new tests based on the growing state of the art knowledge. The following samples and biomarkers will be examined:

- Whole blood samples will be collected for interferon stimulated gene (ISG) mRNA measurements
- Whole blood samples will be collected, mononuclear cells isolated, and frequency and phenotype (activation, maturation, exhaustion) of lymphocyte populations will be enumerated by flow cytometry.
- Whole blood samples will be collected, mononuclear cells isolated and the frequency of HIV-specific T-cells will be quantitated by ex vivo IFN-γ ELISPOT assay and poly-functional ICS.
- Levels of cytokines, chemokines, and inflammatory markers will be quantified by immunoassays.
- Stool samples will be collected in Cohorts 5 to 9 for testing of the fecal microbiome and exploratory analysis

# 1.6. Compliance

This study will be conducted in compliance with this protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements.

# 2. OBJECTIVES

The primary objective of this study is:

- To evaluate the safety and tolerability of GS-9620 at escalating, multiple doses of GS-9620 in HIV-1 infected virologically suppressed adults on ART
- To evaluate the virologic effect of GS-9620 as measured by changes in plasma HIV-1 RNA

The secondary objectives of this study are:

- To evaluate the plasma pharmacokinetics (PK) of GS-9620
- To evaluate the pharmacodynamics (PD) of GS-9620 as measured by changes in interferon-stimulated genes (ISGs) and serum cytokines in whole blood compared to placebo
- To evaluate effects of GS-9620 on whole blood immune cell activation (T cell, B cell, NK cell)

The exploratory objectives of this study are:



## 3. STUDY DESIGN

# 3.1. Endpoints

The primary safety endpoint of this study is:

• Incidence of treatment-emergent SAEs and all treatment-emergent adverse events

The primary virology endpoint of this study is:

• Maximum change from baseline in plasma HIV-1 RNA at any post-dose time point

The secondary endpoints of this study are:

- Change from baseline in plasma HIV-1 RNA at post-baseline visits
- Proportion of subjects with plasma HIV-1 RNA > 50 copies/mL at any post-dose timepoint

The exploratory endpoints of this study are:



## 3.2. Study Design

This protocol describes a randomized, double-blind, multi-cohort dose escalation study that will evaluate the safety and efficacy of 1 mg, 2 mg, 4 mg, 6 mg, 8 mg, 10 mg and 12 mg of GS-9620 or placebo administered orally every other week for 71 days (for Cohorts 1 to 3), 127 days (for Cohorts 4 to 6), CCI in HIV-1 infected, ARV-treated, virologically suppressed adults. For each cohort, subjects will be randomized in a 6:2 ratio to receive GS-9620 or placebo. For Cohorts 5, 6 CCI eight unique subjects per cohort will receive GS-9620 or placebo after an overnight fast. CCI

All subjects will receive a total of 6 doses (for Cohorts 1 to 3), 10 doses (for Cohorts 4 to 9) of their assigned study treatment administered once every other week. For all subjects in Cohort 6, Dose 4 (Day 43) will occur after SEC review has been
completed. If dose escalation is approved by the SEC, subjects in Cohort 6 will receive 12 mg of GS-9620 or placebo from Doses 4 to 10; if dose escalation is not approved by the SEC, subjects will continue receiving 10 mg of GS-9620 or placebo from Doses 4 to 10.

Subjects will continue their

ARV regimen for the entire study duration.

Subjects will return for an end of study visit 30 days after the last dose of study drug is taken.

Enrollment will initially be opened for Cohort 1 only. The SEC will review study progress, safety and virology data of enrolled subjects. After all subjects in a cohort have received at least three doses (Cohorts 1 to 3, and 6) or five doses (Cohorts 4 to 5), the SEC will review safety data from that cohort, including adverse events, clinical laboratory results and plasma HIV-1 RNA, before approving the next dose escalation.

**cohort may be suspended** if  $\geq 2$  out of 6 subjects receiving GS-9620 experience one or more DLTs considered related to study drug. The SEC will consist of members not directly involved with the conduct of the study. Please refer to the SEC Charter for additional details.

Figure 3-1. High-Level Study Schema





Figure 3-2. Cohort 6 Visit Schema



# 3.3. Study Treatments

For each cohort, 8 subjects will be randomized in a 6:2 ratio to receive GS-9620 or placebo. All subjects will receive a total of 6 doses (for Cohorts 1 to 3), 10 doses (for Cohorts 4 to 6), CCI of their assigned study treatment administered once every other week. Subjects will continue their existing ARV regimen for the entire study duration.

Cohort 1 (n=8): GS-9620 1 mg (n=6) or placebo-to-match (n=2)

Cohort 2 (n=8): GS-9620 2 mg (n=6) or placebo-to-match (n=2)

Cohort 3 (n=8): GS-9620 4 mg (n=6) or placebo-to-match (n=2)

Cohort 4 (n=8): GS-9620 6 mg (n=6) or placebo-to-match (n=2)

Cohort 5 (n=8): GS-9620 8 mg (n=6) or placebo-to-match (n=2) administered following overnight fasting

Cohort 6 (n=8): GS-9620 10 mg with potential to escalate to 12 mg (n=6) or placebo-to-match (n=2) administered following overnight fasting



#### 3.4. Duration of Treatment

The treatment duration is 71 days (Cohorts 1 to 3), 127 days (Cohorts 4 to 6), CCI

## 4. SUBJECT POPULATION

# 4.1. Number of Subjects and Subject Selection

Approximately up to seventy two (72) subjects who meet the inclusion/exclusion criteria will be enrolled. Subjects who discontinue study participation before completion of dosing for reasons other than study-treatment related adverse events may be replaced.

## 4.2. Inclusion Criteria (All Cohorts)

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

- 1) The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
- 2) HIV-1 infected males and non-pregnant, non-lactating females ≥ 18 years at Pre-Baseline/Day -13
- 3) On antiretroviral (ARV) regimen for  $\geq 12$  consecutive months prior to Pre-Baseline/Day -13
  - a) The following agents are allowed as part of the current ARV regimen: NRTIs, raltegravir, dolutegravir, rilpivirine, and maraviroc
  - b) The following agents are NOT allowed as part of the current ARV regimen: HIV protease inhibitors (including low dose ritonavir), cobicistat-containing regimens, elvitegravir, efavirenz, etravirine, and nevirapine
  - c) A change in ARV regimen ≥ 45 days prior to Baseline/Day 1 for reasons other than virologic failure (e.g. tolerability, simplification, drug-drug interaction profile) is allowed
- 4) Plasma HIV-1 RNA levels < 50 copies/mL at screening
- 5) Documented plasma HIV-1 RNA levels < 50 copies/mL (according to the local assay being used) for ≥ 12 months preceding the screening visit (measured at least twice using a licensed assay with a lower limit of quantitation of at least 40 copies/mL)
  - a) Unconfirmed virologic elevations of ≥ 50 copies/mL (transient detectable viremia, or "blip") prior to screening are acceptable. (If the lower limit of detection of the local HIV-1 RNA assay is < 50 copies/mL, the plasma HIV-1 RNA level cannot exceed 50 copies/mL on two consecutive HIV-1 RNA tests)
  - b) If ARV regimen is changed ≥ 45 days prior to Pre-Baseline/Day -13, plasma HIV-1 RNA <50 copies/mL at Pre-baseline/Day -13 visit is required.
- 6) No documented history of resistance to any components of the current ARV regimen

- 7) Availability of a fully active alternative ARV regimen, in the opinion of the Investigator, in the event of discontinuation of the current ARV regimen with development of resistance
- 8) Hemoglobin  $\geq 11.5$  g/dL (males) or  $\geq 11$  g/dL (females)
- 9) White blood cell  $\geq 4000 \text{ cells/}\mu\text{L}$
- 10) Platelets  $\geq 150,000/\text{mL}$
- 11) Absolute Neutrophil Count ≥ 1500 cells/µL
- 12) CD4 count  $\geq$  400 cells/ $\mu$ L
- 13) Albumin  $\geq$  3.9 g/dL
- 14) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 × upper limit of normal (ULN)
- 15) Estimated GFR ≥ 60 mL/min according to the Cockcroft-Gault formula for creatinine clearance {Cockcroft 1976}:
  - i. Male:  $(140 age in years) \times (wt in kg) = CLer (mL/min)$

 $72 \times (\text{serum creatinine in mg/dL})$ 

- ii. Female:  $(140 age in years) \times (wt in kg) \times 0.85 = CLcr (mL/min)$  $72 \times (serum creatinine in mg/dL)$
- 16) All subjects must agree to utilize male or female condoms during sexual activity, or practice sexual abstinence for the duration of the study.
- 17) Females of childbearing potential must agree to utilize highly effective contraception methods (as described in Appendix 5) or be non-heterosexually active or practice sexual abstinence from screening through the duration of study treatment and for 36 days following the last dose of study drug.
  - a) Female subjects who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
  - b) Female subjects who have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure must have a serum follicle stimulating hormone (FSH) level at screening within the post-menopausal range based on the Central Laboratory reference
- 18) Male subjects must agree to utilize a highly effective method of contraception during heterosexual intercourse (as described in Appendix 5) or be non-heterosexually active, or practice sexual abstinence from screening throughout the study period and for 90 days following discontinuation of investigational medicinal product

# 4.3. Exclusion Criteria (All Cohorts)

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study.

- 1) A new AIDS-defining condition diagnosed within 90 days prior to screening (refer to Appendix 6)
- 2) Hepatitis B surface antigen (HBsAg) positive
  - a) Positive anti-HBs antibody and negative HBsAg results are acceptable
- 3) Hepatitis C antibody (HCVAb) positive
  - a) Positive anti-HCV antibody and negative HCV PCR results are acceptable
- 4) Documented history of pre-ART CD4 nadir < 200 cells/µL
  - a) Unknown pre-ART CD4 nadir is acceptable
- 5) History of autoimmune disease (e.g. lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, sarcoidosis, moderate or severe psoriasis)
- 6) Acute febrile illness within 35 days prior to Pre-Baseline/Day -13
- 7) Participation in any other clinical trial (including observational trials) without prior approval from the sponsor is prohibited while participating in this trial
- 8) Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
- 9) History or presence of allergy or intolerance to the study drug or their components
- 10) Any vaccination or immunomodulatory concomitant medication within 30 days prior to Pre-Baseline/Day -13. Elective vaccination (e.g. flu shot, hepatitis A or B vaccine) during the course of the study will require prior approval from Sponsor.
- 11) Use of any other prohibited concomitant medications as described in Section 5.4 within 14 days prior to Baseline/Day 1 visit. Refer to the current Prescribing Information for the medications that are contraindicated with the current ARV regimen
- 12) Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.

## 4.4. Other Protocol Restrictions

Subjects will be encouraged to avoid strenuous or prolonged exercise, as well as saunas, steam baths, and sunbathing or other prolonged UV exposure, (eg in a tanning salon) from the screening evaluation until completion of end of study procedures, as these activities are known to affect certain clinical laboratory test parameters, (eg CPK) and may provide false indicators of a potentially treatment-related toxicity.

Subjects will also be prohibited from blood donation (in excess of that required for clinical care) within 30 days prior to Screening and 30 days after end of study.

Smokers and other current tobacco users should keep their tobacco use relatively consistent while enrolled in the study. Non-smokers or ex-smokers should not start or resume smoking.

Other restrictions include all illegal or illicit drug use and use of prescription drugs outside the care of the prescribing physician.

#### 5. INVESTIGATIONAL MEDICINAL PRODUCTS

# 5.1. Randomization, Blinding and Treatment Codes

The randomization will be performed via an Interactive Web Response System (IWRS), whereby study treatment will be assigned to subjects according to the randomization schedule.

The subject number assignment may be performed up to 3 days prior to the in-clinic Pre-Baseline/Day -13 visit, provided that all other screening procedures have been completed and subject eligibility has been confirmed. Once a subject number has been assigned, it will not be reassigned to any other subject.

Eligible subjects (n= 72, 8 per cohort) will be randomized in a 6:2 ratio to receive GS-9620 1 mg or placebo (Cohort 1), 2 mg or placebo (Cohort 2), 4 mg or placebo (Cohort 3), 6 mg or placebo (administered as three 2 mg tablets) (Cohorts 4 CCI 8 mg or placebo (administered as two 4 mg tablets) (Cohort 5), 10 mg or placebo (Cohort 6) (administered as five 2 mg tablets), with the potential to escalate to 12 mg or placebo (administered as six 2 mg tablets, or three 4 mg tablets) with prior approval from SEC, CCI

Clinical Packaging & Labeling for purposes of managing blinded labeling and Clinical Supply Management for purposes of inventory management will remain unblinded throughout the study to prepare and manage the study drug. The Pharmacokinetics File Administrator, or designee, who facilitates data transfer of PK files between Gilead and vendors, will remain unblinded.

# **5.1.1.** Procedures for Breaking Treatment Codes

In the event of a medical emergency where breaking the blind is required to provide medical care to the subject, the investigator may obtain treatment assignment directly from the IWRS system for that subject. Gilead recommends but does not require that the investigator contact the Gilead medical monitor before breaking the blind. Treatment assignment should remain blinded unless that knowledge is necessary to determine subject emergency medical care. The rationale for unblinding must be clearly explained in source documentation and on the electronic case report form (eCRF), along with the date on which the treatment assignment was obtained. The investigator is requested to contact the Gilead medical monitor promptly in case of any treatment unblinding.

Blinding of study treatment is critical to the integrity of this clinical trial and therefore, if a subject's treatment assignment is disclosed to the investigator, the subject may have study treatment discontinued at SEC discretion. All subjects will be followed until study completion unless consent to do so is specifically withdrawn by the subject.

Gilead Pharmacovigilance and Epidemiology (PVE) may independently unblind cases for expedited reporting of suspected unexpected serious adverse reactions (SUSARs).

The SEC may also recommend unblinding of treatment assignments for one or more subjects to help determine if dosing can be resumed in subjects or cohorts where dosing has been suspended.

# 5.2. Description and Handling of GS-9620 and Placebo to match

#### **5.2.1.** Formulation

GS-9620 is available as 1 mg, 2 mg or 4 mg strength tablets. The tablets are round, biconvex, plain-faced, and film-coated white. Total tablet weight is 100 mg.

GS-9620 tablets contain lactose, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyethylene glycol, polyvinyl alcohol, talc, and titanium dioxide in addition to the active ingredient.

Placebo-to-match GS-9620 tablets are round, biconvex, plain-faced, and film-coated white. Total tablet weight is 100 mg.

Placebo tablets contain lactose, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyethylene glycol, polyvinyl alcohol, talc, and titanium dioxide.

## 5.2.2. Packaging and Labeling

GS-9620 tablets and placebo-to-match GS-9620 tablets are packaged in white, high density polyethylene bottles. Each bottle contains 5 tablets, silica gel desiccant, and polyester packing material. Each bottle is capped with a child-resistant polypropylene screw cap fitted with an induction seal, aluminum-faced liner.

Study drug(s) to be distributed to centers in the US shall be labeled to meet applicable requirements of the United States Food and Drug Administration (FDA) and/or other local regulations.

### **5.3.** Dosage and Administration of GS-9620

A blinded study staff member will utilize the IWRS system to obtain bottle numbers and dispense blinded GS-9620 or placebo-to-match tablets from these bottles to randomized subjects in the planned cohorts on their dosing days. Up to six bottles of study drug (5 tablets per bottle) may be assigned by the IWRS for each subject at randomization.

All subjects must remain on the same formulation throughout the duration of treatment. Subjects will be given their dose in the clinic once every two weeks, and will not take the study medication with them.

## 5.3.1. Fasting and food/liquids Requirement

The following fasting guidelines should be followed by subjects on *all* dosing days

Table 5-1. Fasting and food/liquids Requirement

| Cohort | Fasting Period | Water/liquids Permitted | Water/liquids at Dosing |
|---|---|---|---|
| 1 to 4 | At least 2 hours prior to and after dosing <sup>a</sup> | 1 hour prior to and 2 hours after dosing | 240 mL of water |
| 5, 6, <b>CCI</b> | Overnight <sup>b</sup> (at least 8hrs before dosing for Cohorts 5, 6 CCI and at least 2 hours after dosing | 1 hour prior to and 2 hours<br>after dosing | 240 mL of water |



- If subjects eat prior to the 2 hour fasting period before study drug dosing, no more than a light meal should be eaten (as described in the PK Sample Collection, Processing, Storage, and Shipment Manual).
- b If subjects did not fast overnight, plasma GS-9620 Intensive PK must not be completed. The subject should be counseled regarding proper fasting requirement and asked to return for the Intensive PK collection.

For Cohorts 1 to 4, GS-9620 or placebo should be taken by subjects with approximately 240 mL of water on an empty stomach. Food will not be permitted between at least 2 hours prior to and until 2 hours after dosing. Aside from the 240 mL of water provided at dosing, water/liquids will not be permitted from 1 hour prior to until 2 hours after dosing. If subjects eat prior to the 2 hour fasting period before study drug dosing, no more than a light meal should be eaten (as described in the PK Sample Collection, Processing, Storage, and Shipment Manual).

For Cohorts 5, 6 CCI, GS-9620 or placebo should be administered with 240 mL of water after an overnight fast (nothing but water for  $\geq 8$  hours prior to dosing).



[Note: For all cohorts, other than the water or cranberry juice provided with dosing, water and other fluids will be prohibited for 1 hour before and 2 hours after dosing.]





# 5.3.3. Storage and Handling

GS-9620 and placebo-to-match tablets should be stored at controlled room temperature of 25 °C (77 °F); excursions are permitted between 15 °C and 30 °C (59 °F and 86 °F). Storage conditions are specified on the label.

Until needed for IMP dispensation to the subjects, bottles of GS-9620 and placebo-to-match should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability of the tablets and proper product identification, the drug products should be stored in the containers in which they are supplied until needed. Keep the bottles tightly closed.

Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure through inhalation when handling GS-9620.

#### 5.4. Prior and Concomitant Medications

No clinical drug-drug interaction studies have been conducted with GS-9620. GS-9620 is predominantly metabolized by CYP3A with minor contribution of CYP2C8 and CYP2D6 in vitro, and was shown to be a substrate of P-gp and BCRP in vitro. GS-9620 plasma exposure may increase or decrease on co-administration with CYP3A/P-gp/BCRP inhibitors or inducers.

ARV agents known to inhibit or induce CYP3A/P-gp/BCRP are excluded from use in this protocol. The following agents are NOT allowed as part of the current ARV regimen: HIV protease inhibitors (including low dose ritonavir), cobicistat-containing regimens, elvitegravir, efavirenz, etravirine, and nevirapine.

Concomitant use of herbal/natural supplements with GS-9620 may result in pharmacokinetic interactions resulting in alterations in exposure of GS-9620. Administration of GS-9620 with grapefruit juice or Seville orange juice may result in higher exposures to GS-9620. Subjects will refrain from consumption of grapefruit juice, grapefruits, and Seville orange juice throughout participation in the study.

Subjects are restricted from receiving therapy with any medication listed in Table 5-3. Administration of any of the disallowed medications listed in Table 5-3 must be discontinued at least 14 days prior to the Baseline/Day 1 visit and through completion of treatment or the Early Study Drug Discontinuation Visit. Any medications not on the list must be reviewed with the Sponsor prior to randomization and during the study treatment period. Vitamins and/or acetaminophen and/or ibuprofen and/or hormonal contraceptive medications are exceptions and are allowed during the study period. No immunomodulatory concomitant medications are allowed for at least 30 days prior to Pre-Baseline/Day -13.

Subjects' ARV regimens must be used in accordance with their Prescribing Information.

At clinically achieved plasma concentrations, GS-9620 is not expected to be a perpetrator of systemic drug-drug interactions. GS-9620 concentrations estimated to be achieved in the gut at the ≥10 mg GS-9620 doses may transiently inhibit intestinal P-gp and increase systemic exposures of the drugs that are known P-gp substrates. It is recommended that oral P-gp substrates are administered with caution in combination with GS-9620 ≥10 mg doses.

**Table 5-3.** Prohibited Concomitant Medications

| Drug Class | Agents Disallowed | Use Discouraged and To be Used with Caution |
|---|---|---|
| Acid Reducing Agents | Proton Pump Inhibitors | H2-receptor antagonists <sup>a</sup> |
| ACAT inhibitor | Avasimibe | |
| ACE Inhibitors | Captopril | |
| Analeptic | Modafinil | |
| Angiotensin II inhibitors | Telmisartan | |
| Anti-anginals | Ranolazine | |
| Anti-arrhythmics | Amiodarone, Dronedarone, Quinidine | |
| Antibiotics | Azithromycin, Clarithromycin, Erythromycin,<br>Nafcillin, Telithromycin | Ciprofloxacin, Trimethoprim |
| Anticonvulsants | Carbamazepine, Phenytoin, Phenobarbital,<br>Oxcarbazepine | |
| Antidepressants | Nefazodone, Venlafaxine, Ziprasidone,<br>Paroxetine | |
| Antidiabetics | Pioglitazone | |
| Anti-epileptics | Divalproex | |
| Antiemetics | | Aprepitant, Casopitant |
| Antifungals | Caspofungin, Ketoconazole, Itraconazole, Voriconazole, Posaconazole, Fluconazole | |
| Antimycobacterials | Rifampin, Rifampentine, Rifabutin, Isoniazid | |
| Antiretroviral Agents | HIV Protease Inhibitors (including low dose<br>Ritonavir), Cobicistat-containing regimens,<br>Elvitegravir, Efavirenz, Etravirine and<br>Nevirapine | |
| Beta-Blockers | Carvedilol, Talinolol | |
| Calcium Channel Blockers | Diltiazem, Felodipine Mibefradil, Nicardipine,<br>Nifedipine, Nitrendipine, Verapamil | |
| Diuretics | Conivaptan | |
| Endothelin Receptor Antagonists | Bosentan | |
| Herbal/Natural Supplements* | St. John's Wort, Echinacea, Gingko, Milk<br>thistle, Chinese herb shosaiko-to<br>(or Xiao-Shai-Hu-Tang) | |
| HMG-Coa Reductase Inhibitors | Atorvastatin | Pitavastatin, Pravastatin,<br>Rosuvastatin, Lovastatin, Fluvastatin,<br>Simvastatin |
| Immunosuppressants | Cyclosporine, Rapamycin, Sirolimus,<br>Tacrolimus | |
| Systemic Corticosteroids | All agents, including dexamethasone | Use of Prednisone as a steroid burst (≤ 1 week of use) should be monitored appropriately |
| Systemic Chemotherapeutic (antineoplastic) Agents | All agents | |

a Dose not to exceed 20 mg famotidine or equivalent and dose should be administered not less than 24 hours prior to dosing with GS-9620 and not less than 12 hours after dosing with GS-9620.

<sup>\*</sup> Use of complementary or alternative medicines is prohibited at least 14 days prior to Baseline (Day 1) through the end of the follow-up

Should subjects have a need to initiate treatment with any concomitant medication, the Gilead Medical Monitor must be consulted prior to initiation of the new medication. In instances where a medication is initiated prior to discussion with the Sponsor, the Investigator must notify Gilead as soon as he/she is aware of the use of the medication.

## 5.5. Accountability for GS-9620

The investigator is responsible for ensuring adequate accountability of all used and unused study drug. This includes acknowledgement of receipt of each shipment of study drug (quantity and condition).

GS-9620 accountability records will be provided to each study site to:

- Record the date received and quantity of study drug bottles
- Record the date, subject number, subject initials, the study drug bottle number the pills were dispensed from.
- Record the date, quantity of used and unused study drug returned or destroyed, along with the initials of the person recording the information.

# 5.5.1. Investigational Medicinal Product Return or Disposal

Gilead recommends that used and unused IMP supplies be returned to the shipping facility from which it came for eventual destruction. The study monitor will provide instructions for return. If return is not possible, the study monitor will evaluate each study center's IMP disposal procedures and provide appropriate instruction for destruction of unused IMP supplies. If the site has an appropriate standard operating procedure (SOP) for drug destruction as determined by Gilead QA, the site may destroy used (empty or partially empty) and unused IMP supplies in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for central files.

If IMP is destroyed on site, the investigator must maintain accurate records for all IMP destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the IMP. Upon study completion, copies of the IMP accountability records must be filed at the site. Another copy will be returned to Gilead. If drug is destroyed on site, the investigator must maintain accurate records for all study drug bottles destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and person who disposed of the drug. All study drug records must be maintained at the site and copies must be submitted to Gilead Sciences at the end of the study.

The study monitor will review IMP supplies and associated records at periodic intervals.

## 6. STUDY PROCEDURES

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows.

The investigator must document any deviation from protocol procedures and notify the sponsor or contract research organization (CRO).

# 6.1. Subject Enrollment and Treatment Assignment

It is the responsibility of the investigator to ensure that subjects are eligible to participate in the study prior to enrollment. Each study candidate must sign an Informed Consent Form prior to the conduct of any screening procedures, in accordance with regulatory and local Institutional Review Board requirements. Once consent has been obtained, all screening tests and procedures have been completed, and study eligibility has been confirmed, subjects will be randomized using an IWRS. Subjects will receive study drug within their assigned treatment group as described in Section 5.1. With Gilead Medical Monitor approval, candidates who fail to meet eligibility criteria by screening evaluations may be re-screened if there is a reasonable expectation that the candidate will be eligible after repeat screening. The Medical Monitor must approve all re-screening requests.

Retests of screening labs are permitted only if there is reason to believe the retest value will be within accepted parameters, if the initial value was either due to a sample processing error or due to an extenuating circumstance (e.g. intercurrent infection). Reasons for any re-tests should be documented.

## 6.2. Pretreatment Assessments Screening Visit (all cohorts)

Subjects will be screened within 35 days before randomization to determine eligibility for participation in the study. The following will be performed and documented at screening:

- 6.2.1.1. Obtain written informed consent
- 6.2.1.2. Obtain medical history including history of HIV-1 disease-related events and prior medications within 35 days of the screening visit
- 6.2.1.2.1. Collect ARV history for at least 12 months
- 6.2.1.2.2. Collect pre-ARV viral set point, pre-ARV CD4 nadir and historical genotype(s), if available
- 6.2.1.3. Complete physical examination including vital signs (blood pressure, pulse, respiration rate and temperature), body weight, and height. Urogenital/anorectal exams will be performed at the discretion of the Investigator
- 6.2.1.4. 12-lead ECG performed supine
- 6.2.1.5. Obtain urine collection for urinalysis

- 6.2.1.6. Obtain blood samples for:
- 6.2.1.6.1. Serum pregnancy test (females of childbearing potential only). If the test is positive, the subject will not be enrolled
- 6.2.1.6.2. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid
- 6.2.1.6.3. Estimated GFR  $\geq$  60 mL/min according to the Cockcroft-Gault formula for creatinine clearance:

Male:  $(140 - age in years) \times (wt in kg) = CLcr (mL/min)$ 

 $72 \times (\text{serum creatinine in mg/dL})$ 

Female:  $(140 - age in years) \times (wt in kg) \times 0.85 = CLcr (mL/min)$ 

 $72 \times (\text{serum creatinine in mg/dL})$ 

- 6.2.1.6.4. Hematology profile: complete blood count (CBC) with differential and platelet count
- 6.2.1.6.5. CD4+ cell count
- 6.2.1.6.5.1. CD8+ cell count, CD4/CD8 ratio and CD4 % (for Cohorts 5 to 9 only)
- 6.2.1.6.6. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.2.1.6.7. Hepatitis B virus surface antigen serology
- 6.2.1.6.8. Hepatitis C virus serology
- 6.2.1.6.9. Plasma ART trough PK (for Cohorts 5 to 9 only)
- 6.2.1.7. Record any serious adverse events and all adverse events related to protocol mandated procedures occurring after signing of the consent form.

Subjects meeting all of the inclusion criteria and none of the exclusion criteria will return to the clinic within 35 days after the screening visit for the Pre-Baseline/Day -13 study visit.

From the time of obtaining informed consent through the first administration of investigational medicinal product, record all serious adverse events (SAEs), as well as any adverse events related to protocol-mandated procedures on the adverse events electronic case report form (eCRF). All other untoward medical occurrences observed during the screening period, including exacerbation or changes in medical history are to be captured on the medical history eCRF. See Section 7 Adverse Events and Toxicity Management for additional details.

# 6.2.2. Pre-Baseline/Day -13 Assessments (all Cohorts)

The following evaluations are to be completed at the Pre-Baseline/Day -13 visit. The Pre-Baseline/Day -13 visit is to be completed within  $\pm$  3 days of the protocol specified visit date.

- 6.2.2.1. Review of Inclusion/Exclusion criteria to confirm subject eligibility
- 6.2.2.2. Review of AEs and changes in concomitant medications
- 6.2.2.3. Review medical history
- 6.2.2.4. Symptom-directed physical examination as needed
- 6.2.2.5. Blood sample collection for the following laboratory analyses:
- 6.2.2.5.1. PBMC for HIV specific T cell response by ELISPOT CCI
- 6.2.2.5.2. TLR7 genotyping
- 6.2.2.5.3. Pharmacokinetic Blood Collection Details of pharmacokinetic blood sampling procedures and sample management for all PK samples in the study will be documented in the Pharmacokinetic Sample Collection, Processing, Storage, and Shipment Manual.
- 6.2.2.5.3.1. Pharmacokinetic assessments (**for Cohorts 1 to 3 only**) Plasma ARV concentrations: a single trough PK sample will be collected. The timing of the ARV trough collection is to be 20-24 hours following the subject's previous QD regimen dose (and, for any subject on a regimen containing a BID component, the trough collection must also occur 8-12 hours following the subject's previous dose of that BID component).
- 6.2.2.5.5. HIV specific polyfunctional T cell ICS (for Cohorts 4 to 9).
- 6.2.2.5.6. HIV-1 reservoir measurements (for Cohorts 4 to 9). CCI
- 6.2.2.5.7. Blood sample collection for future biomarker and virology studies (**for Cohorts 4 to 9**). CCI

- 6.2.2.6. Obtain subject number and randomize the subject via IWRS. The subject number assignment and randomization may be performed up to 3 days prior to the in-clinic Pre-Baseline/Day -13 visit provided that all screening procedures have been completed and subject eligibility has been confirmed.
- 6.2.2.7. Subjects should be reminded to come in for Day 1 visit in an overnight fasted state for Cohorts 5 to 9.

## 6.2.3. Baseline/Day 1 Assessments (all Cohorts)

Subjects are to arrive in a fasting state for the Baseline/Day 1 visit. Initiation of the treatment with the study drug must take place in the clinic and will be administered by blinded study staff. Fasting requirement and food/liquids consumption requirement is shown in Table 5-1.

For all cohorts, subjects will remain on-site for 12 hours after the first dose for safety assessments and phlebotomy. The following evaluations are to be completed at the Baseline/Day 1 Visit:

- 6.2.3.1. Review medical history
- 6.2.3.2. Review of AEs and changes in concomitant medication



- 6.2.3.4. Symptom-directed physical examination as needed
- 6.2.3.5. Vital signs (blood pressure, pulse, respiration rate and temperature)
- 6.2.3.6. Weight
- 6.2.3.7. VAS Adherence Questionnaire to be completed by the subject. Subject is to read questionnaire by himself/herself and write/mark answers directly onto questionnaires. (Cohorts 5 to 9 only)
- 6.2.3.8. Urine collection for the following laboratory procedures:
- 6.2.3.8.1. Urinalysis
- 6.2.3.8.2. Urine pregnancy test (females of childbearing potential only). If the urine pregnancy test is positive at Baseline/Day 1, study drug will not be dispensed. The positive result will be confirmed with a serum pregnancy test. If the serum pregnancy test is positive, the subject will not be able to participate

- 6.2.3.9. Blood sample collection for the following laboratory analyses:
- 6.2.3.9.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid
- 6.2.3.9.2. Estimated glomerular filtration rate according to the Cockcroft-Gault formula for creatinine clearance
- 6.2.3.9.3. Hematology profile: complete blood count (CBC) with differential and platelet count
- 6.2.3.9.4. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.2.3.9.5. CD4+ cell count
- 6.2.3.9.5.1 CD8+ cell count, CD4/CD8 ratio and CD4 % (Cohorts 5 to 9 only)
- 6.2.3.9.6. Serum for cytokine/soluble biomarker studies
- 6.2.3.9.7. Whole blood ISG mRNA panel
- 6.2.3.9.8. Cell-associated HIV-1 RNA/DNA (CAVR/CAVD) with stored PBMC.
- 6.2.3.9.9. Plasma HIV-1 RNA Single Copy Assay with stored plasma
- 6.2.3.9.10. Whole blood for immune cell activation (T, B, NK) and FoxP3+Treg level
- 6.2.3.9.11. PBMC intracellular cytokine staining (ICS) for Treg cells (for Cohorts 1 to 3 only)
- 6.2.3.9.12. Pharmacokinetic Blood Collection

Intensive PK sampling will occur at the following time points

- Pre-dose (≤5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 12 hours post dose at Baseline/Day 1;
- Then one sample on Day 3 at time = 48 hours post dose.

Details of pharmacokinetic blood sampling procedures and sample management for all PK samples in the study will be documented in the Pharmacokinetic Sample Collection, Processing, Storage, and Shipment Manual.

- 6.2.3.10. Stool sample collection before dosing for microbiome analysis (if subject is able to provide) (Cohorts 5 to 9).
- 6.2.3.11. In-Clinic Dosing
- Dose GS-9620 or placebo with 240 mL of water (All Cohorts, CCI
- 6.3. Treatment Assessments (Cohorts 1 to 3)
- 6.3.1. Treatment Assessments on Non Dosing Days 3, 5, 11, 17, 19, 25, 31, 33, 39, 45, 47, 53, 59, 61, 67, 73, 75 and 81

All study visits are to be scheduled relative to the Baseline/Day 1 visit. All study visits listed above **except for Day 3** allow a visit window within  $\pm$  1 day of the protocol specified visit date. The following procedures will be performed:

- 6.3.1.1. Review of AEs and changes in concomitant medications
- 6.3.1.2. Symptom-directed physical examination as needed
- 6.3.1.3. Blood sample collection for the following laboratory analyses:
- 6.3.1.3.1. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.3.1.3.2. Hematology profile: complete blood count (CBC) with differential and platelet count (Days 3, 17, 31, 45, 59 and 73 only)
- 6.3.1.3.3. CD4+ cell count (Days 3, 17, 31, 45, 59 and 73 only)
- 6.3.1.3.4. Serum for cytokine/soluble biomarker studies (Days 3, 17, 31, 45, 59 and 73 only)
- 6.3.1.3.5. Whole blood ISG mRNA panel (**Days 3, 17, 31, 45, 59 and 73 only**)
- 6.3.1.3.6. Cell-associated HIV-1 RNA/DNA with stored PBMC (Days 3, 45, and 73 only)
- 6.3.1.3.7. Plasma HIV-1 RNA Single Copy Assay with stored plasma (**Days 3, 45, and 73 only**)

- 6.3.1.3.8. Whole blood for immune cell activation (T, B, NK) (Days 3, 31 and 73 only)
- 6.3.1.3.9. PBMC Intracellular cytokine staining (ICS) for Treg cells (Days 3 and 73 only)
- 6.3.1.3.10. GS-9620 plasma pharmacokinetic assessment (**Day 3 only**)

## 6.3.2. Treatment Assessments on Non Dosing Days 8, 22, 36, 50, 64 and 78

All study visits are to be scheduled relative to the Baseline/Day 1 visit. Study visits on Days 8, 22, 36, 50, 64 and 78 are to be completed within  $\pm$  1 day of the protocol specified visit date. The following procedures will be performed:

- 6.3.2.1. Review of AEs and changes in concomitant medications
- 6.3.2.2. Symptom-directed physical examination as needed
- 6.3.2.3. Urine collection for urinalysis
- 6.3.2.4. Blood sample collection for the following laboratory analyses:
- 6.3.2.4.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid
- 6.3.2.4.2. Hematology profile: complete blood count (CBC) with differential and platelet count
- 6.3.2.4.3. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.3.2.4.4. CD4+ cell count
- 6.3.2.4.5. Serum for cytokine/soluble biomarker studies
- 6.3.2.4.6. Whole blood ISG mRNA panel

## 6.3.3. Treatment Assessments on Dosing Days 15, 29, 43, 57 and 71

On dosing days, GS-9620 or placebo should be taken by subject with approximately 240 mL of water on an empty stomach. Food will not be permitted between at least 2 hours prior to and until 2 hours after dosing. Aside from the 240 mL of water provided at dosing, water/liquids will not be permitted from 1 hour prior to until 2 hours after dosing. If subjects eat prior to the 2 hour fasting period before study drug dosing, no more than a light meal should be eaten (as described in the PK Sample Collection, Processing, Storage, and Shipment Manual).

These fasting guidelines should be followed by subjects on <u>all</u> dosing days.

Prior to the subject being administered the in-clinic dose the Investigator must verify the subject's continued eligibility for in-clinic dosing, including the absence of Dose Limiting Toxicities (DLTs) described in Section 7.6.1.

All doses will be directly administered to the study subject by blinded site staff.

| 6.3.3.1. | Review of AEs and changes in concomitant medication |
|---|---|
| 6.3.3.2. | Symptom-directed physical examination as needed |
| 6.3.3.3. | Vital signs (blood pressure, pulse, respiration rate and temperature) |
| 6.3.3.4. | Urine collection for the following laboratory procedures: |
| 6.3.3.4.1. | Urinalysis |
| 6.3.3.4.2. | Urine pregnancy test (females of childbearing potential only). If the urine pregnancy test is positive at a dosing visit, study drug will not be dispensed. The positive result will be confirmed with a serum pregnancy test. If the serum pregnancy test is positive, the subject will be discontinued from the study |
| 6.3.3.5. | Blood sample collection for the following laboratory analyses: |
| 6.3.3.5.1. | Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid |
| 6.3.3.5.2. | Hematology profile: complete blood count (CBC) with differential and platelet count |
| 6.3.3.5.3. | Plasma HIV-1 RNA (TaqMan® v2.0) |
| 6.3.3.5.4. | CD4+ cell count |
| 6.3.3.5.5. | Cell-associated HIV-1 RNA/DNA with stored PBMC (Days 43 and 71 only) |
| 6.3.3.5.6. | Serum for cytokine/soluble biomarker studies collected pre-dose |
| 6.3.3.5.7. | Whole blood ISG mRNA panel collected pre-dose |
| 6.3.3.5.8. | Plasma HIV-1 RNA Single Copy Assay with stored plasma collected pre-dose (Days 43 and 71 only) |
| 6.3.3.5.9. | Whole blood for immune cell activation (T, B, NK,) and FoxP3+Treg level collected pre-dose (Days 29 and 71 only) |

- 6.3.3.5.10. PBMC for ELISPOT collected pre-dose (Day 71 only)
- 6.3.3.5.11 PBMC Intracellular cytokine staining (ICS) for Treg cells (Day 71 only)
- 6.3.3.6. The Investigator will verify the subject's continued eligibility for in-clinic dosing, including the absence of DLTs described in Section 7.6.1.
- 6.3.3.7. In-Clinic Dosing
- 6.4. Treatment Assessments (Cohorts 4 to 9)

#### CCI

# 6.4.1. Treatment Assessments on Non Dosing Days 2, 58 and 128

All study visits are to be scheduled relative to the Baseline/Day 1 visit. The following procedures will be performed:

- 6.4.1.1. Review of AEs and changes in concomitant medications
- 6.4.1.2. Symptom-directed physical examination as needed
- 6.4.1.3. Urine collection for urinalysis (**Day 2 only**)
- 6.4.1.4. Blood sample collection for the following laboratory analyses:
- 6.4.1.4.2. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid (**Day 2 only**)
- 6.4.1.4.3. Hematology profile: complete blood count (CBC) with differential and platelet count (**Day 2 only**)
- 6.4.1.4.4. Plasma HIV-1 RNA (TagMan® v2.0)
- 6.4.1.4.5. Serum for cytokine/soluble biomarker studies
- 6.4.1.4.6. Whole blood ISG mRNA panel
- 6.4.1.4.7. Whole blood for immune cell activation (T, B, NK)

# 6.4.2. Treatment Assessments on Non Dosing Days 3, 59 and 129

All study visits are to be scheduled relative to the Baseline/Day 1 visit. The following procedures will be performed:

- 6.4.2.1. Review of AEs and changes in concomitant medications
- 6.4.2.2. Symptom-directed physical examination as needed
- 6.4.2.3. Urine collection for urinalysis (**Days 59 and 129 only**)
- 6.4.2.4. Blood sample collection for the following laboratory analyses:
- 6.4.2.4.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid (**Days 59 and 129 only**)
- 6.4.2.4.2. Hematology profile: complete blood count (CBC) with differential and platelet count (**Days 59 and 129 only**)
- 6.4.2.4.3. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.4.2.4.4. Serum for cytokine/soluble biomarker studies
- 6.4.2.4.5. Whole blood ISG mRNA panel
- 6.4.2.4.6. Cell-associated HIV-1 RNA/DNA with stored PBMC
- 6.4.2.4.7. Plasma HIV-1 RNA Single Copy Assay with stored plasma
- 6.4.2.4.8. Whole blood for immune cell activation (T, B, NK)
- 6.4.2.4.9. GS-9620 plasma pharmacokinetic assessment (Day 3 only)

# 6.4.3. Treatment Assessments on Non Dosing Days 8, 22, 36, 50, 64, 78, 92, 106, 120 and 134

All study visits are to be scheduled relative to the Baseline/Day 1 visit. Study visits on Days 8, 22, 36, 50, 64, 78, 92, 106, 120 and 134 are to be completed within  $\pm$  1 day of the protocol specified visit date. The following procedures will be performed:

- 6.4.3.1. Review of AEs and changes in concomitant medications
- 6.4.3.2. Symptom-directed physical examination as needed
- 6.4.3.3. Urine collection for urinalysis (Days 50, 64, 78, 92, 120 and 134 only)

- 6.4.3.4. Blood sample collection for the following laboratory analyses:
- 6.4.3.4.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid (Days 50, 64, 78, 92, 120 and 134 only)
- 6.4.3.4.2. Hematology profile: complete blood count (CBC) with differential and platelet count (Days 50, 64, 78, 92, 120 and 134 only)
- 6.4.3.4.3. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.4.3.4.4. CD4+ cell count (Days 50, 64, 78, 92, 120 and 134)
- 6.4.3.4.4.1 CD8+ cell count, CD4/CD8 ratio and CD4 % (Days 50, 64, 78, 92, 120 and 134 for Cohorts 5 to 9 only)
- 6.4.3.4.5. Serum for cytokine/soluble biomarker studies (Days 50, 64 and 134 only)
- 6.4.3.4.6. Whole blood ISG mRNA panel (**Days 50, 64 and 134 only**)
- 6.4.4. Treatment Assessments on Dosing Days 15, 29, 43, 57, 71, 85, 99, 113 and 127

Subjects are to arrive in a fasting state for the Dosing Days 15, 29, 43, 57, 71, 85, 99, 113 and 127 and to follow fasting and food/liquids consumption requirement shown in 1. Initiation of the treatment with the study drug must take place in the clinic and will be administered by blinded study staff.

For all subjects in Cohort 6, Dose 4 (Day 43) will occur after SEC review has been completed.

Prior to the subject being administered the in-clinic dose the Investigator must verify the subject's continued eligibility for in-clinic dosing, including the absence of Dose Limiting Toxicities (DLTs) described in Section 7.6.1.

All doses will be directly administered to the study subject by blinded site staff.

- 6.4.4.1. Review of AEs and changes in concomitant medication
- 6.4.4.2. Symptom-directed physical examination as needed
- 6.4.4.3. Vital signs (blood pressure, pulse, respiration rate and temperature)
- 6.4.4.4. Observe, if possible, and record the exact time that subject starts consuming the meal, the time that (s)he finishes the meal, and what (if anything) is not eaten and how much is consumed (**Cohort 9 only**)

- 6.4.4.5. VAS Adherence Questionnaire to be completed by the subject. Subject is to read questionnaire by himself/herself and write/mark answers directly onto questionnaires. (Days 29, 57, 99 and 127 for **Cohorts 5 to 9 only**)
- 6.4.4.6. Urine collection for the following laboratory procedures:
- 6.4.4.6.1. Urinalysis
- 6.4.4.6.2. Urine pregnancy test (females of childbearing potential only). If the urine pregnancy test is positive at a dosing visit, study drug will not be dispensed. The positive result will be confirmed with a serum pregnancy test. If the serum pregnancy test is positive, the subject will be discontinued from the study
- 6.4.4.7. Blood sample collection for the following laboratory analyses:
- 6.4.4.7.1 Plasma ART trough PK (Days 29, 57, 85 and 99 for Cohort 5; Days 57 and 99 for Cohorts 6
- 6.4.4.7.2. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid
- 6.4.4.7.3. Hematology profile: complete blood count (CBC) with differential and platelet count
- 6.4.4.7.4. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.4.4.7.5. CD4+ cell count
- 6.4.4.7.5.1 CD8+ cell count, CD4/CD8 ratio and CD4 % (Cohorts 5 to 9 only)
- 6.4.4.7.6. Cell-associated HIV-1 RNA/DNA (CAVR/CAVD) with stored PBMC (**Days 57** and 127 only)
- 6.4.4.7.7. Serum for cytokine/soluble biomarker studies **collected pre-dose (Day 43** for Cohort 6 subjects who receive 12 mg at Dose 4; **Days 57 and 127** for all subjects)
- 6.4.4.7.8. Whole blood ISG mRNA panel **collected pre-dose (Day 43** for Cohort 6 subjects who receive 12 mg at Dose 4; **Days 57 and 127** for all subjects)
- 6.4.4.7.9. Plasma HIV-1 RNA Single Copy Assay with stored plasma **collected pre-dose** (Days 57 and 127 only)
- 6.4.4.7.10. Whole blood for immune cell activation (T, B, NK,) and FoxP3+Treg level collected pre-dose (Days 57 and 127 only)

# 6.4.4.7.11. Pharmacokinetic Blood Collection (only if the SEC approves the dose escalation to 12 mg in Cohort 6, starting from Dose 4 and onwards)

Intensive PK sampling will occur at the following time points

- Pre-dose ( $\leq$ 5 minutes prior to dosing), 0.5, 1, 2, 4, 6, 8, 10, and 12 hours post dose at Day 43;
- Then one sample on Day 45 (48 hours post dose)

Details of pharmacokinetic blood sampling procedures and sample management for all PK samples in the study will be documented in the Pharmacokinetic Sample Collection, Processing, Storage, and Shipment Manual.

- 6.4.4.8. The Investigator will verify the subject's continued eligibility for in-clinic dosing, including the absence of DLTs described in Section 7.6.1.
- 6.4.4.9. In-Clinic Dosing

# 6.4.5. Treatment Assessments on Non Dosing Days 31, 45, 73, 87, 101 and 115 (For Cohorts 5 to 9 only)

All study visits are to be scheduled relative to the Baseline/Day 1 visit. Study visits on Day 31, Day 45, Day 73, Day 87, Day 101 and Day 115 Day are to be completed within  $\pm$  1 day of the protocol specified visit date. The following procedures will be performed:

- 6.4.5.1. Review of AEs and changes in concomitant medication
- 6.4.5.2. Symptom-directed physical examination as needed
- 6.4.5.3. Urine collection for urinalysis (Days 73, 87, 101 and 115 only)
- 6.4.5.4. Blood sample collection for the following laboratory analyses:
- 6.4.5.4.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid (Days 73, 87, 101 and 115 only)
- 6.4.5.4.2. Hematology profile: complete blood count (CBC) with differential and platelet count (**Days 73, 87, 101 and 115 only**)
- 6.4.5.4.3. Plasma HIV-1 RNA (TaqMan<sup>®</sup> v2.0)
- 6.4.5.4.4. Serum for cytokine/soluble biomarker studies (**Day 45**, only if the SEC approves the dose escalation to 12 mg in Cohort 6 starting from Dose 4)
- 6.4.5.4.5. Whole blood ISG mRNA panel (**Day 45**, only if the SEC approves the dose escalation to 12 mg in Cohort 6 starting from Dose 4)

## 6.5. Post-treatment Assessments

# 6.5.1. End of Study Visit (all Cohorts)

30 days after the last administration of study drug, subjects will return to the study center to complete an end of study visit. For the purpose of scheduling the end of study visit,  $a \pm 3$  days window may be used. The following evaluations and/or procedures will be performed at the end of study visit for all cohorts, unless otherwise specified:

- 6.5.1.1. Review of AEs and changes in concomitant medication
- 6.5.1.2. Symptom-directed physical examination as needed
- 6.5.1.3. Weight
- 6.5.1.4. Urine collection for the following laboratory procedures:
- 6.5.1.4.1. Urinalysis
- 6.5.1.4.2. Urine pregnancy test (females of childbearing potential only, if not done within the previous 30 days).
- 6.5.1.5. Stool sample collection for microbiome analysis (if subject is able to provide)

  (Cohorts 5 to 9 only). CCI
- 6.5.1.6. Blood sample collection for the following laboratory analyses:
- 6.5.1.6.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid
- 6.5.1.6.2. Estimated glomerular filtration rate according to the Cockcroft-Gault formula for creatinine clearance
- 6.5.1.6.3. Hematology profile: complete blood count (CBC) with differential and platelet count
- 6.5.1.6.4. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.5.1.6.5. CD4+ cell count
- 6.5.1.6.5.1 CD8+ cell count, CD4/CD8 ratio and CD4 % (Cohorts 5 to 9 only)
- 6.5.1.6.6. Cell-associated HIV-1 RNA/DNA (CAVR/CAVD) with stored PBMC



Subjects who prematurely discontinue study drug will be required to complete an Early Study Drug Discontinuation Visit (ESDD) within 30 days after their last dose of study treatment.

If a subject discontinues study dosing (for example, as a result of an AE) every attempt should be made to keep the subject in the study and continue to perform the required study-related follow-up and procedures.

At the ESDD Visit, any evaluations showing abnormal results indicating that <u>there is a possible or probable causal relationship with the study drug</u>, should be repeated weekly (or as often as deemed prudent by the Investigator) until the abnormality is resolved, returns to baseline, or is otherwise explained.

The following evaluations are to be completed at the Early Study Drug Discontinuation Visit for all cohorts, unless otherwise specified:

- 6.5.2.1. Review of AEs and changes in concomitant medication
- 6.5.2.2. Symptom-directed physical examination as needed
- 6.5.2.3. Weight

- 6.5.2.4. Urine collection for the following laboratory procedures:
- 6.5.2.4.1. Urinalysis
- 6.5.2.4.2. Urine pregnancy test (females of childbearing potential only).
- 6.5.2.5. Stool sample for microbiome analysis (if subject is able to provide)

(Cohorts 5 to 9). CCI

- 6.5.2.6. Blood sample collection for the following laboratory analyses:
- 6.5.2.6.1. Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, phosphorus, magnesium, potassium, sodium, uric acid
- 6.5.2.6.2. Estimated glomerular filtration rate according to the Cockcroft-Gault formula for creatinine clearance
- 6.5.2.6.3. Hematology profile: complete blood count (CBC) with differential and platelet count
- 6.5.2.6.4. Plasma HIV-1 RNA (TaqMan® v2.0)
- 6.5.2.6.5. CD4+ cell count
- 6.5.2.6.5.1 CD8+ cell count, CD4/CD8 ratio and CD4 % (Cohorts 5 to 9 only)
- 6.5.2.6.6. Serum for cytokine/soluble biomarker studies
- 6.5.2.6.7. Whole blood ISG mRNA panel

# 6.6. Criteria for Discontinuation of Study Treatment

Study medication may be discontinued in the following instances:

- Intercurrent illness that would, in the judgment of the investigator, affect assessments of clinical status to a significant degree
- Unacceptable toxicity, or toxicity that, in the judgment of the investigator, compromises the ability to continue study-specific treatment and/or procedures or is considered to not be in the subject's best interest
- Subject receives GS-9620 and experiences one or more DLTs (at discretion of SEC)

- Subject request to discontinue for any reason
- Subject noncompliance
- Pregnancy during the study; refer to Appendix 5
- Discontinuation of the study at the request of Gilead, a regulatory agency or an institutional review board (IRB)



# 6.8. Prolonged Viremia

Subjects will be considered to have prolonged viremia if they have two consecutive plasma HIV-1 RNA levels  $\geq$  200 copies/mL during a single dosing period.

# **6.8.1.** Management of Prolonged Viremia

If plasma HIV-1 RNA level is  $\geq 200$  copies/mL at any visit post-dose, viral load will be tested at next scheduled visit or retested within 4 days. The next dose will be withheld and only given after viral load of  $\leq 200$  copies/mL is achieved. The study procedure schedule will be reset relative to the next dose of study drug.

If HIV-1 RNA viral load  $\geq$  200 copies/mL is confirmed during a single dosing period, then this subject will be considered to have prolonged viremia and blood samples from this visit will be used for HIV-1 genotype/phenotype testing with assays corresponding to the antiretroviral medications the subject is taking.

If primary resistance mutations to the subject's existing ART regimen are identified, a new ART regimen will be configured at the discretion of the Investigator and the subject will be discontinued from the study. If the genotyping/phenotyping assay fails to provide results or no drug resistance mutations are identified, a new ART regimen may be configured at the discretion of the Investigator. Subjects who start a new ART regimen will not be allowed to receive further doses of study drug, but can be monitored for the study duration at the discretion of the study Investigator. Subjects who remain on their current ART regimen must show confirmed HIV-1 RNA levels <200 copies/mL before resuming study drug dosing at the discretion of the Investigator.

## 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

# 7.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

#### 7.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or post-treatment complications that occur as a result of protocol specified procedures, lack of efficacy, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported.
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the screening visit that do not worsen
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions)
- Overdose without clinical sequelae (see Section 7.7.1)
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history eCRF.

#### 7.1.2. Serious Adverse Events

A serious adverse event (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
- In-patient hospitalization or prolongation of existing hospitalization

- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is a reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

# 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to IMP interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

For specific information on handling of clinical laboratory abnormalities in this study, please refer to Section 7.5.

#### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

## 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to IMP therapy using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the IMP. For SAEs, an alternative causality must be provided (eg, pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the event may have been caused by the investigational medicinal product.

It should be emphasized that ineffective treatment should not be considered as causally related in the context of adverse event reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures, (eg., venipuncture)

# 7.2.2. Assessment of Severity

A distinction should be drawn between seriousness and severity of AEs. An AE that is assessed as Grade 4 (potentially life-threatening) should not be confused with an SAE. Severity is a category utilized for rating the intensity of an event; and both AEs and SAEs can be assessed as Grade 4. An event is defined as "serious" when it meets one of the predefined outcomes described above in Section 7.1.2.

Severity should be recorded and graded according to the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities (Appendix 4) For adverse events associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events to Gilead

## Requirements for collection prior to study drug initiation:

After informed consent, but prior to initiation of study medication, the following types of events should be reported on the case report form (eCRF): all serious adverse events (SAEs) and adverse events related to protocol-mandated procedures.

#### **Adverse Events**

Following initiation of study medication, collect all AEs, regardless of cause or relationship, until 30 days after last administration of study IMP must be reported to the eCRF database as instructed.

All AEs should be followed up until resolution or until the adverse event is stable, if possible. Gilead Sciences may request that certain AEs be followed beyond the protocol defined follow up period.

#### **Serious Adverse Events**

All SAEs, regardless of cause or relationship, that occurs after the subject first consents to participate in the study (ie, signing the informed consent) and throughout the duration of the study, including the protocol-required post treatment follow-up period, must be reported to the eCRF database and Gilead Pharmacovigilance and Epidemiology (PVE) as instructed. This also includes any SAEs resulting from protocol-associated procedures performed after informed consent is signed.

Any SAEs and deaths that occur after the post treatment follow-up visit but within 4 weeks of the last dose of study IMP, regardless of causality, should also be reported.

Investigators are not obligated to actively seek SAEs after the protocol defined follow up period, however, if the investigator learns of any SAEs that occur after study participation has concluded and the event is deemed relevant to the use of IMP, he/she should promptly document and report the event to Gilead PVE.

• All AEs and SAEs will be recorded in the eCRF database within the timelines outlined in the eCRF completion guideline.

# **Electronic Serious Adverse Event (eSAE) Reporting Process**

- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead PVE within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form and submit within 24 hours to Gilead PVE:

Gilead Sciences PVE Representative: Fax: PPD E-mail: PPD

- As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF database according to instructions in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.
- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other
  documents are also to be submitted by e-mail or fax when requested and applicable.
   Transmission of such documents should occur without personal subject identification,
  maintaining the traceability of a document to the subject identifiers.
- Additional information may be requested to ensure the timely completion of accurate safety reports.
- Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's eCRF and the event description section of the SAE form.

# 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports associated with any study IMP. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

# 7.5. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities are usually not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, urinalysis) independent of the underlying medical condition that require medical or surgical intervention or lead to investigational medicinal product interruption or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE (or SAE) as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (ie, anemia) not the laboratory result (ie, decreased hemoglobin).

Severity should be recorded and graded according to the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities (Appendix 4) For adverse events associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.
## 7.6. Toxicity Management

## 7.6.1. Management of Dose-Limiting Toxicities (DLTs)

Prior to the subject being administered the in-clinic dose the Investigator will verify the subjects continued eligibility for dosing, including the absence of DLTs listed below:

- ALT elevation as defined as:
  - ALT  $\geq 10 \times \text{ULN OR}$
  - Confirmed ALT elevation (ie. Grade shift or 2× previous value) with evidence of worsened hepatic function (e.g. total bilirubin > 2mg/dL above Baseline, serum albumin > 1 g/dL decrease from Baseline)
- A confirmed ≥ Grade 3 AE considered drug related by the Investigator
- A confirmed, clinically significant ≥ Grade 3 laboratory abnormality considered study drug-related by the investigator
- A persistent (≥ 72 hours) ≥ Grade 2 flu-like symptom (pyrexia, fatigue, myalgia, arthralgia, headache, chills) considered study drug-related by the investigator
- A post-dose increase in plasma HIV-1 RNA that fails to resolve to < 50 copies/mL within 10 days in Cohorts 1 to 3
- A post-dose increase in plasma HIV-1 RNA that fails to resolve to < 200 copies/mL within 10 days in Cohorts 4 to 9

The designated Safety Evaluation Committee contact will be notified within 24 hours of the Investigator's knowledge of a subject having any of the above DLTs. Dosing must be withheld until the Safety Evaluation Committee determines the appropriate next steps, including but not limited to additional safety, pharmacokinetic and pharmacodynamic assessments. The SEC may also suspend dosing in additional subjects or cohorts.

The SEC may hold or discontinue study drug dosing for a subject if they receive GS-9620 and experience one or more DLTs. The SEC may hold or discontinue study drug dosing for a cohort if  $\geq 2$  out of 6 subjects receiving GS-9620 experience one or more DLTs.

## 7.6.2. Management of Other Toxicities

Unless otherwise specified in Section 7.6.1, toxicities will be managed according to the guidelines below.

- All clinical and clinically significant laboratory toxicities will be managed according to uniform guidelines detailed in Appendix 3.
- Grade 3 and 4 clinically significant laboratory abnormalities should be confirmed by repeat testing within 3 calendar days of receipt of results and before investigational medicinal product (IMP) discontinuation, unless such a delay is not consistent with good medical practice.
- Clinical events and clinically significant laboratory abnormalities will be graded according to the Table for GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities (Appendix 4).
- When restarting IMP following resolution of the adverse event, the investigational medicinal product should be restarted at full dose or modified dose that is dependent upon discussion with the Gilead Sciences Medical Monitor.
- Any recurrence of the Grade 3 or 4 clinical or clinically significant laboratory adverse event following dose interruption mandates permanent discontinuation of IMP.
- Any questions regarding toxicity management should be directed to the Gilead Sciences Medical Monitor.

## 7.6.2.1. Grades 1 and 2 Laboratory Abnormality or Clinical Event

Continue investigational medicinal product at the discretion of the Investigator.

## 7.6.2.2. Grade 3 Laboratory Abnormality or Clinical Event

- For a Grade 3 clinical event or clinically significant Grade 3 laboratory abnormality confirmed by repeat testing, IMP should be withheld until the toxicity returns to ≤ Grade 2.
- If a laboratory abnormality recurs to ≥ Grade 3 following rechallenge with IMP, then IMP should be permanently discontinued and the subject managed according to local practice.

## 7.6.2.3. Grade 4 Laboratory Abnormality or Clinical Event

• For a Grade 4 clinical event or clinically significant Grade 4 laboratory abnormality confirmed by repeat testing, IMP should be withheld until the toxicity returns to ≤ Grade 2.

• For a Grade 4 clinical event or clinically significant Grade 4 laboratory abnormality confirmed by repeat testing that is considered related to IMP, IMP should be permanently discontinued and the subject managed according to local practice. The subject should be followed as clinically indicated until the laboratory abnormality returns to baseline or is otherwise explained, whichever occurs first. A clinically significant Grade 4 laboratory abnormality that is not confirmed by repeat testing should be managed according to the algorithm for the new toxicity grade.

Investigational medicinal product may be continued without dose interruption for a clinically non-significant (and therefore not an AE), Grade 4 laboratory abnormality (eg, Grade 4 CK after strenuous exercise, or triglyceride elevation that is non-fasting or that can be medically managed).

## 7.7. Special Situations Reports

## 7.7.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, reports of adverse events associated with product complaints, occupational exposure with an AE, AE in an infant following exposure from breastfeeding and pregnancy reports regardless of an associated AE.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labelling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging, or distribution of the medicinal product.

## 7.7.2. Instructions for Reporting Special Situations

## 7.7.2.1. Instructions for Reporting Pregnancies

Subjects should be instructed to notify the investigator if they become pregnant at any time during the study, or if they become pregnant within 4 weeks of last study drug dose. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator, and seek the investigator's advice regarding action required with study drug immediately. The investigator should counsel the subject regarding the possible effects of prior study drug exposure on the fetus and the need to inform the study site of the outcome of the pregnancy.

The investigator should report pregnancies in female study subjects that are identified after initiation of study medication and throughout the study, including the post study drug follow-up period, to Gilead PVE using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of pregnancy reporting.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in the Adverse and Serious Adverse Section 7.1.1 and 7.1.2. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to Gilead PVE.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to Gilead PVE using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead PVE. Gilead PVE contact information is as follows:

Gilead Sciences PVE Representative:

Fax:
PPD
PPD
PPD

Pregnancies of female partners of male study subjects exposed to Gilead or other study drugs must also be reported and relevant information should be submitted to or Gilead PVE using the pregnancy and pregnancy outcome forms within 24 hours. Monitoring of the subject should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead PVE, fax number PPD or email PPD

Refer to Appendix 5 for Pregnancy Precautions, Definition for Female of Childbearing Potential and Contraceptive Requirements.

## 7.7.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to or Gilead PVE within 24 hours of the investigator becoming aware of the situation. These reports must consist of situations that involve study IMP and/or Gilead concomitant medications, but do not apply to non-Gilead concomitant medications.

Special situations involving non-Gilead concomitant medications do not need to be reported on the special situations report form; however, for special situations that result in AEs due to a non-Gilead concomitant medication, the AE should be reported on the AE form.

Any inappropriate use of concomitant medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to section and the eCRF completion guidelines for full instructions on the mechanism of special situations reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

Special Situations reports should be sent to Gilead Sciences PVE:

Gilead Sciences PVE Representative: Fax: PPD E-mail: PPD

CONFIDENTIAL Page 77 16 January 2019

## 8. STATISTICAL CONSIDERATIONS

## 8.1. Analysis Objectives and Endpoints

## 8.1.1. Analysis Objectives

The primary analysis objectives are:

- To evaluate the safety and tolerability of escalating, multiple doses of GS-9620 in HIV-1 infected virologically suppressed adults on ART
- To evaluate the virologic effect of GS-9620 as measured by changes in plasma HIV-1 RNA.

The secondary analysis objectives are:

- To evaluate the PK of GS-9620
- To evaluate the PD of GS-9620 as measured by changes in ISGs and serum cytokines in whole blood compared to placebo
- To evaluate effects of GS-9620 on whole blood immune cell activation (T cell, B cell, NK cell)

The exploratory analysis objectives are:



## 8.1.2. Primary Endpoint

- The primary safety endpoint is incidence of treatment-emergent SAEs and all treatment-emergent adverse events.
- The primary virology endpoint is maximum change from baseline in plasma log<sub>10</sub> HIV-1 RNA at any post-dose timepoint

## 8.1.3. Secondary Endpoint

The secondary endpoints are:

- Change from baseline in plasma HIV-1 RNA at post-baseline visits
- Proportion of subjects with plasma HIV-1 RNA > 50 copies/mL at any post-dose timepoint

## 8.1.4. Other Endpoints of Interest

Other endpoints include:

- Change from baseline in the levels of serum cytokines
- Change from baseline and fold induction in mRNA for ISGs
- Change from baseline in peripheral blood lymphocyte count for T/B/NK/pDC/mDC including: CD4 and CD8 populations, CD4/CD8 ratio, CD4 % and lymphocyte activation (T, B and NK cells)

## 8.1.5. Exploratory Endpoints



## 8.2. Analysis Conventions

## 8.2.1. Analysis Sets

### 8.2.1.1. All Randomized

The randomized analysis set includes all subjects who are randomized into the study. This is the primary analysis set for by-subject listings.

### 8.2.1.2. Efficacy

## 8.2.1.2.1 Full Analysis Set

The full analysis set (FAS) will include all subjects who (1) are randomized into the study and (2) have received at least one dose of study drug. Subjects with major eligibility violations that are identifiable based on pre-randomization characteristics will be excluded.

Subjects will be grouped according to the treatment to which they were randomized.

## 8.2.1.3. Safety

The safety analysis set will include all randomized subjects who received at least one dose of study drug. All the data collected up to 30 days after subjects permanently discontinue their study drug will be included in the safety summaries. Subjects will be grouped according to the treatment they actually received.

### 8.2.1.4. Phamacokinetics

## 8.2.1.4.1 GS-9620 Pharmacokinetic Analysis Set

The GS-9620 pharmacokinetic (PK) analysis set will include all subjects who are randomized and have received at least one dose of study drug and for whom PK parameters of analyte GS-9620 are available.

### 8.2.1.4.2 ARV Pharmacokinetic Analysis Set

The ARV PK analysis set will include all subjects who are randomized and have received at least one dose of study drug and for whom the PK concentration of any analyte of the ARV is available.

### 8.2.1.5. Biomarkers

The biomarker analysis set will include all subjects who are randomized and have received at least one dose of study drug and for whom the biomarkers are available.

## **8.3.** Data Handling Conventions

Natural logarithm transformation for key PK parameters, such as C<sub>max</sub>, AUC<sub>last</sub> and AUC<sub>inf</sub>, will be applied for pharmacokinetic analysis, as appropriate.

PK concentration values below the limit of quantitation (BLQ) will be presented as "BLQ" in the concentration data listing, will be treated as zero for the determination of summary and order statistics, and will be excluded for natural logarithm transformation. PK parameter values that are BLQ will be presented as "BLQ" in the parameter data listing and will be excluded in any calculation of geometric means or ratios.

## 8.4. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods by treatment group.

Demographic summaries will include sex, race/ethnicity, and age.

Baseline data including body weight, height, body mass index, HIV-1 infection will be summarized.

### 8.5. Efficacy Analysis

### 8.5.1. Primary Analysis

The primary virology endpoint is the maximum change from baseline in plasma  $log_{10}$  HIV-1 RNA at any post-dose timepoint. It will be summarized by treatment group. The primary analysis of the efficacy will be based on the full analysis set (FAS).

## 8.5.2. Secondary Analyses

The change from baseline in plasma  $log_{10}$  HIV-1 RNA at post-baseline visits will be summarized by treatment group.

The number and proportion of subjects with plasma HIV-1 RNA > 50 copies/mL at any post-dose timepoint will be summarized by treatment group.

## 8.6. Safety Analysis

All safety analyses will be performed using the safety analysis set.

All safety data collected on or after the date that study drug was first taken up to the date of last dose of study drug plus 30 days will be summarized by treatment group according to the study drug received. Data for the pretreatment period and the period post the date of last dose of study drug plus 30 days will be included in data listings.

### 8.6.1. Extent of Exposure

A subject's extent of exposure to study drug will be generated from the study drug administration data. Exposure data will be summarized by treatment group.

Duration of exposure to study drug will be expressed as the number of weeks between the first and last dose of the study drug, inclusive, regardless of temporary interruptions in study drug administration and summarized by treatment.

Dosing information for individual subjects will be listed.

### **8.6.2.** Adverse Events

Clinical and laboratory adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database.

Treatment-emergent AEs are 1) any AEs with onset date on or after the study drug start date and no later than 30 days after the study drug stop date, or 2) any AEs leading to study drug discontinuation.

Summaries (number and percentage of subjects) of treatment-emergent adverse events (by SOC and PT) will be provided by treatment group. Additional summaries will include summaries for adverse events by grade, Investigator's assessment of relationship to study drug, and effect on study drug dosing.

On an ongoing basis adverse events will be reviewed for events that might meet the definition of Category C events that are indicative of an AIDS-Defining Diagnoses. The Gilead medical personnel will review the possible Category C events and approve the events that meet the definition. Those events that do meet the Category C definition of an AIDS-Defining Diagnosis will be listed.

A listing of Category C, AIDS-Defining Diagnosis can be found in Appendix 6.

### 8.6.3. Laboratory Evaluations

Selected laboratory data will be summarized using only observed data. Absolute values and changes from baseline at all scheduled visits will be summarized.

Graded laboratory abnormalities will be defined using the grading scheme defined in Grading of laboratory abnormalities provided in Appendix 4.

Incidence of treatment-emergent laboratory abnormalities, defined as values that increase at least one toxicity grade from baseline at any time post baseline up to and including the date of last dose of study drug plus 30 days, will be summarized by treatment group. If baseline data are missing, any graded abnormality (i.e., at least a Grade 1) will be considered treatment emergent. The maximum toxicity grade will be summarized by laboratory parameter.

Laboratory abnormalities that occur before the first dose of study drug or after the subject has been discontinued from treatment plus 30 days will be included in a data listing.

## 8.7. Pharmacokinetic Analysis

The concentration data of GS-9620 and ARV (trough samples), if analyzed, will be summarized by nominal sampling time using descriptive statistics. For GS-9620, pharmacokinetic parameters ( $C_{max}$ ,  $T_{max}$ ,  $C_{last}$ ,  $T_{last}$ ,  $\lambda z$ ,  $AUC_{inf}$ ,  $AUC_{last}$ , and  $t_{1/2}$ ) will be listed and summarized using descriptive statistics (e.g., sample size, arithmetic mean, geometric mean, coefficient of variation (%), standard deviation, median, minimum, and maximum). Plasma concentrations over time will be plotted in semi-logarithmic and linear formats as mean  $\pm$  standard deviation, and median (Q1, Q3). For ARVs, trough sample concentrations for an individual will be descriptively compared to historical data.

## 8.8. Sample Size

This is an exploratory study to characterize the safety and efficacy of GS-9620; therefore, no power calculation was performed. Sample size is determined based on empirical considerations. A total of up to 54 subjects receiving GS-9620 will provide reasonable preliminary assessment of safety.

## 8.9. Safety Evaluation Committee

A Safety Evaluation Committee (SEC) will review study progress, virology and safety of enrolled subjects. The SEC will consist of members not directly involved with the conduct of the study. After all subjects in a cohort have received at least three doses (Cohorts 1 to 3, and 6) or five doses (Cohorts 4 and 5), the SEC will review safety data from that cohort, including adverse events, clinical laboratory results, and plasma HIV-1 RNA, before approving opening of enrollment in the next cohort. For Cohort 6, SEC will confer once all subjects have completed 3 doses of 10 mg GS-9620, and recommend whether or not subjects may proceed with a dose escalation to 12 mg starting with Dose 4.

A cohort may be suspended if  $\geq 2$  out of 6 subjects receiving GS-9620 experience one or more DLTs considered related to study drug. Please refer to the SEC Charter for additional details.

### 8.10. Analysis Schedule

## **Interim Unblinded Analyses**

Prior to the final analysis, selected individuals from Gilead will be unblinded to assess the interim safety, virology, biomarker, and PK data of GS-9620. This group may consist of at least one representative from Clinical Research, Biostatistics, Clinical Pharmacology, Pharmacovigilance/Epidemiology, Biomarkers, Clinical Virology and may include other personnel as necessary.

The access to individual unblinded data (safety, virology, biomarker and PK) will be limited only to data relevant for analysis by the function representatives and will be summarized at the group level for regulatory documents and external submissions without revealing individual subject identification to protect study blind at the subject level. This group will review data (safety, virology, biomarker and PK) to support development of new clinical protocols, regulatory documents, and conference submissions.

## Final analysis

The Sponsor will conduct a final analysis of all data after the last subject in the study completes the last visit (Day 157) or prematurely discontinues from the study.

## 9. **RESPONSIBILITIES**

## 9.1. Investigator Responsibilities

## 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki (as amended in Edinburgh, Tokyo, Venice, Hong Kong, and South Africa), International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. These standards are consistent with the European Union Clinical Trials Directive 2001/20/EC and Good Clinical Practice Directive 2005/28/EC.

The investigator will ensure adherence to the basic principles of Good Clinical Practice, as outlined in 21 CFR 312, subpart D, "Responsibilities of Sponsors and Investigators," 21 CFR, part 50, "Protection of Human Subjects", and 21 CFR, part 56, "Institutional Review Boards".

The investigator and all applicable subinvestigators will comply with 21 CFR, Part 54, "Financial Disclosure by Clinical Investigators", providing documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug under study. This documentation must be provided prior to the investigator's (and any subinvestigators') participation in the study. The investigator and sub-investigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

### 9.1.2. Institutional Review Board (IRB) Review and Approval

The investigator (or sponsor as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an. The investigator will not begin any study subject activities until approval from the IRB has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the any modifications made to the protocol or any accompanying material to be provided to the subject after initial approval, with the exception of those necessary to reduce immediate risk to study subjects.

### 9.1.3. Informed Consent

The investigator is responsible for obtaining written informed consent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The investigator must use the most current approved consent form for documenting written informed consent. Each informed consent (or assent as applicable) will be appropriately signed and dated by the subject or the subject's legally authorized representative and the person conducting the consent discussion, and also by an impartial witness if required by.

## 9.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, another unique identifier (as allowed by local law) and an identification code will be recorded on any form or biological sample submitted to the Sponsor, or laboratory. Laboratory specimens must be labeled in such a way as to protect subject identity while allowing the results to be recorded to the proper subject. Refer to specific laboratory instructions NOTE: The investigator must keep a screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the trial. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator brochure, this protocol, eCRF, the IMP, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

### 9.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, eCRF and query forms, and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, ie, history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);
- Documentation of the reason(s) a consented subject is not enrolled
- Participation in study (including study number);
- Study discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol specific procedures were performed;

- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of IMP, including dates of dispensing and return;
- Record of all adverse events and other safety parameters (start and end date, and including causality and severity);
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, United States, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

## 9.1.6. Case Report Forms

For each subject consented, an eCRF will be completed by an authorized study staff member whose training for this function is documented according to study procedures. eCRF should be completed on the day of the subject visit to enable the sponsor to perform central monitoring of safety data. Subsequent to data entry, a study monitor will perform source data verification within the EDC system. Original entries as well as any changes to data fields will be stored in the audit trail of the system. Prior to database lock (or any interim time points as described in the clinical data management plan), the investigator will use his/her log in credentials to confirm that the forms have been reviewed, and that the entries accurately reflect the information in the source documents. The eCRF capture the data required per the protocol schedule of events and procedures. System-generated or manual queries will be issued to the investigative site staff as data discrepancies are identified by the monitor or internal Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site coordinator is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (e.g. data entry error). At the conclusion of the trial, Gilead will provide the site with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.5.

## 9.1.7. Investigational Medicinal Product Accountability and Return

Gilead recommends that used and unused IMP supplies be returned to the shipping facility from which it came for eventual destruction. The study monitor will provide instructions for return. If return is not possible, the study monitor will evaluate each study center's IMP disposal procedures and provide appropriate instruction for destruction of unused IMP supplies. If the site has an appropriate standard operating procedure (SOP) for drug destruction as determined by Gilead QA, the site may destroy used (empty or partially empty) and unused IMP supplies in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for central files.

If IMP is destroyed on site, the investigator must maintain accurate records for all IMP destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the IMP. Upon study completion, copies of the IMP accountability records must be filed at the site. Another copy will be returned to Gilead.

The study monitor will review IMP supplies and associated records at periodic intervals.

## 9.1.8. Inspections

The investigator will make available all source documents and other records for this trial to Gilead's appointed study monitors, to IRBs, or to regulatory authority or health authority inspectors.

## 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

## 9.2. Sponsor Responsibilities

## 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. The investigator must submit all protocol modifications to the IRB in accordance with local requirements and receive documented approval before modifications can be implemented.

## 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agency. Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

- The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form or the study has been completed at all study sites for at least 2 years
- The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation.
- No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.4).
- The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

## 9.3. Joint Investigator/Sponsor Responsibilities

## 9.3.1. Payment Reporting

Investigators and their study staff may be asked to provide services performed under this protocol, e.g. attendance at Investigator's Meetings. If required under the applicable statutory and regulatory requirements, Gilead will capture and disclose to Federal and State agencies any expenses paid or reimbursed for such services, including any clinical trial payments, meal, travel expenses or reimbursements, consulting fees, and any other transfer of value.

## 9.3.2. Access to Information for Monitoring

In accordance with regulations and guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the accuracy of the data recorded in the eCRF.

The monitor is responsible for routine review of the eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries on the eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

## 9.3.3. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

## 9.3.4. Study Discontinuation

Both the sponsor and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs, and IECs. In terminating the study, Gilead and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.

## 10. REFERENCES

- Bar KJ, Sneller MC, Harrison LJ, Justement JS, Overton ET, Petrone ME, et al. Effect of HIV Antibody VRC01 on Viral Rebound after Treatment Interruption. N Engl J Med 2016;375 (21):2037-50.
- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.
- European Medicines Agency (EMA). Pegasys: EPAR Scientific Discussion: 8 August 2006. 8 Aug, 2006.
- Fosdick A, Zheng J, Pflanz S, Frey CR, Hesselgesser J, Halcomb RL, et al. Pharmacokinetic and Pharmacodynamic Properties of GS-9620, a Novel TLR7 Agonist, Demonstrates ISG Induction without Detectable Serum Interferon at Low Oral Doses. J Pharmacol Exp Ther 2013.
- Joint United Nations Programme on HIV/AIDS (UNAIDS). Global Aids Update 2016. Available at: http://www.unaids.org/en/resources/documents/2016/Global-AIDS-update-2016. 31 May. 2016.
- Kubicek WG, Anderson WD, Geber WF. Effects of hypoxia on the course of induced fever in dogs and monkeys. Am J Physiol 1958;195 (3):601-13.
- Lanford RE, Guerra B, Chavez D, Giavedoni L, Hodara VL, Brasky KM, et al. GS-9620, an Oral Agonist of Toll-Like Receptor-7, Induces Prolonged Suppression of Hepatitis B Virus in Chronically Infected Chimpanzees. Gastroenterology 2013;144 (7):1508-17 e10.
- Li JZ, Etemad B, Ahmed H, Aga E, Bosch RJ, Mellors JW, et al. The size of the expressed HIV reservoir predicts timing of viral rebound after treatment interruption. AIDS 2016;30 (3):343-53.
- Lim SY, Osuna CE, Hraber PT, Hesselgesser J, Gerold JM, Barnes TL, et al. TLR7 agonists induce transient viremia and reduce the viral reservoir in SIV-infected rhesus macaques on antiretroviral therapy [Research Article]. Science translational medicine 2018;10:eaao452.
- Mocroft A, Vella S, Benfield TL, Chiesi A, Miller V, Gargalianos P, et al. Changing patterns of mortality across Europe in patients infected with HIV-1. EuroSIDA Study Group. Lancet 1998;352 (9142):1725-30.
- Palella FJ, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, et al. Declining Morbidity and Mortality Among Patients With Advanced Human Immunodeficiency Virus Infection. N Eng J Med 1998;338 (13):853-60.

- Pilaro AM, Green MD. Toxicologist's Review: Pegylated interferon-a 2b for the Treatment of Chronic Hepatitis C Infection (Biologics License Application # 99-1488). Clinical Pharmacology/Toxicology Branch, Division of Clinical Trials Design and Analysis, Center for Biologics Evaluation and Research. December 19. 2000.
- Schneider E, Whitmore S, Glynn KM, Dominguez K, Mitsch A, McKenna MT. Revised surveillance case definitions for HIV infection among adults, adolescents, and children aged <18 months and for HIV infection and AIDS among children aged 18 months to <13 years--United States, 2008. MMWR Recomm Rep 2008;57 (RR-10):1-12.
- Sogaard OS, Graversen ME, Leth S, Olesen R, Brinkmann CR, Nissen SK, et al. The Depsipeptide Romidepsin Reverses HIV-1 Latency In Vivo. PLoS pathogens 2015;11 (9):e1005142.
- Sterne J, Hernán M, Ledergerber B, Tilling K, Weber R, Sendi P, et al. Long-term effectiveness of potent antiretroviral therapy in preventing AIDS and death: a prospective cohort study. Lancet 2005;366 (9483):378-84.
- U. S. Department of Health and Human Services (DHHS), Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER). Guidance for Industry. Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. Rockville, MD. July, 2005.
- Vial T, Descotes J. Clinical toxicity of the interferons. Drug Saf 1994;10 (2):115-50.
- Vibholm L, Schleimann MH, Hojen JF, Benfield T, Offersen R, Rasmussen K, et al. Short-Course Toll-Like Receptor 9 Agonist Treatment Impacts Innate Immunity and Plasma Viremia in Individuals With Human Immunodeficiency Virus Infection. Clin Infect Dis 2017;64 (12):1686-95.

# 11. APPENDICES

| Appendix 1. | Investigator Signature Page |
|---|---|
| Appendix 2. | Study Procedures Table |
| Appendix 3. | Management of Clinical and Laboratory Adverse Events |
| Appendix 4. | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities |
| Appendix 5. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and |
| | Contraceptive Requirements |
| Appendix 6. | Definitions of Stage 3 Opportunistic Illnesses in HIV (CDC Guidelines) |

### Appendix 1.

## **Investigator Signature Page**

GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404

### STUDY ACKNOWLEDGEMENT

A Phase 1b, Randomized, Blinded, Placebo-Controlled Dose-Escalation Study of the Safety and Biological Activity of GS-9620 in HIV-1 Infected, Virologically Suppressed Adults

## GS-US-382-1450, Amendment 7, 16 January 2019

This protocol has been approved by Gilead Sciences, Inc. The following signature documents this approval.

| PPD | PPD |
|-------------------------------|------------------------|
| PPD (Printed) Medical Monitor | Signature |
| Date Dayuary 20 | 719 |
| ] | INVESTIGATOR STATEMENT |

I have read the protocol, including all appendices, and I agree that it contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Gilead Sciences, Inc. I will discuss this material with them to ensure that they are fully informed about the drugs and the study.

| Principal Investigator Name (Printed) | Signature |
|---------------------------------------|-------------|
| Date | Site Number |

#### Appendix 2. **Study Procedures Table**

| Study Proced | ures | Tabl | e (Co | hort | s 1 to | 3) | | | | | | | | | | | | | _ | | | | | | | | | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screena | Pre-Baseline | Dose 1 <sup>b</sup> | | | | | Dose 2 | | | · · | Pe | Dose 3 | Base | line | stud | ly vi | Stis Dose 4 | | | | | Dose 5 | | | | | Dose 6 | | | | | End of Study | 4400 |
| Study<br>Procedure | Day -48 | Day -13 | Baseline/<br>Day 1 | Day 3 | Day 5 | Day 8 | Day 11 | Day 15 | Day 17 | Day 19 | Day 22 | Day 25 | Day 29 | Day 31 | Day 33 | Day 36 | Day 39 | Day 43 | Day 45 | Day 47 | Day 50 | Day 53 | Day 57 | Day 59 | Day 61 | Day 64 | Day 67 | Day 71 | Day 73 | Day 75 | Day 78 | Day 81 | Day 101 | |
| Informed<br>Consent | X | | | | | | , | | | | | | | | | | 2,- | | | | | | | | | | | e : | | | | | | |
| Review I/E<br>Criteria | | X | | | | | | | | | | | | | 13 70 | 13 | er u | | | | | | | | | | | | | | | | | |
| Medical History <sup>d</sup> | X | X | X | | 2 | | 3 | | | | | | | 7 | 5 - 3 | \$ - S | 2, 3 | | | | | | | | S | 5 - 3 | | f= .7 | 1. | | | | | Г |
| AEs and Con<br>Meds | X | X | Х | X | X | X | X | X | X | X | X | X | x | X | X | X | X | X | X | X | X | X | x | X | X | X | X | x | X | X | X | X | X | X |
| Complete<br>Physical Exam <sup>e</sup> | X | | | | | | | | | | | | | | | | er e. | | | | | | | | | | | | | | | | | |
| Symptom<br>Directed<br>Physical Exam <sup>f</sup> | | Х | х | X | X | X | х | X | X | X | X | X | X | X | X | X | X | х | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х |
| 12-Lead ECG<br>(performed supi<br>ne) | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Vital Signs | X | | Х | | | | | X | | | | $\Box$ | X | | | | | X | | | | | X | | | | | X | | | | $\Box$ | | Γ |
| Weight | X | | X | * | 13 | | | | | | | | | | 7 | | | | | | | | | | 2 | | | e | | | | | X | X |
| Height | X | | | | | | | | | | | İ | | 2 | 35 | | | | | | | | | | | | | | | | | | | |

| | Screena | Pre-Baseline | Dose 1b | | | 3.1 | | se 2 | | | | | Dose 3 | Š. | | | | se 4 | | | | | se 5 | | | | | se 6 | | | | | End of Study | ESDD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sci | Pre | Do | ÷F | - 6 | S | | Dose | | | | D | | 2000 | line | | | Dose | _ | | | | Dose | 47 | | 5 - X | 4 4 | Dose | Ť | 1 | Ś | | En | ES |
| | | | | | · · | , | 97 | | | | | P | ost-I | oase | nne | stuc | ly VI | SILS | | | | | | | is . | 3 | | | | - 2 | | | _ | $\vdash$ |
| Study<br>Procedure | Day -48 | Day -13 | Baseline/<br>Day 1 | Day 3 | Day 5 | Day 8 | Day 11 | Day 15 | Day 17 | Day 19 | Day 22 | Day 25 | Day 29 | Day 31 | Day 33 | Day 36 | Day 39 | Day 43 | Day 45 | Day 47 | Day 50 | Day 53 | Day 57 | Day 59 | Day 61 | Day 64 | Day 67 | Day 71 | Day 73 | Day 75 | Day 78 | Day 81 | Day 101 | |
| Randomization | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Plasma HIV-1<br>RNA | X | | х | X | X | X | x | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CD4+ cell count | X | | X | X | 2 3 | X | 8 | X | X | | X | | X | X | \$ - A | X | 2 - 2 | X | X | | X | | X | X | S | X | 2 | X | X | | X | | X | X |
| Chemistry profile | X | | х | | | X | | x | | | X | | X | × | 3.6 X.0 | X | 0.00 NO | x | | | X | | X | Ni. | | X | 3.6 | x | 96 | | X | | X | X |
| Hematology<br>profile | X | | Х | X | | X | | X | X | | X | | X | X | 30 YA | X | | X | X | | X | | X | X | 8 | X | | X | X | | X | | X | X |
| HBV/HCV<br>Serology | X | | | | | | | | | | | | | | | | | | | | | | | | | | 50 St | S 10 | 3,0 | | | | | |
| Estimated GFR | X | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | X | X |
| Urinalysis | X | | X | | | X | | X | | | X | | X | | 7,1 | X | | X | | | X | | X | | 7 | X | | X | | | X | | X | X |
| Serum<br>Pregnancy Test <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | | | | S W | | | Ĭ | | | |
| Urine Pregnancy<br>Test <sup>g</sup> | | | X | | 2.4 | | | х | | | | | X | V. | 7.6 2.6 | 02 10 | 0.5. | X | | | | | X | 0 | | 24 2.0 | | x | 54 | 3 | | | X | X |
| Plasma GS-9620<br>Intensive PK <sup>h</sup> | | | Х | X | | ky c | 78 | | | | | | | 0<br>% | (3 Y) | | KV LL | | | | | | | | 50 | 31 73<br>74 July | | e 3 | | | | | | |
| Plasma ARV<br>Trough PK <sup>h</sup> | | х | | | | | | | | | | | | | | | | | | | | | | | | | | (a ) | 4 | | | | | |

| 8 | Screena | Pre-Baseline | Dose 1° | | | | | Dose 2 | | | | | Dose 3 | | | | | Dose 4 | | | | | Dose 5 | | | | | Dose 6 | | | | | End of Study | ESDD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <b>V</b> 1 | # 1 | - 1 | l <sub>g</sub> | | | | | | | | P | | Base | line | stud | ly vi | | | | | | | | | | | | Ý | | | | | |
| Study<br>Procedure | Day -48 | Day -13 | Baseline/<br>Day 1 | Day 3 | Day 5 | Day 8 | Day 11 | Day 15 | Day 17 | Day 19 | Day 22 | Day 25 | Day 29 | Day 31 | Day 33 | Day 36 | Day 39 | Day 43 | Day 45 | Day 47 | Day 50 | Day 53 | Day 57 | Day 59 | Day 61 | Day 64 | Day 67 | Day 71 | Day 73 | Day 75 | Day 78 | Day 81 | Day 101 | |
| TLR7<br>genotyping | | X | | | - N | | | | | | | | | 53 | | | <i>u</i> = = | | | | | | | v | | | | | | | | | | |
| Serum for<br>cytokine/<br>soluble<br>biomarker<br>studies <sup>i</sup> | | | x | X | | х | | х | X | | X | | х | X | | X | | X | x | | X | | x | x | | X | | x | X | | X | | X | х |
| Whole blood<br>ISG mRNA <sup>i</sup> | | 3 | X | X | . /2 | X | 2 | X | X | | X | | X | X | 1.0 | X | | X | X | | X | | X | X | | X | | X | X | | X | | X | X |
| Cell associated<br>HIV-1<br>RNA/DNA with<br>stored PBMCs <sup>i</sup> | | | х | X | | | | | | | | | | | | | E. | x | X | | | | | | | 4.5 | | x | X | | | | X | |
| Plasma HIV-1<br>RNA Single<br>Copy Assay<br>with stored<br>plasma <sup>i</sup> | | | x | x | | | | | | | | | | | | | | X | x | | | | | | | | | x | X | | | | X | |
| PBMC –<br>ELISPOT <sup>i</sup> | | X | | g: | | | -Si | | | | | | | | | | | | | | | | | | | | | x | | | | | X | |
| Whole blood –<br>immune cell<br>activation <sup>i</sup> | | | X | X | | | | | | | | | X | X | | | | | | | | | | | | | | X | X | | | | | |

| | Screena | Pre-Baseline | Dose 1b | 1300 | | | 5 | | Dose 2 | | | | p | Dose 3 | Sase | line | stud | v vis | Dose 4 | | | | | Dose 5 | d | | | | Dose 6 | , | 1 | | | End of Study | ESDD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>Procedure | Day -48 | | Day -13 | Baseline/<br>Day 1 | Day 3 | Day 5 | Day 8 | Day 11 | Day 15 | Day 17 | Day 19 | Day 22 | 25 | | Day 31 | Day 33 | Day 36 | Day 39 | 43 | Day 45 | Day 47 | Day 50 | Day 53 | Day 57 | Day 59 | Day 61 | Day 64 | Day 67 | Day 71 | Day 73 | Day 75 | Day 78 | Day 81 | Day 101 | 3.5 |
| Whole blood -<br>flow FoxP3+<br>Treg <sup>i</sup> | | | 1 | Х | | | | | | | | | | x | | | | | | | | | | | | | | | X | | | | | | |
| PBMC ICS for<br>Treg <sup>i</sup> | | | | X | X | 2.0 | 02. 0 | | | | | | | | 90 | | 2 22 | 12. 90 | | | | | | | | | 20 4.0 | 200 - 921 | X | X | | | | | 3.5 |
| Review DLTs to<br>confirm dosing<br>can proceed | | | | | 3 | , | | | X | | | | | X | | 7,0 | | | X | | | | | X | 3 | | 7,1 | | X | | | | | | |
| In-Clinic<br>Dosing <sup>j</sup> | | | 1 | х | | | | | x | | | | | X | | | | | x | | | | | X | | | | | X | | | | | | |

- Evaluation to be completed within 35 days prior to Pre-Baseline/Day -13
- b Subjects should be administered study drug after Baseline/Day 1 visit assessments (except for post-dose intensive PK)
- c All study visits are to be scheduled relative to the Baseline/Day 1 visit date.
- d Collect ART history for at least 12 months; Pre-ARV viral set point, pre-ARV CD4 nadir and historical genotype will be collected if available
- e Urogenital/anorectal exams may be performed at discretion of the Investigator
- f Symptom-directed physical examination as needed
- g Females of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test at any visit. At End of Study visit (Day 101), urine pregnancy test only performed if not done within past 30 days.
- h Details of pharmacokinetic blood sampling procedures and sample management for all PK samples in the study will be documented in the Pharmacokinetic Sample Collection, Processing, Storage, and Shipment Manual.
- i To be collected pre-dose on dosing days
- On dosing days, study drug should be taken with approximately 240 mL of water on an empty stomach. Food will not be permitted between at least 2 hours prior to and until 2 hours after dosing. Aside from the 240 mL of water provided at dosing, water/liquids will not be permitted from 1 hour prior to until 2 hours after dosing. If subjects eat prior to the 2 hour fasting period before study drug dosing, no more than a light meal should be eaten (as described in the PK Sample Collection, Processing, Storage, and Shipment Manual).

## **Study Procedures Table (Cohort 4)**

| | Screena | Pre-Baseline | Dose 1 <sup>b</sup> | | | | Dose 2 | | Dose 3 | | Dose 4 | | Dose 5 | | | | Dose 6 | | Dose 7 | | Dose 8 | | Dose 9 | | Dose 10 | | | | End of Study | ESDD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 7 | | 14 195T | | P 7 | | D 93 | | P 2 | | Post- | Basel | ine | stud | y vis | its <sup>c</sup> | | e | | 2 | | | | | | | | |
| Study Procedure | Day -48 | Day -13 | Baseline/ | Day 2 | Day 3 | Day 8 | Day 15 | Day 22 | Day 29 | Day 36 | Day 43 | Day 50 | Day 57 | Day 58 | Day 59 | Day 64 | Day 71 | Day 78 | Day 85 | Day 92 | 66 ÅeQ | Day 106 | Day 113 | Day 120 | Day 127 | Day 128 | Day 129 | Day 134 | Day 157 | |
| Informed Consent | X | | | | | | | | | | | | | | | | | | | | | | | Jally | | | 12. | | | |
| Review I/E Criteria | | X | | | | | | | | | | | | | 5 7 | | | | | | | | | | | | | | | |
| Medical History <sup>d</sup> | X | X | X | | | | | | | | | | | | (45 - 55)<br>(42 - 55) | 1 | | 14 | 10 | (V ) | 9 | | 9 | | | | | | | |
| AEs and Con Meds | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х | X | X | X | X | X | X | X | х | X | X | X | X | X | X | X |
| Complete Physical Exame | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Symptom Directed Physical Exam <sup>f</sup> | | X | X | X | X | X | X | X | x | X | x | X | X | X | X | X | x | X | x | X | X | X | X | X | X | X | X | X | X | X |
| 12-Lead ECG<br>(performed supine) | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Vital Signs | X | | X | | | | X | | X | | X | | X | | (42 - 53) | | X | ry . | X | | X | | X | | X | | | | | |
| Weight | X | | X | | | | | | | | | | | | | | | | | | | | | | | | | | X | X |
| Height | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | | | | | | | | | П | | | | |
| Plasma HIV-1 RNA | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CD4+ cell count | X | | X | | | | X | | X | | X | X | X | | | X | X | X | X | X | X | | X | X | X | | | X | X | X |
| Chemistry profile | X | | X | | | | X | | X | | X | X | X | | | X | X | X | X | X | X | | X | X | X | | | X | X | X |
| Hematology profile | X | | X | | | | X | | X | | X | X | X | | | X | X | X | X | X | X | | X | X | X | | | X | X | X |
| HBV/HCV Serology | X | | | | | | | | | | | | | | | | | | | | | | | | | П | | | | |

| | | line | 10 01 | | 1. 31 | | | | 2 | | | | | | 91 10 | | | | | | | | | | | | | | udy | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | Pre-Baseline | Dose 1b | | | | Dose 2 | | Dose 3 | | Dose 4 | | Dose 5 | | | | Dose 6 | | Dose 7 | | Dose 8 | | Dose 9 | | Dose 10 | | | | End of Study | ESDD |
| | | | 0 | 5 | 3 | | | | × × | | | | Post-l | Basel | ine | stud | y vis | its <sup>c</sup> | | | | | | | 3 | | | | | .es 9 |
| Study Procedure | Day -48 | Day -13 | Baseline/<br>Day 1 | Day 2 | Day 3 | Day 8 | Day 15 | Day 22 | Day 29 | Day 36 | Day 43 | Day 50 | Day 57 | Day 58 | Day 59 | Day 64 | Day 71 | Day 78 | Day 85 | Day 92 | Day 99 | Day 106 | Day 113 | Day 120 | Day 127 | Day 128 | Day 129 | Day 134 | Day 157 | |
| Estimated GFR | X | | X | | | | | | | | | | | | | | | | | | | | | | | | | | X | X |
| Urinalysis | X | | X | | | | X | | X | | X | X | X | | | X | X | X | X | X | X | | X | X | X | | | X | X | X |
| Serum Pregnancy Testg | X | | | | | | | | | | | | | | | | | čr | | | | ē | | | | | | | | |
| Urine Pregnancy Test <sup>g</sup> | | | X | | | | X | | X | | X | | X | | | | X | (f | X | | X | 65 - 1<br>62 - 1 | X | | X | | | | X | X |
| Plasma GS-9620 Intensive<br>PK <sup>h</sup> | | | X | | X | | | | | | | | | | | | | | | | | | | | | | | | | |
| TLR7 genotyping | 2 | X | | | | | | | | | | | | | 20 20 | | | 300 | | 35. | | 8 8 | | 100 C | | | | | | 25 2 |
| Serum for cytokine/<br>soluble biomarker studies | | | Xi | X | X | X | | | | | | | Xi | X | X | X | | | | | | | | | Xi | х | X | X | | X |
| Whole blood ISG mRNA | | | Xi | X | X | X | | | | | | | Xi | X | X | X | | | | | | | | | Xi | X | X | X | $\Box$ | X |
| Cell associated HIV-1<br>RNA/DNA with stored<br>PBMCs | | | Xi | | X | | | | | | | | Xi | | Х | | | | | | | | | | Xi | | X | | X | |
| Plasma HIV-1 RNA Single<br>Copy Assay with stored<br>plasma | | | Xi | | X | | | | | | | | Xi | | X | | | | | | | | | | Xi | | X | | X | |
| PBMC – ELISPOT | | X | | | | | | | | | | | | | | | | 5 | | 8 | | 02 | | | | | | | X | 34 3<br>5 3 |
| Whole blood – immune cell activation | 5 | | Xi | X | X | | | | | | | | Xi | X | X | | | | * | | | | *** | | Xi | X | X | | | |
| Whole blood - flow FoxP3+<br>Treg | | | Xi | | | | | | | | | | Xi | | | | | | | | | | | | Xi | | | | | |
| T cell ICS | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | X | |

| | Screena | Pre-Baseline | Dose 1b | | | | | Dose 2 | | Dose 3 | | Dose 4 | | Post-I | Basel | ine | stud | y visi | | Dose 7 | | Dose 8 | | Dose 9 | | Dose 10 | | | | End of Study | ESDD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Day -48 | Day -13 | Baseline/ | Dav 1 | Day 2 | Day 3 | Day 8 | Day 15 | Day 22 | Day 29 | Day 36 | Day 43 | Day 50 | Day 57 | Day 58 | Day 59 | Day 64 | Day 71 | Day 78 | Day 85 | Day 92 | Day 99 | Day 106 | Day 113 | Day 120 | Day 127 | Day 128 | Day 129 | Day 134 | Day 157 | |
| HIV reservoir measurement | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | X | A |
| Future Biomarker/Virology analysis Blood Sample | | X | | - 60 | | | | | | | | | | | 7. | 07 73 | | | 25 | * | | | | | | | | | | X | |
| Review DLTs to confirm dosing can proceed | | | | | | | | X | | X | | X | | X | | | | X | | X | | X | | X | | X | | | | | |
| In-Clinic Dosing <sup>j</sup> | | | X | | | | | X | | X | | X | | X | | | | X | | X | | X | | X | | X | | | | | |

- a Evaluation to be completed within 35 days prior to Pre-Baseline/Day -13
- b Subjects should be administered study drug after Baseline/Day 1 visit assessments (except for post-dose intensive PK)
- c All study visits are to be scheduled relative to the Baseline/Day 1 visit date
- d Collect ART history for at least 12 months; Pre-ARV viral set point, pre-ARV CD4 nadir and historical genotype will be collected if available
- e Urogenital/anorectal exams may be performed at discretion of the Investigator
- f Symptom-directed physical examination as needed
- g Females of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test at any visit. At End of Study visit (Day 157), urine pregnancy test only performed if not done within past 30 days.
- h Details of pharmacokinetic blood sampling procedures and sample management for all PK samples in the study will be documented in the Pharmacokinetic Sample Collection, Processing, Storage, and Shipment Manual
- i To be collected pre-dose on dosing days
- j On dosing days, study drug should be taken with approximately 240 mL of water on an empty stomach. Food will not be permitted between at least 2 hours prior to and until 2 hours after dosing. Aside from the 240 mL of water provided at dosing, water/liquids will not be permitted from 1 hour prior to until 2 hours after dosing. If subjects eat prior to the 2 hour fasting period before study drug dosing, no more than a light meal should be eaten (as described in the PK Sample Collection, Processing, Storage, and Shipment Manual).

## Study Procedures Table (Cohorts 5 to 9)<sup>a</sup>

| Study 110ccuure | 3 1 | ant | 10 | UII | or t. | , , | | , | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scree | PreBaselin | Dose | Day 1 Post E | Day 2 Post E | Day 7 Post E | Dose | Day 7 Post L | Dose | Day 2 Post E | Day 7 Poos | Dosed | Day 2 Post E | Day 7 Post E | Dos | | | | 2// | | | Dose | Day 2 Post L | Day 7 Post L | Dose | Day 2 Post L | Day 7 Post L | Dose | Day 2 Post E | Day 7 Post L | Dose 1 | Day 1 Post L | Day 2 Post L | Day 7 Post E | End of Stu | Ecni |
| | | 2 70 | | _ | | | . 6 | K 5 | | | | ľ | | | | Post | -Ba | selir | ie st | udy | visit | Se | | 12 - 25 | e o | | | | .1 | 4 4 | | | | | Ta a | F |
| Study Procedure <sup>a</sup> | Day-48 | Day-13 | Baselin | Day | Day | Day | Day 1 | Day 2 | Day 2 | Day 3 | Day 3 | Day43 | Day 4 | Day 5 | Day 5 | Day 5 | Day 5 | Day 6 | Day 7 | Day 7 | Day 7 | Day 8 | Day 8 | Day 9 | Day 9 | Day 10 | Day 10 | Day 11 | Day 11 | Day 12 | Day 12 | Day 12 | Day 12 | Day 13 | Day 15 | |
| Informed Consent | X | 3 - 15 | | | | | | | | | V | | | | | | 7.00 | | | | | | | | | | | | 20 | | | | 7 721 | | | |
| Review I/E Criteria | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Medical History <sup>f</sup> | X | X | X | | | | | 2, | | | | | 2 0 | | | | | | 7. 7 | | | | | | | | | | | | | | | | 10 0 | |
| AEs and Con Meds | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Complete Physical<br>Exam <sup>g</sup> | X | 10 1.0 | | | | | | 03. W | | | | | | | | | | (d 20 | | | | | | 26 | | | | | | 35 53 | | | | | | 0.5 |
| Symptom Directed<br>Physical Exam <sup>h</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-Lead ECG<br>(performed supine) | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Vital Signs | X | | X | | | | X | | X | | | X | | | X | | | | X | | | X | | | X | | | X | | | X | | | | | |
| Weight | X | S - 19 | X | | | | | 4 | | | | | | | | | | 0 45 | | | | | | o | | | | | | | | | | | X | X |
| Height | X | £ 2 | | | | | 70 10 | a c | | | | | | 3.5 | | | | | | | | | | 2 3 | | | | | 1 | | e: 3 | | | | 71 2 | |
| Randomization | | X | | | | | | | | | | | | | | | | | | | | | 5 | | | | | | S) | 5 6 | | | | | 6 d | |
| Stool sample for<br>microbiome analysis <sup>i</sup> | | 9 (5 | X | | | | | e e | | | | | | 2 | | | | | | | | | | | | | | | | 3 50 | | | | | X | X |
| VAS Questionnaire | | 61 | X | | | | | S* | X | | | | | | X | | | | | | | | | 9 | X | | | | | | X | | | | | S.r. |
| Plasma HIV-1 RNA | X | 25 75 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| | Scree | PreBaselin | Dose | Day 1 Post E | Day 2 Post E | Day 7 Post E | Dose | Day 7 Post L | Dose | Day 2 Post E | Day 7 PdOos | Dosed | Day 2 Post L | Day 7 Post L | Dose | _ | Ba Day 2 Post E | | Dos | | | | Day 2 Post L | Day 7 Post L | Dose | Day 2 Post L | Day 7 Post E | Dose | Day 2 Post E | Day 7 Post L | Dose 1 | Day 1 Post L | Day 2 Post E | Day 7 Post L | End of Stu | ESDI |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure <sup>a</sup> | Day48 | Day-13 | Baselin | Day | Day | Day | Day 1 | Day 2 | Day 2 | Day 3 | Day 3 | Day43 | Day 4 | Day 5 | Day 5 | | | | | | | | Day 8 | Day 9 | Day 9 | Day 1( | Day 10 | Day 11 | Day 11 | Day 12 | Day 12 | Day 12 | Day 12 | Day 13 | Day 15 | |
| CD4+ cell count,<br>CD8+ cell count,<br>CD4/CD8 ratio and<br>CD4 % | X | | x | | | | X | | X | | | X | | X | X | | | X | x | | X | X | | X | X | | | X | | X | X | | | X | X | X |
| Chemistry profile | X | | X | Xm | | | X | | X | | | X | | X | X | | Xm | X | X | Xm | X | X | Xm | X | X | Xm | | X | Xm | X | X | | Xm | X | X | X |
| Hematology profile | Х | 2 22 | X | Xm | | | X | 0. | X | | | X | | X | X | | Xm | X | X | Xm | X | X | Xm | X | X | Xm | | X | Xm | X | X | | Xm | X | X | X |
| HBV/HCV Serology | X | | | | | | | | | | | | 5 5 | | | | | | | | | | | 25 - 25 | | | | | | | | | | | 8 8 | |
| Estimated GFR | Х | 3 3 | X | | | ò | | 2 6 | 2 | | | | ē 4 | 8 | | | | 1 3 | (C. 7) | | | | | 3 4 | | 3 | | | 22 | 4 | G 2 | | | | X | X |
| Urinalysis | X | 2 - 15 | X | Xm | | | X | | X | | | X | ii - 5. | X | X | | Xm | X | X | Xm | X | X | Xm | X | X | Xm | | X | Xm | X | X | | Xm | X | X | X |
| Urine Pregnancy Test <sup>j</sup> | | | X | | | | X | | X | | | X | | | X | | | | X | | | X | | | X | | | X | | | X | | | | X | X |
| Serum Pregnancy Test <sup>j</sup> | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Plasma GS-9620<br>Intensive PK <sup>k</sup> | | v - 45 | Х | | X | | | | | | | Xn | Xn | | | | , | | | 3 | | | | | | | | | | | | | | | | g s |
| Plasma ART PKP | X | | | | | | | | X | | | | | | X | | | | | | | X | | | X | | | | | | | | | | | |
| TLR7 genotyping | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Serum for<br>cytokine/soluble<br>biomarker studies | | | Χ° | X | Х | | | | | | | Xn | Xn | Xn | Xº | X | X | X | | | | | | | | | | | | | Xº | X | X | X | | X |
| Whole blood ISG<br>mRNA | | | Xº | X | X | | | | | | | Xn | Xn | Xn | Xº | X | X | X | | | | | | | | | | | | | Xº | X | X | X | | X |

| - | | | | | | $\neg$ | | - | - | | - | | | | | | Ī | | | | | | | | | ī | $\neg$ | | | - | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scree | PreBaselin | Dose | Day 1 Post L | Day 2 Post L | Day 7 Post L | Dose | Day 7 Post L | Dose | Day 2 Post L | Day 7 Poos | Dosed | Day 2 Post I | Day 7 Post L | | | | | | | | | Day 2 Post L | Day 7 Post I | Dose | Day 2 Post L | Day 7 Post L | Dose | Day 2 Post L | Day 7 Post L | Dose 1 | Day 1 Post L | Day 2 Post I | Day 7 Post L | End of Stu | ESDI |
| | | | | | | | | | | | | | | _ | | Post | t-Ba | selir | ie st | udy | visit | se | | | | _ | _ | | | | | | | | | _ |
| Study Procedure <sup>a</sup> | Day-48 | Day-13 | Baselin<br>Dov | Day | Day | Day | Day 1 | Day 2 | Day 2 | Day 3 | Day 3 | Day43 | Day 4 | Day 5 | Day 5 | Day 5 | Day 5 | Day 6 | Day 7 | Day 7 | Day 7 | Day 8 | Day 8 | Day 9 | Day 9 | Day 1( | Day 10 | Day 11 | Day 11 | Day 12 | Day 12 | Day 12 | Day 12 | Day 13 | Day 15 | |
| Cell associated HIV-1<br>RNA/DNA<br>(CAVR/CAVD) with<br>stored PBMCs | | | Xº | | X | | | | | | | | | | Χ° | | X | | | | | | | | | | | | | | Χ° | | X | | X | |
| Plasma HIV-1 RNA<br>Single Copy Assay<br>with stored plasma | | | X° | | X | | | | | | | | | | Χ° | | X | | | | | | | | | | | | | | Χ° | | X | | X | |
| PBMC – ELISPOT <sup>i</sup> | | X | | | | | | | | | | | | | | | | | | | | | | | | | | | CI | | | | | | X | |
| Whole blood –<br>immune cell activation | | | Xº | X | X | | | | | | | | | | Xº | X | X | | | | | | | | | | | | | | Xº | X | X | | | |
| Whole blood - flow<br>FoxP3+ Treg | | | Xº | | | | | | | | | | | | Xº | | | | | | | | | | | | | | 5 | | Xº | | | | | |
| T cell ICSi | | X | | | | | | 5 6 | , | | | | 8 8 | | | | 0 | )<br>1 - 17 | e e e | | | | | | | 3 | | | | 5 5 | | | | | X | |
| HIV-1 Reservoir<br>measurement <sup>i</sup> | | X | | | | | 9 23 | 2, 19 | , y | | | | 8 | | | | | 3 3 | * C | | | | 9 | S 43 | | | | | 2 | 5 - 6 | (# % | | | | X | |
| CCI | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Review DLTs to<br>confirm dosing can<br>proceed | | | | | | | X | | X | | | X | | | X | | | | X | | | X | | | X | | | X | | | X | | | | | |
| In-Clinic Dosing <sup>1</sup> | | | X | | | | X | | X | | | X | | | X | | | | X | | | X | | | X | | ヿ | X | | | X | | | | | |

Evaluation to be completed within 35 days prior to Pre-Baseline/Day -13
Subjects should be administered study drug after Baseline/Day 1 visit assessments (except for post-dose intensive PK)

- d Dose 4 (Cohort 6 only) cannot occur until SEC completes review of the safety data from all subjects' first three doses (GS-9620 10 mg dose). If the GS-9620 10mg dose is found to be safe, Dose 4 and subsequent Doses (5-10) will escalate to GS-9620 12 mg. If dose escalation is not approved by the SEC, subjects will continue receiving 10 mg of GS-9620 or placebo from Doses 4 to 10
- e All study visits are to be scheduled relative to the Baseline/Day 1 visit date
- f Collect ART history for at least 12 months; Pre-ARV viral set point, pre-ARV CD4 nadir and historical genotype will be collected if available
- g Urogenital/anorectal exams may be performed at discretion of the Investigator
- h Symptom-directed physical examination as needed
- j Females of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test at any visit. At End of Study visit, urine pregnancy test only performed if not done within past 30 days
- k Details of pharmacokinetic blood sampling procedures and sample management for all PK samples in the study will be documented in the Pharmacokinetic Sample Collection, Processing, Storage, and Shipment Manual.
- 1 In Cohorts 5 and 6, CCI , the study drug will be administered following an overnight fast.

m Cohorts 6 only

- n Cohort 6 only, if dose escalation to 12mg is approved by SEC
- o To be collected pre-dose on dosing days
- p Cohorts 6 coloring only required at Screening, Days 57 and Days 99





Appendix 4. GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

Antiviral Toxicity Grading Scale Version: 01 April 2015

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin HIV POSITIVE Adult and Pediatric ≥ 57 Days | 8.5 to 10.0 g/dL<br>85 to 100 g/L | 7.5 to < 8.5 g/dL<br>75 to < 85 g/L | 6.5 to < 7.5 g/dL<br>65 to < 75 g/L | < 6.5 g/dL<br>< 65 g/L |
| HIV NEGATIVE Adult and Pediatric ≥ 57 Days | 10.0 to 10.9 g/dL<br>100 to 109 g/L<br>OR<br>Any decrease from Baseline<br>2.5 to < 3.5 g/dL<br>25 to < 35 g/L | 9.0 to < 10.0 g/dL<br>90 to < 100 g/L<br>OR<br>Any decrease from Baseline<br>3.5 to < 4.5 g/dL<br>35 to < 45 g/L | 7.0 to $<$ 9.0 g/dL<br>70 to $<$ 90 g/L<br>OR<br>Any decrease from Baseline<br>$\ge 4.5$ g/dL<br>$\ge 45$ g/L | < 7.0 g/dL<br>< 70 g/L |
| Infant, 36–56 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 8.5 to 9.4 g/dL<br>85 to 94 g/L | 7.0 to < 8.5 g/dL<br>70 to < 85 g/L | 6.0 to < 7.0 g/dL<br>60 to < 70 g/L | < 6.0 g/dL<br>< 60 g/L |
| Infant, 22–35 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 9.5 to 10.5 g/dL<br>95 to 105 g/L | 8.0 to < 9.5 g/dL<br>80 to < 95 g/L | 7.0 to < 8.0 g/dL<br>70 to < 80 g/L | < 7.0 g/dL<br>< 70 g/L |
| Infant, 1–21 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 12.0 to 13.0 g/dL<br>120 to 130 g/L | 10.0 to < 12.0 g/dL<br>100 to < 120 g/L | 9.0 to < 10.0 g/dL<br>90 to < 100 g/L | < 9.0 g/dL<br>< 90 g/L |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Neutrophil Count (ANC) Adult and Pediatric, ≥ 7 Months# | 1000 to 1300/mm <sup>3</sup> 1.00 to 1.30 GI/L | 750 to < 1000/mm <sup>3</sup><br>0.75 to < 1.00 GI/L | 500 to < 750/mm <sup>3</sup><br>0.50 to < 0.75 GI/L | < 500/mm <sup>3</sup><br>< 0.50 GI/L |
| Absolute CD4+ Count HIV NEGATIVE ONLY Adult and Pediatric > 13 Years | 300 to 400/mm <sup>3</sup><br>300 to 400/μL | $200 \text{ to} < 300/\text{mm}^3 \\ 200 \text{ to} < 300/\mu\text{L}$ | $100 \text{ to} < 200/\text{mm}^3$ $100 \text{ to} < 200/\mu L$ | $<100/mm^3 \\ <100/\mu L$ |
| Absolute Lymphocyte Count HIV NEGATIVE ONLY Adult and Pediatric > 13 Years | 600 to 650/mm <sup>3</sup><br>0.60 to 0.65 GI/L | 500 to < 600/mm <sup>3</sup><br>0.50 to < 0.60 GI/L | 350 to < 500/mm <sup>3</sup><br>0.35 to < 0.50 GI/L | < 350/mm <sup>3</sup><br>< 0.35 GI/L |
| Platelets | 100,000 to < 125,000/mm <sup>3</sup><br>100 to < 125 GI/L | 50,000 to < 100,000/mm <sup>3</sup><br>50 to < 100 GI/L | 25,000 to < 50,000/mm <sup>3</sup><br>25 to < 50 GI/L | < 25,000/mm <sup>3</sup><br>< 25 GI/L |
| WBCs | 2000/mm <sup>3</sup> to 2500/mm <sup>3</sup><br>2.00 GI/L to 2.50 GI/L | 1,500 to < 2,000/mm <sup>3</sup><br>1.50 to < 2.00 GI/L | 1000 to < 1,500/mm <sup>3</sup><br>1.00 to < 1.50 GI/L | < 1000/mm <sup>3</sup><br>< 1.00 GI/L |
| Hypofibrinogenemia | 100 to 200 mg/dL<br>1.00 to 2.00 g/L | 75 to < 100 mg/dL<br>0.75 to < 1.00 g/L | 50 to < 75 mg/dL<br>0.50 to < 0.75 g/L | < 50 mg/dL<br>< 0.50 g/L |
| Hyperfibrinogenemia | > ULN to 600 mg/dL<br>> ULN to 6.0 g/L | > 600 mg/dL<br>> 6.0 g/L | | |
| Fibrin Split Product | 20 to 40 μg/mL<br>20 to 40 mg/L | > 40 to 50 μg/mL<br>> 40 to 50 mg/L | > 50 to 60 μg/mL<br>> 50 to 60 mg/L | > 60 μg/mL<br>> 60 mg/L |
| Prothrombin Time (PT) | > 1.00 to 1.25 × ULN | > 1.25 to 1.50 × ULN | > 1.50 to 3.00 × ULN | > 3.00 × ULN |

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| International Normalized Ratio of prothrombin time (INR) | 1.1 to 1.5 x ULN | >1.5 to 2.0 x ULN | >2.0 to 3.0 x ULN | >3.0 x ULN |
| Activated Partial Thromboplastin Time (APTT) | > 1.00 to 1.66 × ULN | > 1.66 to 2.33 × ULN | > 2.33 to 3.00 × ULN | > 3.00 × ULN |
| Methemoglobin | 5.0 to 10.0% | > 10.0 to 15.0% | > 15.0 to 20.0% | > 20.0% |

<sup>#</sup> An overlap between the Grade 1 scale and the Lab's normal range for absolute neutrophils may result for pediatric subjects. Please follow the Gilead convention of grading any result within the LLN and ULN a 0.
| | | CHEMISTRY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to <lln l<="" meq="" td=""><td>125 to &lt; 130 mEq/L</td><td>121 to &lt; 125 mEq/L</td><td>&lt; 121 mEq/L</td></lln> | 125 to < 130 mEq/L | 121 to < 125 mEq/L | < 121 mEq/L |
| | 130 to <lln l<="" mmol="" td=""><td>125 to &lt; 130 mmol/L</td><td>121 to &lt; 125 mmol/L</td><td>&lt; 121 mmol/L</td></lln> | 125 to < 130 mmol/L | 121 to < 125 mmol/L | < 121 mmol/L |
| Hypernatremia | >ULN to 150 mEq/L | > 150 to 154 mEq/L | > 154 to 159 mEq/L | > 159 mEq/L |
| | >ULN to 150 mmol/L | > 150 to 154 mmol/L | > 154 to 159 mmol/L | > 159 mmol/L |
| Hypokalemia | 3.0 to <lln l<="" meq="" td=""><td>2.5 to &lt; 3.0 mEq/L</td><td>2.0 to &lt; 2.5 mEq/L</td><td>&lt; 2.0 mEq/L</td></lln> | 2.5 to < 3.0 mEq/L | 2.0 to < 2.5 mEq/L | < 2.0 mEq/L |
| Adult and Pediatric | 3.0 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.0 mmol/L</td><td>2.0 to &lt; 2.5 mmol/L</td><td>&lt; 2.0 mmol/L</td></lln> | 2.5 to < 3.0 mmol/L | 2.0 to < 2.5 mmol/L | < 2.0 mmol/L |
| ≥1 Year | | | | |
| Infant <1 Year | 3.0 to 3.4 mEq/L | 2.5 to < 3.0 mEq/L | 2.0 to < 2.5 mEq/L | < 2.0 mEq/L |
| | 3.0 to 3.4 mmol/L | 2.5 to <3.0 mmolL | 2.0 t o <2.5 mmolL | <2.0 mmolL |
| Hyperkalemia | 5.6 to 6.0 mEq/L | > 6.0 to 6.5 mEq/L | > 6.5 to 7.0 mEq/L | > 7.0 mEq/L |
| Adult and Pediatric | 5.6 to 6.0 mmol/L | > 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mmol/L | > 7.0 mmol/L |
| ≥1 Year | | | | |
| Infant <1 Year | >ULN to 6.0 mEq/L | > 6.0 to 6.5 mEq/L | > 6.5 to 7.0 mEq/L | > 7.0 mEq/L |
| | >ULN to 6.0 mmol/L | > 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mmol/L | > 7.0 mmol/L |
| Hypoglycemia | 55 to 64 mg/dL | 40 to < 55 mg/dL | 30 to < 40 mg/dL | < 30 mg/dL |
| Adult and Pediatric | 3.03 to 3.58 mmol/L | 2.20 to < 3.03 mmol/L | 1.64 to < 2.20 mmol/L | < 1.64 mmol/L |
| ≥ 1 Month | | | | |
| Infant, < 1 Month | 50 to 54 mg/dL | 40 to < 50 mg/dL | 30 to < 40 mg/dL | < 30 mg/dL |
| | 2.8 to 3.0 mmol/L | 2.2 to < 2.8 mmol/L | 1.7 to < 2.2 mmol/L | < 1.7 mmol/L |
| Hyperglycemia, Nonfasting | 116 to 160 mg/dL | > 160 to 250 mg/dL | > 250 to 500 mg/dL | > 500 mg/dL |
| | 6.42 to 8.91 mmol/L | > 8.91 to 13.90 mmol/L | > 13.90 to 27.79 mmol/L | > 27.79 mmol/L |
| Hyperglycemia, Fasting | 110 to 125 mg/dL | >125 to 250 mg/dL | >250 to 500 mg/dL | >500 mg/dL |
| | 6.08 to 6.96 mmol/L | >6.96 to 13.90 mmol/L | >13.90 to 27.79 mmol/L | >27.79 mmol/L |
| Hypocalcemia | 7.8 <lln dl<="" mg="" td=""><td>7.0 to &lt; 7.8 mg/dL</td><td>6.1 to &lt; 7.0 mg/dL</td><td>&lt; 6.1 mg/dL</td></lln> | 7.0 to < 7.8 mg/dL | 6.1 to < 7.0 mg/dL | < 6.1 mg/dL |
| (corrected for albumin if | 1.94 to <lln l<="" mmol="" td=""><td>1.74 to &lt; 1.94 mmol/L</td><td>1.51 to &lt; 1.74 mmol/L</td><td>&lt; 1.51 mmol/L</td></lln> | 1.74 to < 1.94 mmol/L | 1.51 to < 1.74 mmol/L | < 1.51 mmol/L |
| appropriate*) | | | | |
| Adult and Pediatric | | | | |
| ≥2 Years | | | | |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Pediatric ≥7 days -2 Years | 7.8 to 8.4 mg/dL | 7.0 to <7.8 mg/dL | 6.1 to <7.0 mg/dL | < 6.1 mg/dL |
| | 1.94 to 2.10 mmol/L | 1.74 to <1.94 mmolL | 1.51 to < 1.74 mmolL | < 1.51 mmol/L |
| Infant, < 7 Days | 6.5 to 7.5 mg/dL | 6.0 to < 6.5 mg/dL | 5.5 to < 6.0 mg/dL | < 5.5 mg/dL |
| | 1.61 to 1.88 mmol/L | 1.49 to < 1.61 mmol/L | 1.36 to < 1.49 mmol/L | < 1.36 mmol/L |
| Hypercalcemia (corrected | | | | |
| for albumin if appropriate*) | >ULN to 11.5 mg/dL | > 11.5 to 12.5 mg/dL | > 12.5 to 13.5 mg/dL | > 13.5 mg/dL |
| Adult and Pediatric ≥<br>7 Days | >ULN to 2.88 mmol/L | > 2.88 to 3.13 mmol/L | > 3.13 to 3.38 mmol/L | > 3.38 mmol/L |
| Infant, < 7 Days | 11.5 to 12.4 mg/dL | > 12.4 to 12.9 mg/dL | > 12.9 to 13.5 mg/dL | > 13.5 mg/dL |
| | 2.86 to 3.10 mmol/L | > 3.10 to 3.23 mmol/L | > 3.23 to 3.38 mmol/L | > 3.38 mmol/L |
| Hypocalcemia (ionized) | 3.0 mg/dL to < LLN | 2.5 to < 3.0 mg/dL | 2.0 to < 2.5 mg/dL | < 2.0 mg/dL |
| | 0.74 mmol/L to < LLN | 0.62 to < 0.74 mmol/L | 0.49 to < 0.62 mmol/L | < 0.49 mmol/L |
| Hypercalcemia (ionized) | > ULN to 6.0 mg/dL | > 6.0 to 6.5 mg/dL | > 6.5 to 7.0 mg/dL | > 7.0 mg/dL |
| | > ULN to 1.50 mmol/L | > 1.50 to 1.63 mmol/L | > 1.63 to 1.75 mmol/L | > 1.75 mmol/L |
| Hypomagnesemia | 1.40 to <lln dl<="" mg="" td=""><td>1.04 to &lt; 1.40 mg/dL</td><td>0.67 to &lt; 1.04 mg/dL</td><td>&lt; 0.67 mg/dL</td></lln> | 1.04 to < 1.40 mg/dL | 0.67 to < 1.04 mg/dL | < 0.67 mg/dL |
| | 1.2 to <lln l<="" meq="" td=""><td>0.9 to &lt; 1.2 mEq/L</td><td>0.6 to &lt; 0.9 mEq/L</td><td>&lt; 0.6 mEq/L</td></lln> | 0.9 to < 1.2 mEq/L | 0.6 to < 0.9 mEq/L | < 0.6 mEq/L |
| | 0.58 to <lln l<="" mmol="" td=""><td>0.43 to &lt; 0.58 mmol/L</td><td>0.28 to &lt; 0.43 mmol/L</td><td>&lt; 0.28 mmol/L</td></lln> | 0.43 to < 0.58 mmol/L | 0.28 to < 0.43 mmol/L | < 0.28 mmol/L |
| Hypophosphatemia | | | | |
| Adult and Pediatric | 2.0 to < LLN mg/dL | 1.5 to < 2.0 mg/dL | 1.0 to < 1.5 mg/dL | < 1.0 mg/dL |
| > 14 Years | 0.63 to < LLN mmol/L | 0.47 to < 0.63 mmol/L | 0.31 to < 0.47 mmol/L | < 0.31 mmol/L |
| Pediatric 1 Year–14 Years | 3.0 to <lln dl<="" mg="" td=""><td>2.5 to &lt; 3.0 mg/dL</td><td>1.5 to &lt; 2.5 mg/dL</td><td>&lt; 1.5 mg/dL</td></lln> | 2.5 to < 3.0 mg/dL | 1.5 to < 2.5 mg/dL | < 1.5 mg/dL |
| roundle i ioni i i ioni | 0.96 to <lln l<="" mmol="" td=""><td>0.80 to &lt; 0.96 mmol/L</td><td>0.47 to &lt; 0.80 mmol/L</td><td>&lt; 0.47 mmol/L</td></lln> | 0.80 to < 0.96 mmol/L | 0.47 to < 0.80 mmol/L | < 0.47 mmol/L |
| Pediatric < 1 Year | 3.5 to <lln dl<="" mg="" td=""><td>2.5 to &lt; 3.5 mg/dL</td><td>1.5 to &lt; 2.5 mg/dL</td><td>&lt; 1.5 mg/dL</td></lln> | 2.5 to < 3.5 mg/dL | 1.5 to < 2.5 mg/dL | < 1.5 mg/dL |
| | 1.12 to <lln l<="" mmol="" td=""><td>0.80 to &lt; 1.12 mmol/L</td><td>0.47 to &lt; 0.80 mmol/L</td><td>&lt; 0.47 mmol/L</td></lln> | 0.80 to < 1.12 mmol/L | 0.47 to < 0.80 mmol/L | < 0.47 mmol/L |

| | CHEMISTRY | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyperbilirubinemia Adult and Pediatric > 14 Days | > 1.0 to 1.5 × ULN | > 1.5 to 2.5 × ULN | > 2.5 to 5.0 × ULN | > 5.0 × ULN |
| Infant, ≤ 14 Days (non-hemolytic) | NA | 20.0 to 25.0 mg/dL<br>342 to 428 μmol/L | > 25.0 to 30.0 mg/dL<br>> 428 to 513 μmol/L | > 30.0 mg/dL<br>> 513 μmol/L |
| Infant, ≤ 14 Days (hemolytic) | NA | NA | 20.0 to 25.0 mg/dL<br>342 to 428 μmol/L | > 25.0 mg/dL<br>> 428 μmol/L |
| Blood Urea Nitrogen | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Hyperuricemia | >ULN to 10.0 mg/dL<br>>ULN to 597 μmol/L | > 10.0 to 12.0 mg/dL<br>> 597 to 716 μmol/L | > 12.0 to 15.0 mg/dL<br>> 716 to 895 μmol/L | > 15.0 mg/dL<br>> 895 μmol/L |
| Hypouricemia Adult and Pediatric | 1.5 mg/dL to < LLN<br>87 µmol/L to < LLN | 1.0 to < 1.5 mg/dL<br>57 to < 87 μmol/L | 0.5 to < 1.0 mg/dL<br>27 to < 57 μmol/L | < 0.5 mg/dL<br>< 27 μmol/L |
| ≥1 year<br>Infant <1 Year | N/A | 1.0 mg/dl to <lln-<br>57 μmol to <lln< td=""><td>0.5 to &lt; 1.0 mg/dL<br/>27 to &lt; 57 μmol/L</td><td>&lt; 0.5 mg/dL<br/>&lt; 27 μmol/L</td></lln<></lln-<br> | 0.5 to < 1.0 mg/dL<br>27 to < 57 μmol/L | < 0.5 mg/dL<br>< 27 μmol/L |
| Creatinine** | > 1.50 to 2.00 mg/dL<br>> 133 to 177 μmol/L | > 2.00 to 3.00 mg/dL<br>> 177 to 265 μmol/L | > 3.00 to 6.00 mg/dL<br>> 265 to 530 μmol/L | > 6.00 mg/dL<br>> 530 μmol/L |
| Bicarbonate Adult and Pediatric ≥ 4 Years | 16.0 mEq/L to < LLN<br>16.0 mmol/L to < LLN | 11.0 to < 16.0 mEq/L<br>11.0 to < 16.0 mmol/L | 8.0 to < 11.0 mEq/L<br>8.0 to < 11.0 mmol/L | < 8.0 mEq/L<br>< 8.0 mmol/L |
| Pediatric < 4 Years | NA | 11.0 mEq/Lto <lln<br>11.0 mmol/L to <lln< td=""><td>8.0 to &lt; 11.0 mEq/L<br/>8.0 to &lt; 11.0 mmol/L</td><td>&lt; 8.0 mEq/L<br/>&lt; 8.0 mmol/L</td></lln<></lln<br> | 8.0 to < 11.0 mEq/L<br>8.0 to < 11.0 mmol/L | < 8.0 mEq/L<br>< 8.0 mmol/L |
| Triglycerides (Fasting) | NA | 500 to 750 mg/dL<br>5.64–8.47 mmol/L | > 750 to 1200 mg/dL<br>> 8.47–13.55 mmol/L | > 1200 mg/dL<br>> 13.55 mmol/L |

| CHEMISTRY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| LDL (Fasting) | 130 to 160 mg/dL | >160 to 190 mg/dL | > 190 mg/dL | NA |
| Adult | 3.35 to 4.15 mmol/L | >4.15 to 4.92 mmol/L | >4.92 mmol/L | |
| LDL (Fasting) | 110 to 130 mg/dL | >130 to 190 mg/dL | > 190 mg/dL | NA |
| Pediatric >2 to <18 years | 2.84 to 3.37 mmol/L | >3.37 to 4.92 mmol/L | >4.92 mmol/L | |
| Hypercholesterolemia | 200 to 239 mg/dL | > 239 to 300 mg/dL | > 300 mg/dL | NA |
| (Fasting) | 5.16 to 6.19 mmol/L | > 6.19 to 7.77 mmol/L | > 7.77 mmol/L | |
| Pediatric < 18 Years | 170 to 199 mg/dL<br>4.39 to 5.15 mmol/L | > 199 to 300 mg/dL<br>> 5.15 to 7.77 mmol/L | > 300 mg/dL<br>> 7.77 mmol/L | NA |
| Creatine Kinase | 3.0 to < 6.0 × ULN | 6.0 to < 10.0 × ULN | 10.0 to < 20.0 × ULN | ≥ 20.0 × ULN |

Calcium should be corrected for albumin if albumin is < 4.0 g/dLAn overlap between the Grade 1 scale and the Lab's normal range for creatinine may result for Male subjects > 70 yrs. Please follow the Gilead convention of grading any result within the LLN and ULN a 0.

| | | <b>ENZYMES</b> | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| ALT (SGPT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| GGT | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Alkaline Phosphatase | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Total Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Pancreatic Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Lipase | > 1.0 to 1.5 × ULN | > 1.5 to 3.0 × ULN | > 3.0 to 5.0 × ULN | > 5.0 × ULN |
| Albumin Pediatrics <16 years | - | 2.0 to < LLN g/dL<br>20 to < LLN g/L | < 2.0 g/dL<br>< 20 g/L | NA |
| ≥ 16 years | 3.0 g/dL to < LLN<br>30 g/L to < LLN | 2.0 to < 3.0 g/dL<br>20 to < 30 g/L | < 2.0 g/dL<br>< 20 g/L | NA |

| URINALYSIS | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hematuria (Dipstick) | 1+ | 2+ | 3-4+ | NA |
| Hematuria (Quantitative)<br>See Note below | | | | |
| Females | >ULN - 10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Males | 6-10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Proteinuria (Dipstick) | 1+ | 2–3+ | 4+ | NA |
| Proteinuria, 24 Hour Collection Adult and Pediatric ≥ 10 Years | 200 to 999 mg/24 h | >999 to 1999 mg/24 h | >1999 to 3500 mg/24 h | > 3500 mg/24 h |
| Pediatric > 3 Mo to<br>< 10 Years | 201 to 499 mg/m <sup>2</sup> /24 h | >499 to 799 mg/m <sup>2</sup> /24 h | >799 to 1000 mg/m <sup>2</sup> /24 h | > 1000 mg/ m <sup>2</sup> /24 h |
| Glycosuria (Dipstick) | 1+ | 2-3+ | 4+ | NA |

#### Notes:

- Toxicity grades for Quantitative and Dipstick Hematuria will be assigned by Covance Laboratory, however for other laboratories, toxicity grades will only be assigned to Dipstick Hematuria.
- With the exception of lipid tests, any graded laboratory test with a result that is between the LLN and ULN should be assigned Grade 0.
- If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE.

| | | CARDIOVASCULAR | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Arrhythmia (general)<br>(By ECG or physical exam) | Asymptomatic AND No intervention indicated | Asymptomatic AND Non-<br>urgent medical intervention<br>indicated | Symptomatic, non-life-<br>threatening AND Non-<br>urgent medical intervention<br>indicated | Life-threatening arrhythmia OR Urgent intervention indicated |
| Cardiac-ischemia/Infarction | NA | NA | Symptomatic ischemia (stable angina) OR Testing consistent with ischemia | Unstable angina OR Acute myocardial infarction |
| Hemorrhage (significant acute blood loss) | NA | Symptomatic AND No transfusion indicated | Symptomatic AND Transfusion of ≤ 2 units packed RBCs (for children ≤ 10 cc/kg) indicated | Life-threatening hypotension<br>OR Transfusion of > 2 units<br>packed RBCs indicated (for<br>children ≤ 10 cc/kg) indicated |
| Hypertension (with repeat testing at same visit) | 140–159 mmHg systolic<br>OR<br>90–99 mmHg diastolic | > 159–179 mmHg systolic<br>OR<br>> 99–109 mmHg diastolic | > 179 mmHg systolic<br>OR<br>> 109 mmHg diastolic | Life-threatening consequences<br>(eg, malignant hypertension)<br>OR Hospitalization (other than<br>ER visit) indicated |
| Pediatric ≤ 17 Years (with repeat testing at same visit) | NA | 91st–94th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | ≥ 95th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | Life-threatening consequences<br>(eg, malignant hypertension)<br>OR Hospitalization indicated<br>(other than emergency room<br>visit) |
| Hypotension | NA | Symptomatic, corrected with oral fluid replacement | Symptomatic, IV fluids indicated | Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Pericardial Effusion | Asymptomatic, small effusion requiring no intervention | Asymptomatic, moderate or larger effusion requiring no intervention | Effusion with non-life-<br>threatening physiologic<br>consequences OR Effusion<br>with nonurgent intervention<br>indicated | Life-threatening consequences<br>(eg, tamponade) OR Urgent<br>intervention indicated |
| Prolonged PR Interval | PR interval 0.21 to 0.25 sec | PR interval > 0.25 sec | Type II 2nd degree AV<br>block OR Ventricular pause<br>> 3.0 sec | Complete AV block |

| | | CARDIOVASCULAR | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Pediatric ≤ 16 Years | 1st degree AV block<br>(PR > normal for age and<br>rate) | Type I 2nd degree AV block | Type II 2nd degree AV block | Complete AV block |
| Prolonged QTc | Asymptomatic, QTc interval 0.45 to 0.47 sec OR Increase interval < 0.03 sec above baseline | Asymptomatic, QTc interval 0.48 to 0.49 sec OR Increase in interval 0.03 to 0.05 sec above baseline | Asymptomatic, QTc interval ≥ 0.50 sec OR Increase in interval ≥ 0.06 sec above baseline | Life-threatening consequences, eg, Torsade de pointes or other associated serious ventricular dysrhythmia |
| Pediatric ≤ 16 Years | Asymptomatic, QTc interval 0.450 to 0.464 sec | Asymptomatic, QTc interval 0.465 to 0.479 sec | Asymptomatic, QTc interval ≥ 0.480 sec | Life-threatening consequences, eg, Torsade de pointes or other associated serious ventricular dysrhythmia |
| Thrombosis/Embolism | NA | Deep vein thrombosis AND<br>No intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Deep vein thrombosis AND<br>Intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Embolic event (eg, pulmonary embolism, life-threatening thrombus) |
| Vasovagal Episode (associated with a procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | NA | NA |
| Ventricular Dysfunction<br>(congestive heart failure,<br>CHF) | NA | Asymptomatic diagnostic finding AND intervention indicated | New onset with symptoms<br>OR Worsening symptomatic<br>CHF | Life-threatening CHF |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bronchospasm (acute) | FEV1 or peak flow reduced to 70% to 80% | FEV1 or peak flow 50% to 69% | FEV1 or peak flow 25% to 49% | Cyanosis OR FEV1 or peak flow < 25% OR Intubation |
| Dyspnea or Respiratory<br>Distress | Dyspnea on exertion with no or minimal interference with usual social & functional activities | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities | Dyspnea at rest causing inability to perform usual social & functional activities | Respiratory failure with ventilatory support indicated |
| Pediatric < 14 Years | Wheezing OR minimal increase in respiratory rate for age | Nasal flaring OR Intercostal retractions OR Pulse oximetry 90% to 95% | Dyspnea at rest causing inability to perform usual social & functional activities OR Pulse oximetry < 90% | Respiratory failure with ventilatory support indicated |

| OCULAR/VISUAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Uveitis | Asymptomatic but detectable on exam | Symptomatic anterior uveitis OR<br>Medical intervention indicated | Posterior or pan-uveitis OR<br>Operative intervention<br>indicated | Disabling visual loss in affected eye(s) |
| Visual Changes (from baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |

| | | SKIN | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alopecia | Thinning detectable by study participant or caregiver (for disabled adults) | Thinning or patchy hair loss detectable by health care provider | Complete hair loss | NA |
| Cutaneous Reaction – Rash | Localized macular rash | Diffuse macular,<br>maculopapular, or<br>morbilliform rash OR Target<br>lesions | Diffuse macular,<br>maculopapular, or morbilliform<br>rash with vesicles or limited<br>number of bullae OR<br>Superficial ulcerations of<br>mucous membrane limited to<br>one site | Extensive or generalized<br>bullous lesions OR<br>Stevens-Johnson syndrome<br>OR Ulceration of mucous<br>membrane involving two<br>or more distinct mucosal<br>sites OR Toxic epidermal<br>necrolysis (TEN) |
| Hyperpigmentation | Slight or localized | Marked or generalized | NA | NA |
| Hypopigmentation | Slight or localized | Marked or generalized | NA | NA |
| Pruritis (itching – no skin lesions) (See also Injection Site Reactions: Pruritis associated with injection) | Itching causing no or<br>minimal interference with<br>usual social & functional<br>activities | Itching causing greater than minimal interference with usual social & functional activities | Itching causing inability to perform usual social & functional activities | NA |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite associated with decreased oral intake without significant weight loss | Loss of appetite associated with significant weight loss | Life-threatening consequences<br>OR Aggressive intervention<br>indicated [eg, tube feeding or<br>total parenteral nutrition] |
| Ascites | Asymptomatic | Symptomatic AND Intervention indicated (eg, diuretics or therapeutic paracentesis) | Symptomatic despite intervention | Life-threatening consequences |
| Cholecystitis | NA | Symptomatic AND Medical intervention indicated | Radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences (eg, sepsis or perforation) |
| Constipation | NA | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (eg, obstruction) |
| Diarrhea | | | | |
| Adult and Pediatric<br>≥ 1 Year | Transient or intermittent episodes of unformed stools OR Increase of $\leq 3$ stools over baseline/24 hr | Persistent episodes of unformed<br>to watery stools OR Increase of<br>4–6 stools over baseline per<br>24 hrs. | Bloody diarrhea OR Increase<br>of ≥ 7 stools per 24-hour<br>period OR IV fluid<br>replacement indicated | Life-threatening consequences (eg, hypotensive shock) |
| Pediatric < 1 Year | Liquid stools (more<br>unformed than usual) but<br>usual number of stools | Liquid stools with increased<br>number of stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Liquid stools resulting in<br>severe dehydration with<br>aggressive rehydration<br>indicated OR Hypotensive<br>shock |
| Dysphagia-Odynophagia | Symptomatic but able to eat usual diet | Symptoms causing altered dietary intake without medical intervention indicated | Symptoms causing severely altered dietary intake with medical intervention indicated | Life-threatening reduction in oral intake |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucositis/Stomatitis<br>(clinical exam)<br>See also Proctitis,<br>Dysphagia-Odynophagia | Erythema of the mucosa | Patchy pseudomembranes or ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Tissue necrosis OR Diffuse<br>spontaneous mucosal bleeding<br>OR Life-threatening<br>consequences (eg, aspiration,<br>choking) |
| Nausea | Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake | Persistent nausea resulting in decreased oral intake for 24–48 hours | Persistent nausea resulting in minimal oral intake for > 48 hours OR Aggressive rehydration indicated (eg, IV fluids) | Life-threatening consequences (eg, hypotensive shock) |
| Pancreatitis | NA | Symptomatic AND Hospitalization not indicated (other than ER visit) | Symptomatic AND<br>Hospitalization indicated<br>(other than ER visit) | Life-threatening consequences (eg, sepsis, circulatory failure, hemorrhage) |
| Proctitis (functional-<br>symptomatic)<br>Also see Mucositis/<br>Stomatitis for Clinical<br>Exam | Rectal discomfort AND No intervention indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social/ functional activities OR Operative intervention indicated | Life-threatening consequences (eg, perforation) |
| Vomiting | Transient or intermittent vomiting with no or minimal interference with oral intake | Frequent episodes of vomiting with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated | Life-threatening consequences (eg, hypotensive shock) |

| | | NEUROLOGICAL | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alteration in Personality-<br>Behavior or in Mood (eg,<br>agitation, anxiety,<br>depression, mania,<br>psychosis) | Alteration causing no or minimal interference with usual social & functional activities | Alteration causing greater than minimal interference with usual social & functional activities | Alteration causing inability to perform usual social & functional activities | Behavior potentially harmful<br>to self or others (eg,<br>suicidal/homicidal ideation or<br>attempt, acute psychosis) OR<br>Causing inability to perform<br>basic self-care functions |
| Altered Mental Status For Dementia, see Cognitive and Behavioral/Attentional Disturbance (including dementia and ADD) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or somnolence causing greater than minimal interference with usual social & functional activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR obtundation, OR coma |
| Ataxia | Asymptomatic ataxia detectable on exam OR Minimal ataxia causing no or minimal interference with usual social & functional activities | Symptomatic ataxia causing greater than minimal interference with usual social & functional activities | Symptomatic ataxia causing inability to perform usual social & functional activities | Disabling ataxia causing inability to perform basic self-care functions |
| Cognitive and Behavioral/Attentional Disturbance (including dementia and Attention Deficit Disorder) | Disability causing no or<br>minimal interference with<br>usual social & functional<br>activities OR Specialized<br>resources not indicated | Disability causing greater than<br>minimal interference with<br>usual social & functional<br>activities OR Specialized<br>resources on part-time basis<br>indicated | Disability causing inability to<br>perform usual social &<br>functional activities OR<br>Specialized resources on a<br>full-time basis indicated | Disability causing inability to<br>perform basic self-care<br>functions OR<br>Institutionalization indicated |
| CNS Ischemia (acute) | NA | NA | Transient ischemic attack | Cerebral vascular accident (CVA, stroke) with neurological deficit |
| Developmental delay – Pediatric ≤ 16 Years | Mild developmental delay,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate<br>for the setting | Moderate developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Severe developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Developmental regression,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate for<br>the setting |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated (other than ER visit) OR Headache with significant impairment of alertness or other neurologic function |
| Insomnia | NA | Difficulty sleeping causing greater than minimal interference with usual social/functional activities | Difficulty sleeping causing inability to perform usual social & functional activities | Disabling insomnia causing inability to perform basic self-care functions |
| Neuromuscular Weakness (including myopathy & neuropathy) | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & functional activities | Muscle weakness causing greater than minimal interference with usual social & functional activities | Muscle weakness causing inability to perform usual social & functional activities | Disabling muscle weakness causing inability to perform basic self-care functions OR Respiratory muscle weakness impairing ventilation |
| Neurosensory Alteration<br>(including paresthesia and<br>painful neuropathy) | Asymptomatic with sensory alteration on exam or minimal paresthesia causing no or minimal interference with usual social & functional activities | Sensory alteration or<br>paresthesia causing greater<br>than minimal interference with<br>usual social & functional<br>activities | Sensory alteration or paresthesia causing inability to perform usual social & functional activities | Disabling sensory alteration or paresthesia causing inability to perform basic self-care functions |
| Seizure: (new onset) | NA | 1 seizure | 2–4 seizures | Seizures of any kind that are<br>prolonged, repetitive (eg,<br>status epilepticus), or difficult<br>to control (eg, refractory<br>epilepsy) |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Seizure: (pre-existing) For Worsening of Existing Epilepsy the Grades Should Be Based on an Increase from Previous Level of Control to Any of These Levels | NA | Increased frequency of pre-<br>existing seizures (non-<br>repetitive) without change in<br>seizure character OR<br>infrequent breakthrough<br>seizures while on stable meds<br>in a previously controlled<br>seizure disorder | Change in seizure character<br>from baseline either in<br>duration or quality (eg,<br>severity or focality) | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure — Pediatric < 18 Years | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>< 5 minutes with < 24 hours<br>post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting 5–20<br>minutes with<br>< 24 hours post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>> 20 minutes | Seizure, generalized onset<br>with or without secondary<br>generalization, requiring<br>intubation and sedation |
| Syncope (not associated with a procedure) | NA | Present | NA | NA |
| Vertigo | Vertigo causing no or<br>minimal interference with<br>usual social & functional<br>activities | Vertigo causing greater than<br>minimal interference with<br>usual social & functional<br>activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo causing inability to perform basic self-care functions |

| | MUSCULOSKELETAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia See also Arthritis | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain causing inability to perform basic self-care functions |
| Arthritis<br>See also Arthralgia | Stiffness or joint swelling causing no or minimal interference with usual social & functional activities | Stiffness or joint swelling causing greater than minimal interference with usual social & functional activities | Stiffness or joint swelling causing inability to perform usual social & functional activities | Disabling joint stiffness or<br>swelling causing inability to<br>perform basic self-care<br>functions |
| Bone Mineral Loss | BMD t-score or z-score –2.5 to –1.0 | BMD t-score or z-score < -2.5 | Pathological fracture (including loss of vertebral height) | Pathologic fracture causing life-threatening consequences |
| Pediatric < 21 Years | BMD z-score<br>-2.5 to -1.0 | BMD z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Myalgia<br>(non-injection site) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain causing inability to perform basic self-care functions |
| Osteonecrosis | NA | Asymptomatic with radiographic findings AND No operative intervention indicated | Symptomatic bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain with radiographic findings causing inability to perform basic self-care functions |

| | SYSTEMIC | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Acute Systemic Allergic<br>Reaction | Localized urticaria<br>(wheals) with no medical<br>intervention indicated | Localized urticaria with medical intervention indicated OR Mild angioedema with no medical intervention indicated | Generalized urticaria OR<br>Angioedema with medical<br>intervention indicated OR<br>Symptomatic mild<br>bronchospasm | Acute anaphylaxis OR Life-<br>threatening bronchospasm OR<br>laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Fatigue<br>Malaise | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating fatigue/malaise<br>symptoms causing inability to<br>perform basic self-care<br>functions |
| Fever (nonaxillary) | 37.7°C to 38.6°C<br>99.8°F to 101.5°F | 38.7°C to 39.3°C<br>101.6°F to 102.8°F | 39.4°C to 40.5°C<br>102.9°F to 104.9°F | > 40.5°C<br>> 104.9°F |
| Pain- Indicate Body Site<br>See also Injection Site<br>Pain, Headache,<br>Arthralgia, and Myalgia | Pain causing no or<br>minimal interference with<br>usual social & functional<br>activities | Pain causing greater than minimal interference with usual social & functional activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization (other than ER visit) indicated |
| Unintentional Weight<br>Loss | NA | 5% to 9% loss in body weight from baseline | 10% to 19% loss in body<br>weight from baseline | ≥ 20% loss in body weight<br>from baseline OR Aggressive<br>intervention indicated [eg,<br>tube feeding or total parenteral<br>nutrition] |

| | INJECTION SITE REACTION | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Injection Site Pain (pain without touching) Or Tenderness (pain when area is touched) | Pain/tenderness causing no<br>or minimal limitation of use<br>of limb | Pain/tenderness limiting use of limb OR Pain/tenderness causing greater than minimal interference with usual social & functional activities | Pain/tenderness causing inability to perform usual social & functional activities | Pain/tenderness causing inability<br>to perform basic self-care<br>function OR Hospitalization<br>(other than ER visit) indicated<br>for management of<br>pain/tenderness |
| Injection Site Reaction (Localized), > 15 Years | Erythema OR Induration<br>of $5 \times 5$ cm to $9 \times 9$ cm (or<br>$25-81 \times \text{cm}^2$ ) | Erythema OR Induration OR<br>Edema > 9 cm any diameter<br>(or > 81 cm <sup>2</sup> ) | Ulceration OR Secondary<br>infection OR Phlebitis OR<br>Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pediatric ≤ 15 Years | Erythema OR Induration<br>OR Edema present but<br>≤ 2.5 cm diameter | Erythema OR Induration<br>OR Edema > 2.5 cm<br>diameter but < 50% surface<br>area of the extremity<br>segment (eg, upper<br>arm/thigh) | Erythema OR Induration OR Edema involving ≥ 50% surface area of the extremity segment (eg, upper arm/thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pruritis Associated with<br>Injection<br>See also Skin: Pruritis<br>(itching—no skin lesions) | Itching localized to injection<br>site AND Relieved<br>spontaneously or with<br>< 48 h treatment | Itching beyond the injection site but not generalized OR Itching localized to injection site requiring ≥ 48 h treatment | Generalized itching causing inability to perform usual social & functional activities | NA |

| | ENDOCRINE/METABOLIC | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipodystrophy (eg, back of neck, breasts, abdomen) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious changes on casual visual inspection | NA |
| Diabetes Mellitus | NA | New onset without need to initiate medication OR Modification of current meds to regain glucose control | New onset with initiation of indicated med OR Diabetes uncontrolled despite treatment modification | Life-threatening consequences (eg, ketoacidosis, hyperosmolar non-ketotic coma) |
| Gynecomastia | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |
| Hyperthyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, thyroid storm) |
| Hypothyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, myxedema coma) |
| Lipoatrophy (eg, fat loss from the face, extremities, buttocks) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |

| GENITOURINARY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Intermenstrual Bleeding (IMB) | Spotting observed by participant<br>OR Minimal blood observed<br>during clinical or colposcopic<br>exam | Intermenstrual bleeding not greater in duration or amount than usual menstrual cycle | Intermenstrual bleeding greater in duration or amount than usual menstrual cycle | Hemorrhage with life-<br>threatening hypotension OR<br>Operative intervention<br>indicated |
| Urinary Tract obstruction (eg, stone) | NA | Signs or symptoms of urinary tract obstruction without hydronephrosis or renal dysfunction | Signs or symptoms of urinary tract obstruction with hydronephrosis or renal dysfunction | Obstruction causing life-<br>threatening consequences |

| | INFECTION | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Infection (any other than HIV infection) | Localized, no systemic antiµbial treatment indicated AND Symptoms causing no or minimal interference with usual social & functional activities | Systemic antiµbial treatment indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Systemic antiubial treatment indicated AND Symptoms causing inability to perform usual social & functional activities OR Operative intervention (other than simple incision and drainage) indicated | Life-threatening consequences (eg, septic shock) |

Basic Self-care Functions: Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.

Usual Social & Functional Activities: Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc.

# Appendix 5. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

### 1) Pregnancy and Contraception Requirements for Males and Females of Childbearing Potential

The risks of treatment with GS-9620 during pregnancy have not been evaluated in humans. Please refer to the latest version of the investigator's brochure for GS-9620 for the treatment of chronic hepatitis B virus and HIV-1 infection for additional information.

#### 2) Definition of Female of Childbearing Potential

For the purposes of this study, a female subject of childbearing potential is a nonmenopausal female who has not had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure. This definition includes a pubertal female who has not yet started menstruating. A woman who has had a tubal sterilization is considered to be of childbearing potential.

A female subject may be considered menopausal in either of the following conditions:

- Surgical menopause: Appropriate medical documentation of prior complete bilateral oophorectomy (ie, surgical removal of the ovaries and occurring at the age at which the procedure was performed)
- Spontaneous menopause: Permanent cessation of previously occurring menses as a result of ovarian failure with documentation of hormonal deficiency by a certified health care provider. The worldwide mean age of spontaneous menopause is 49.24 (SD 1.73) years
- A hormonal deficiency should be properly documented in the case of suspected spontaneous menopause as follows:
  - If age ≥54 years and with the absence of normal menses: serum follicle stimulating hormone (FSH) level elevated to within the postmenopausal range based on the laboratory reference range where the hormonal assay is performed
  - If age <54 years and with the absence of normal menses: negative serum or urine human chorionic gonadotropin (hCG) with concurrently elevated serum FSH level in the postmenopausal range, depressed estradiol (E2) level in the postmenopausal range, and absent serum progesterone level, based on the laboratory reference ranges where the hormonal assays are performed

#### 3) Contraceptive Requirements

Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to utilize protocol specified methods of contraception from the screening/enrollment visit throughout the study period and for 36 days following the last dose of study drug. Female study subjects who are not heterosexually active must provide periodic confirmation of continued abstinence from heterosexual intercourse and regular pregnancy testing while taking GS-9620 or placebo. The investigator will counsel subjects on the protocol specified method(s) for avoiding pregnancy in case the subject chooses to engage in heterosexual intercourse.

Protocol specified contraceptive methods are as follows: (1) a combination of one hormonal method and one barrier method; or (2) use of an intrauterine device (IUD) or tubal sterilization; see Appendix Table 1. Acceptable hormonal methods include injectable progesterone, progesterone implants, combination oral contraceptives, transdermal contraceptive patch, and vaginal ring. An acceptable barrier method is the male condom. Female subjects must use a hormonal method if the partner has a vasectomy. If a subject has undergone tubal sterilization or has had a Copper T 380A IUD or LNg 20 IUD inserted, no other contraception is needed.

If tubal sterilization is via the Essure procedure, verification of tubal blockage by hysterosalpingogram (HSP) must be performed approximately 3 months after microinsertion. Prior to verification, Essure is not considered a reliable form of contraception and the contraception methods described below must be used. Female subjects who utilize hormonal contraceptives as one of their birth control methods must have used the same method for at least 3 months before study dosing.

Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline (Day 1) prior to receiving the first dose of study drug. Lactating females must discontinue nursing before IMP administration.

**Appendix Table 1. Protocol Specified Contraceptive Methods** 

| Single Methods | <b>Combination Methods</b> |
|---|---|
| Intrauterine Devices (IUDs) Copper T 380A IUD LNg 20 IUD Tubal Sterilization | Estrogen and Progesterone plus Barrier Combined oral contraceptives plus condom* Transdermal patch plus condom* Vaginal ring plus condom* Implant plus condom* Injection plus condom* Partner's vasectomy must be used with a hormonal method. |

<sup>\* (</sup>without spermicide and excluding lambskin)

The investigator will counsel all subjects on the most effective method(s) for avoiding pregnancy during the study.

## 4) Additional Requirements for Male Subjects and Recommendations for Partners of Female Subjects

Male subjects must agree to use condoms (without spermicide and excluding lambskin) during heterosexual intercourse and avoid sperm donation while enrolled in the study and for at least 90 days after administration of the last dose of study drug. Partners of female subjects should be encouraged to use condoms during heterosexual intercourse while enrolled in the study.

Use of condoms, with or without spermicide, has been proven to decrease the risk of transmission of HIV and other sexually transmitted diseases. The use of spermicide is not recommended if the subject or subject's partner is infected with HIV.

### 5) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study, or if they become pregnant within 30 days or 4 weeks of last study drug dose. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant during the study must report the information to the investigator. Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.7.2.1.

### Appendix 6. Definitions of Stage 3 Opportunistic Illnesses in HIV (CDC Guidelines)

- Candidiasis of bronchi, trachea, or lungs
- Candidiasis of esophagus
- Cervical cancer, invasive
- Coccidioidomycosis, disseminated or extrapulmonary
- Cryptococcosis, extrapulmonary
- Cryptosporidiosis, chronic intestinal (> 1 month duration)
- Cytomegalovirus disease (other than liver, spleen or nodes)
- Cytomegalovirus retinitis (with loss of vision)
- Encephalopathy, HIV-related
- Herpes simplex: chronic ulcer(s) (> 1 month duration); or bronchitis, pneumonitis or esophagitis
- Histoplasmosis, disseminated or extrapulmonary
- Isosporiasis, chronic intestinal (> 1 month duration)
- Kaposi's sarcoma
- Lymphoma, Burkitt's (or equivalent term)
- Lymphoma, immunoblastic (or equivalent term)
- Lymphoma, primary, of brain
- Mycobacterium avium complex or Myobacterium kansasii, disseminated or extrapulmonary
- Mycobacterium tuberculosis, of any site, pulmonary, disseminated or extrapulmonary
- Mycobacterium, other species or unidentified species, disseminated or extrapulmonary
- Pneumocystis jirovecii (previously known as "Pneumocystis carinii) pneumonia
- Pneumonia, recurrent
- Progressive multifocal leukoencephalopathy
- Salmonella septicemia, recurrent
- Toxoplasmosis of brain
- Wasting syndrome attributed to HIV infection

CDC Stage-3-Defining Opportunistic Illnesses in HIV Infection - 2014 (Schneider 2008)